# Statistical Analysis Plan

# TauRx Therapeutics Ltd TRx-237-020

# An Open-Label, Extension Study of the Effects of Leuco-methylthioninium bis(hydromethanesulfonate) in Subjects with Alzheimer's Disease or Behavioral Variant Frontotemporal Dementia

**VERSION 3.0, 24 March 2016** 

**Sponsor:** TauRx Therapeutics Ltd

Liberty Building, Foresterhill Road, Aberdeen AB25 2ZP,

Scotland, UK

Prepared by: Paul A. Pappas, MS

SynteractHCR, Inc.

5759 Fleet Street, Suite 100

Carlsbad, CA 92008

Version: Version 1.3

**Date:** 30 March 2017

# Approval

Upon review of this document, including table, listing, and figure shells, the undersigned approves the Statistical Analysis Plan. The analysis methods and data presentation are acceptable.

| Signature | Date |
|---|---|
| Professor Claude Wischik Executive Chairman TauRx Therapeutics Ltd. | 3/4/17 |
| Dr. W. Maddland, CMO VP Clinical Development TarRx Therapeutics Ltd. | 07APR-17 |
| Charles Davis. Ph.D. Biostatistics Consultant CSD Biostatistics, Inc. | 30 M.AR. 2017 |
| Paul A. Pappas, MS Biostatistician Synteract | 30Mar2017 |

# TABLE OF CONTENTS

| LIS | ST OF | ABBREVIATIONS | 5 |
|---|---|---|---|
| 1. | INT | RODUCTION | 8 |
| 2. | STU | DY OBJECTIVES | 8 |
| 3. | STU | DY DESIGN AND PLAN | 8 |
| | 3.1 | SCHEDULE OF ASSESSMENTS | 10 |
| | 3.2 | ASSIGNMENT OF TREATMENT | |
| | 3.3 | STUDY TREATMENT | |
| 4. | GEN | NERAL ANALYSIS CONSIDERATIONS | 13 |
| | 4.1 | Conventions | 14 |
| | 4.2 | STANDARD CALCULATIONS | |
| | 4.3 | HANDLING PARTIAL DATES | 16 |
| | 4.4 | Visit Windows | 17 |
| 5. | STU | DY POPULATION | 17 |
| | 5.1 | ANALYSIS POPULATION | 17 |
| | 5.2 | SUBJECT DISPOSITION | 18 |
| | 5.3 | PROTOCOL DEVIATIONS | |
| | 5.4 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | |
| | 5.5 | MEDICAL HISTORY | |
| | 5.6 | CONCOMITANT MEDICATIONS | |
| 6. | EXT | TENT OF EXPOSURE | 21 |
| 7. | SAF | ETY ANALYSES | 23 |
| | 7.1 | ADVERSE EVENTS | 23 |
| | 7.2 | CLINICAL LABORATORY EVALUATION | 26 |
| | 7.3 | VITAL SIGNS | 27 |
| | 7.4 | PHYSICAL AND NEUROLOGICAL EXAMINATIONS AND SEROTONIN SYNDROME | |
| | | XICITY) | |
| | 7.5 | ELECTROCARDIOGRAPHY | |
| 8. | OTI | HER ASSESSMENTS | |
| | 8.1 | MMSE | |
| | 8.2 | EQ-5D-5L | |
| | 8.3 | RUD LITE | |
| 9. | CHA | ANGES TO PROTOCOL-SPECIFIED ANALYSES | 31 |
| AP | PENI | DICES | 32 |
| | APP | ENDIX A: POST-DOSE VISIT WINDOWS | 32 |
| | APP | ENDIX B: CRITERIA FOR DETERMINING POTENTIALLY CLINICALLY SIGNIFICANT VA | LUES |
| | in L | ABORATORY TEST RESULTS | 33 |

| APPENDIX C: CRITERIA FOR DETERMINING POTENTIALLY CLINICALLY SIGNIFIC | CANT VALUES |
|---|---|
| IN VITAL SIGNS | 34 |
| APPENDIX D: RULES FOR DETERMINING "WORST" VALUE | 35 |
| APPENDIX E: RULES FOR SCORING THE MMSE | 37 |
| APPENDIX F: LIST OF TABLES, FIGURES AND LISTINGS | 38 |
| APPENDIX G: TABLE LAYOUTS | 54 |
| APPENDIX H: FIGURE LAYOUTS | 105 |
| APPENDIX I: LISTING LAYOUTS | 109 |

| LIST OF ABBRI | EVIATIONS |
|---------------|--------------------------------------------|
| AChEI | acetylcholinesterase inhibitor |
| AD | Alzheimer's Disease |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALK-P | alkaline phosphatase |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | body mass index |
| BP | blood pressure |
| bpm | beats per minute |
| bvFTD | behavioral variant Frontotemporal Dementia |
| °C | degrees Celsius |
| CA | Competent Authority |
| CK | creatine kinase |
| cm | centimeter(s) |
| CNS | central nervous system |
| CRF | case report form |
| CS | clinically significant |
| CSR | clinical study report |
| DBP | diastolic blood pressure |
| EC | Ethics Committee |
| ECG | electrocardiogram |
| eGFR | estimated glomerular filtration rate |
| EQ-5D-5L | EuroQol – 5 Dimension – 5 Level |
| g, kg, mg | gram, kilogram, milligram |
| GGT | gamma-glutamyl transpeptidase |
| HCT | hematocrit |
| HR | heart rate |
| ICH | International Conference on Harmonisation |
| IP | investigational product |

| LIST OF ABBRI | EVIATIONS |
|---------------|---------------------------------------------------|
| IRB | Institutional Review Board |
| IWRS | interactive web response system |
| K | Potassium |
| L, dL, mL | liter, deciliter, milliliter |
| LDH | lactate dehydrogenase |
| LMTM | leuco-methylthioninium bis(hydromethanesulfonate) |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean cell volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mEq | milliequivalent |
| mmHg | millimeters of mercury |
| mmol | millimole |
| MMSE | Mini-Mental State Examination |
| msec | millisecond |
| Na | Sodium |
| NCS | Non-clinically significant |
| PCS | Potentially Clinically Significant |
| PCST | Treatment-emergent PCS post-baseline worsening |
| PT | MedDRA preferred term |
| QTcB | Bazett's QT correction |
| QTcF | Fridericia's QT correction |
| RBC | red blood cell |
| RTF | rich text format |
| RUD Lite | Resource Utilization in Dementia – short version |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAR | serious adverse reaction |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SI | The International System of Units |
| SOC | MedDRA System Organ Class |
| TSH | thyroid stimulating hormone |

| LIST OF ABBR | EVIATIONS |
|--------------|---------------------------|
| ULN | upper limit of normal |
| WBC | white blood cell |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analysis of data collected within the scope of TauRx Therapeutics Ltd Protocol TRx-237-020, An Open-Label, Extension Study of the Effects of Leuco-methylthioninium bis(hydromethanesulfonate) (LMTM) in subjects with Alzheimer's Disease (AD) or Behavioral Variant Frontotemporal Dementia (bvFTD). The purpose of this statistical analysis plan (SAP) is to provide specific guidelines from which the analysis will proceed. Any deviations from these guidelines will be documented in the clinical study report (CSR).

This SAP is based on the final protocol Version 3.0, approved 24 March 2016. The data presented for this study will characterize subjects at study entry and report safety data restricted to study-emergent information.

#### 2. STUDY OBJECTIVES

The primary objectives of this open-label extension study of LMTM in subjects with AD or byFTD are:

- 1. To provide subjects who have completed participation in a Phase 2 or Phase 3 trial continued access to therapy, and
- 2. To evaluate the long-term safety and tolerability of LMTM given in flexible doses of up to 300 mg/day, or in those countries where limited by a Competent Authority (CA) or Ethics Committee (EC), 200 mg/day.

#### 3. STUDY DESIGN AND PLAN

This study is a multicenter, open-label extension study of LMTM in subjects with mild to moderate AD or bvFTD at the time they first enrolled in a double-blind trial sponsored by TauRx. Specifically, participation in this study will be offered to any subject who completed participation in Studies TRx-237-005, TRx-237-008, or TRx-237-015 (AD subjects) or TRx-237-007 (bvFTD subjects). Only AD subjects who have completed the full double-blind period of the originating studies (including the one-month post-treatment follow-up), or bvFTD subjects who completed the full double-blind treatment period through Visit 9 in TRx-237-007, are eligible for inclusion in this open-label extension study.

The study will be open only to approximately 170 participating sites in North America, Asia, Australia, and Europe.

Subjects may enter this study at the final designated visit in the double-blind study, provided subjects and caregivers have had sufficient time to consider the study prior to giving consent, or at any subsequent time. Subjects may continue participation at the same site at which they participated in the originating double-blind study or, if an AD subject, transfer to a geographically close investigational site (that also participated in the same study). Eligibility for continued open-label treatment is to be determined by the original investigator and, if applicable, a referral to a new site made. The new investigator will have access to the subject's prior study case report forms (CRFs) and is to confirm eligibility. Baseline testing can be repeated as necessary in the judgment of the new investigator. The initial visit will be designated Visit 1. Study drug will be dispensed at each visit, beginning with Visit 1. The study drug will be dispensed in 13-week (± 2-week) supplies.

The first on-treatment visit will occur approximately 2 weeks after Visit 1 (designated Visit 2) for the initial post-treatment safety assessment. During the first year, post-Baseline study visits will occur at approximately 2 weeks (Visit 2), 13 weeks (Visit 3), 26 weeks (Visit 4), 39 weeks (Visit 5), and 52 weeks (Visit 6) after Baseline. Required assessments will be performed at all visits as described in the Schedule of Assessments in Section 3.1. Caregivers will be contacted by telephone at the mid-point between Visits 2 and 3; they will also be asked to contact the investigator in response to any safety concern. An unscheduled visit will be arranged to assess the subject as needed.

Continued participation will be re-evaluated approximately every 12 months on the basis of safety, tolerability, and continued benefit as judged by the investigator. Subjects deemed eligible for continued treatment (and their caregivers) must provide informed consent for re-enrollment. Subjects for whom consent is not provided consistent with national requirements and IRB/EC approval will be discontinued.

For subjects who cease to take LMTM, a post-treatment follow-up visit 4 weeks after the last dose of study drug is to be scheduled, regardless of the reason for discontinuation. Subjects who fail to complete the initial 12-month extension period will not be eligible to continue to receive treatment during any subsequent extension period.

A schematic representation of the first 12 months of the study is provided in Table 3-1.

| Table 3-1 Schematic Representation of Study (First 12 Months) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 1 <sup>st</sup><br>Dose | | | | | | Last<br>Dose | Follow-up (4 wks after last |
| Visit | 1 | 2 | (T)* | 3 | 4 | 5 | 6 | dose) |
| Week | 0 | 2 | 5 | 13 | 26 | 39 | 52 | 56 |
| Day | 1 | 15 | 43 | 92 | 183 | 274 | 365 | 393 |
| (±days) | | (3) | (14) | (14) | (14) | (14) | (14) | (14) |

<sup>\*</sup>A telephone contact (T) will occur between the scheduled Weeks 2 and 13 study visits (at approximately Week 6). Note: The same 13-week visit schedule will be maintained for continued treatment beyond the first 12 months (if there is re-consent approximately every 12 months), with no requirement for the Week 2 visit in the second or any subsequent year of participation.

#### 3.1 Schedule of Assessments

Baseline safety assessments may be made at the final designated visit of the prior TauRx study in which the subject was enrolled. For purposes of the open-label extension, these will be designated as Baseline (Visit 1, Day 1). If Visit 1 does not coincide with the final designated visit of the previous double-blind study of participation, medical history, concomitant medication use, and adverse events (AEs) should be updated; serum pregnancy testing should be performed in women of childbearing potential. If more than 42 days have elapsed since that final visit, additional baseline safety assessments must be repeated. The additional safety assessments include clinical laboratory testing (e.g., hematology and serum chemistry panels), vital signs (seated blood pressure and pulse, temperature, and respirations), body weight, targeted physical and neurological examinations (including an assessment for signs and symptoms of serotonin toxicity), and 12-lead Electrocardiogram (ECG). If needed to confirm eligibility or to evaluate an AE, unscheduled local 12-lead ECG testing and/or physical and neurological examinations may be performed if judged to be required by the investigator for any given subject. Baseline assessments may be repeated (also within 42 days) as determined by the new investigator for AD subjects transferring to a different site.

Safety assessments (described further in Section 7 of the TRx-237-020 protocol) will be repeated at each visit, i.e., approximately 2 weeks post-Baseline and at visits occurring approximately every 3 months (13 weeks) relative to Baseline (or upon early termination). These assessments include adverse event and concomitant medication recording, vital signs (seated blood pressure and pulse, temperature, and respirations), body weight, targeted physical and neurological examinations (including an assessment for signs and symptoms of serotonin toxicity), clinical laboratory testing (e.g., hematology and serum chemistry panels), and serum pregnancy testing in women of childbearing potential. A

12-lead ECG will be obtained in triplicate approximately every 6 months (or upon early termination).

The EuroQol – 5 Dimension – 5 Level (EQ-5D-5L) scale, applied to the subject and to the caregiver on behalf of the subject, will be evaluated at Baseline (as it is not used in the Phase 3 studies of prior participation). The Resource Utilization in Dementia – short version (RUD Lite) will be also be evaluated at Baseline if not available from within the prior 42 days. These evaluations will be repeated approximately every 6 months, i.e., approximately 26 and 52 weeks after Baseline.

The same 13-week schedule of in-clinic safety assessments will be maintained for continued treatment beyond the first 12 months (if there is re-consent approximately every 12 months), with no requirement for the Week 2 visit or Week 6 telephone contact in the second or any subsequent year of participation. Continued treatment will be restricted to those subjects for whom continued benefit is expected by the investigator to outweigh risk and informed consent is provided.

Additional targeted examinations may be performed as clinically indicated (e.g., in the event of an AE that requires such follow up or any reported change in the subject's physical condition).

Post-treatment safety assessments will be conducted at the follow-up visit to be scheduled to occur approximately 4 weeks after the last dose of study drug (End of Treatment or Early Termination). These visits should be scheduled for all subjects.

A schedule of assessments (the first 12 months of the study) is shown in Table 3-2.

Table 3-2: Schedule of Assessments (First 12 Months)

| Visit Name | Baseline | F | First 12 | Month C | pen-Lab | el Extension | Follow |
|---|---|---|---|---|---|---|---|
| Overall Visit Number: | 1 | 2* | 3 | 4 | 5 | 6 (End of Treatment or Early Termination) | -up |
| Months Relative to Baseline Days | | | 3 | 6 | 9 | 12 | 13 |
| Weeks Relative to Baseline Days | | 2 | 13 | 26 | 39 | 52 | 56 |
| (Allowable Time Window in days): | | (±3) | (±14) | (±14) | (±14) | (±14) | (±14) |
| Informed Consent (Subject and Caregiver) (M) | X | | | | | X | |
| Inclusion/Exclusion Criteria Review (M) | X | | | | | | |
| Concomitant Medication Recording/<br>Review (M) | X | X | X | X | X | X | X |
| Adverse Events / Medical History Review (M) | X | X | X | X | X | X | X |
| Study Drug Dispensing | X | | X | X | X | X | |
| Study Drug Compliance Assessment | | X | X | X | X | X | |
| Blood Samples for Laboratory Tests | X | X | X | X | X | X | X |
| Serum Pregnancy Test (women of childbearing potential) | X | X | X | X | X | X | X |
| Seated Blood Pressure and Pulse | X | X | X | X | X | X | X |
| Temperature and Respiratory Rate | X | X | X | X | X | X | X |
| Body Weight | X | X | X | X | X | X | X |
| ECG | X | | | X | | X | X |
| Physical and Neurological Exam (including an assessment for signs and symptoms of serotonin toxicity) | X | X | X | X | X | X | X |
| MMSE (to inform the evaluation for possible serotonin toxicity) | X | | | X | | X | X |
| RUD Lite | X | | | X | | X | |
| EQ-5D-5L | X | | | X | | X | |

<sup>\*</sup>A documented telephone contact will occur between the scheduled Visit 2 and 3 study visits, scheduled to occur at approximately Week 6 ( $\pm$  14 days) and will include AE and concomitant medication review.

Note: The same 13-week schedule of in-clinic safety assessments will be maintained for continued treatment beyond the first 12 months (if there is re-consent approximately every 12 months), with no requirement for the Week 2 visit in the second or any subsequent year of participation.

### 3.2 Assignment of Treatment

This is not applicable to this open-label study as all subjects will receive LMTM.

Treatment assignment from the prior double-blind clinical study will be recorded in a listing.

Subjects will be assigned a study identification number with the first three digits for the study (020), the next two letters for the country, the next three digits for the site, and the last two digits for the sequential order of enrollment at a given site. These study identification numbers will be listed along with the subject's study identification number in the prior study. Subjects that have switched sites for this study will be flagged.

#### 3.3 Study Treatment

Study drug is provided as 100-mg tablets. The intended schedule of dosing is twice daily, with or without meals.

The initial LMTM dose for all subjects will be 200 mg/day, except for subjects from Study TRx-237-007 who were taking a reduced dose (i.e., 100 mg/day) and who should continue taking this reduced regimen upon entering this extension study. Thereafter, dosing will be flexible (in 100-mg decrements or increments). The dose may be increased (at Visit 3 or at any subsequent dispensing visit as determined by the investigator during the treatment period) or decreased (at any time at or after Visit 2) in response to benefit as judged by the investigator and safety and tolerability. The maximum allowable dose is 300 mg/day (or in those countries where limited by a CA or EC, 200 mg/day). The dose may also be interrupted at any time as needed (for up to 30 days at any one time). Study drug and regimens, including dose interruptions and modifications in response to adverse events, are further described in Section 6 of the TRx-237-020 protocol.

#### 4. GENERAL ANALYSIS CONSIDERATIONS

The Safety population will include all subjects who take at least one dose of study drug. All analyses described in this SAP will be based on the Safety Population. All subjects entering the study, even if not known to have taken a dose, will be accounted for in a listing.

The statistical analyses will be reported using summary tables, figures, and data listings. Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentage of subjects in corresponding categories.

For purposes of calculations of change from baseline, Baseline (Visit 1) for the open-label study will be used. Depending on the parameter, the data may have been acquired during the double-blind study of prior participation.

Summary tables will present results by diagnosis (AD or bvFTD) and an "All Subjects" column.

Individual subject data obtained from the CRFs (including mapped data<sup>1</sup>), central clinical laboratory (local laboratory results are entered on the CRFs), and any derived data will be presented by subject in data listings. Listings will include relative study day, where negative values will indicate visits prior to first dose of study drug in 020, and any data collected after discontinuation of study drug will be flagged as follow-up. All data captured on the CRF, including specific descriptions of 'other' and comments fields, will be included on the listings. Listings will be sorted by subject number.

All analyses and tabulations will be performed using SAS® Version 9.4 or higher. Tables, listings, and figures will be presented in RTF format. Upon completion, all SAS® programs will be validated by an independent programmer. In addition, all program output will undergo a senior level statistical review. The validation process will be used to confirm that statistically valid methods have been implemented and that all data manipulations and calculations are accurate. Checks will be made to ensure accuracy, consistency with this plan, consistency within tables, and consistency between tables and corresponding data listings. Upon completion of validation and quality review procedures, all documentation will be collected and filed by the project statistician or designee.

#### 4.1 Conventions

The precision of original measurements will be maintained in summaries, when possible. Means, medians and standard deviations will be presented with an increased level of precision; means and medians will be presented to one more decimal place than the raw data, and the standard deviations will be presented to two more decimal places than the raw data.

<sup>&</sup>lt;sup>1</sup> Mapped data consists of medical history, concomitant medication, and AE data obtained during the prior studies and imported into the 020 database (for handling of these data see Sections 5.5, 5.6, and 7.1, respectively).

Unless otherwise specified, summaries of continuous variables that have some values recorded using approximate values (e.g., < or >) will use imputed values. The approximate values will be imputed using the closest exact value for that measurement. For tables where rounding is required, rounding will be done to the nearest round-off unit. For example, if the round-off unit is the ones place (i.e., integers), values  $\ge$  XX.5 will be rounded up to XX+1 while values < XX.5 will be rounded down to XX.

For percentages, unless they are calculated to be exactly 0% or 100%, values of very small or very large percentages will be reported as <0.1% and >99.9%.

For by-visit tables, percentages will be based on available data and denominators will generally exclude subjects with missing values. For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the subjects discontinue due to "lost to follow-up", this reason will be included in the table with a count of 0.

#### 4.2 Standard Calculations

Variables requiring calculation will be derived using the following formulas:

- **Baseline** A baseline value, unless specified otherwise, is the last non-missing value recorded prior to the first dose of study drug in 020. If an assessment has the same date as the date of first dose of study drug in 020, the assessment will be counted as baseline (depending on the parameter, the data may have been acquired during the double-blind study of prior participation).
- **Study day** For a given date (*date*), study day is calculated as days since the date of first dose of study drug in the open-label extension (*firstdose*):

```
Study day = date - firstdose + 1, where date \geq firstdose Study day = date - firstdose, where date \leq firstdose
```

- **Days** Durations, expressed in days, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in days = (date2-date1+1).
- Weeks Durations, expressed in weeks, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in weeks = (date2-date1+1)/7.
- **Months** Durations, expressed in months, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in months = (date2-date1+1)/30.4375.

- Years Durations, expressed in years, between one date (*date1*) and another later date (*date2*) are calculated using the following formula: duration in years = (date2-date1+1)/365.25.
- Body Mass Index (BMI) BMI  $(kg/m^2)$  = weight (kg) /  $[height (cm)/100]^2$
- Estimated Glomerular Filtration Rate (eGFR) eGFR (mL/min/1.73 m<sup>2</sup>) = 175 × (serum creatinine in mg/dL)<sup>-1.154</sup> × (Age in years)<sup>-0.203</sup> × (0.742 if female) × (1.212 if African American).

Note that age on consent date is collected on the CRF and will not be calculated.

#### 4.3 Handling Partial Dates

If only a partial date is available and is required for a calculation, the following standards will be applied:

#### Start dates

- a. For missing start day only in 020 Day will be imputed as the first day of the month (i.e., 1) with the following exception: if the partial date falls in the same month and year as the date being used in the calculation (e.g., first dose date in 020, informed consent date for 020), then the partial date will be imputed to equal the date being used for the calculation. If the partial date is used for multiple calculations, then the earliest date will be used.
- b. For missing start day and month in 020 Day and month will be imputed as the first day of the year (i.e., 1 January) with the following exception: if the partial date falls in the same year as the date being used in the calculation (e.g., first dose date in 020, informed consent date for 020), then the partial date will be imputed to equal the date being used for the calculation. If the partial date is used for multiple calculations, then the earliest date will be used.
- c. For missing start day only that is mapped from a previous study Day will be imputed as the first day of the month (i.e., 1) with the following exception: if the partial date falls in the same month and year as the date being used in the calculation (e.g., first dose date, informed consent date), then the partial date will be imputed to equal the date being used for the calculation. If the partial date is used for multiple calculations, then the earliest date will be used.
- d. For missing start day and month that is mapped from a previous study Day and month will be imputed as the first day of the year (i.e., 1 January) with the following exception: if the partial date falls in the same year as the date

being used in the calculation (e.g., first dose date, informed consent date), then the partial date will be imputed to equal the date being used for the calculation. If the partial date is used for multiple calculations, then the earliest date will be used.

#### Stop dates

- a. For missing stop day only Day will be imputed as the last day of the month (i.e., 28, 29, 30, or 31) or the last day of study contact if earlier
- b. For missing stop day and month Day and month will be imputed as the last day of the year (i.e., 31 December) or the last day of study contact if earlier

The date of last dose of study drug will be taken from the Study Exit Status CRF page. If this is missing, then the last visit date, excluding the follow-up visit, will be used, unless a data review indicates a different date. Similarly, if other key dates are missing, a review will be undertaken to aid imputation of these.

Any partial dates will be displayed in data listings without imputation of missing days and/or months (e.g., MAR2011, 2009).

#### 4.4 Visit Windows

Since study visits do not always take place exactly as scheduled in the protocol, it is necessary to assign the actual observation times to "analysis visit windows" for analysis purposes. Post-baseline visit windows for each target visit are defined in <u>Appendix A</u>, and will be applied to all measurements. For each summary and value if there are multiple values within a visit window, the "worst" value as defined in <u>Appendix D</u> will be used for that visit window summary. These visit windows will be applied to all visits, including scheduled, unscheduled, and early termination visits.

#### 5. STUDY POPULATION

#### 5.1 Analysis Population

The safety population is defined as all subjects who received at least one dose of LMTM in 020. Subjects dispensed study medication who subsequently are lost to follow up without any contact are not included in the Safety Population but will be included in the study disposition tabulation and listings. With the exception of study disposition, all tables and listings will be generated on the basis of the Safety Population.

#### 5.2 Subject Disposition

Subject disposition information will be summarized for all subjects, overall and by region, country and site. Summaries will include: the number of subjects, (discontinued or completed), all reasons for discontinuation, and the primary reason for discontinuation.

The timing of the early discontinuations will be assessed by summarizing discontinuations by reason during each of the following time periods, overall and by region:

- Day 1
- Days 2 53
- Days 54 137
- Days 138 228
- Days 229 319
- Days 320 410
- Days 411 501
- Days 502 591
- Days 592 683
- > 683 Days

#### **5.3** Protocol Deviations

In accordance with ICH E3, Sponsor-defined eligibility violations and important post-baseline protocol deviations will be identified and listed separately by study site and subject. Sources for these deviations may include IWRS, CTMS (Clinical Trial Management System) and the clinical database. Deviations will be classified as follows:

Deviation type/code as provided by Sponsor:

- Informed consent
- Safety
- IP / Treatment deviation
- Other protocol deviations

Deviations are then categorized into:

- Critical
- Major
- Minor

A tabulation of protocol deviations by type/code overall and by categorization will be provided. A by-subject listing of deviations will also be provided.

#### 5.4 Demographic and Baseline Characteristics

Tabular summaries of demographics will be prepared based on data collected at the Baseline visit for the prior study and at the baseline for the open-label extension study. These include the following: age, sex, ethnicity, race and geographic region. Age at informed consent for participation in the prior study will be imported into the 020 CRF from IWRS (it is not entered by the site).

General study-specific baseline characteristics to be summarized include the following: height, weight and body mass index (BMI).

Summaries of demographic and baseline characteristics will also be provided by region, country and site.

Additional demographic and baseline characteristics will be presented in a listing only, including childbearing status (for females), main method of adequate contraception, subject's living accommodation, and with whom they live.

#### 5.5 Medical History

There are two CRFs contributing medical history data.

- Prior Study Medical History CRF: Medical history as recorded during prior studies 005, 007 and 015 will be automatically uploaded to the Prior Study – Medical History CRF and medical history recorded during the 008 study will be recopied from the 008 records by the site to the Prior Study – Medical History CRF.
- Medical History CRF: Medical History discovered since the last visit in the prior study that is considered clinically relevant by the Investigator as well as prior study AEs that, at the Investigator's discretion, are judged clinically relevant will be recorded on the Medical History CRF.

Verbatim terms on CRFs will be coded to preferred term (PT) and system organ class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA) (version 16.0). The coding process is described in the Data Management Plan.

The number and percentage of subjects with a given medical history will be summarized for both CRFs combined for each system organ class and preferred term. The verbatim and coded medical histories from both CRFs will also be included in a listing. Newly added medical history will be flagged.

#### 5.6 Concomitant Medications

There are two CRFs contributing concomitant medication data.

- Prior Study Concomitant Medications CRF: Concomitant medications as recorded during prior studies 005, 007 and 015 will be automatically uploaded to the Prior Study Concomitant Medications CRF. These mapped medications will be available to the investigator at Visit 1 to use as a resource for completing the Concomitant Medications CRF. Concomitant medications recorded during the 008 study will be recopied from the 008 records by the site to the Prior Study Concomitant Medications CRF.
- Concomitant Medications CRF: During Visit 1, all medications that were ongoing at the end of the prior study will be recopied by the site to the Concomitant Medications CRF. At each visit, any changes to existing concomitant medications and any new concomitant medications will be reviewed and recorded in the Concomitant Medications CRF. The date of commencement, dose, and date of any change of dose of concomitant medications are to be recorded.

Verbatim terms on case report forms will be coded to Anatomical Therapeutic Chemical (ATC) classes and Generic Drug Names using the World Health Organization (WHO) dictionary (WHODDE B2, March 1, 2013 release). The coding process is described in the Data Management Plan.

Each of the below summaries will be presented for each of the following:

- 1. Concomitant medications that were ongoing on Day 1 of dosing (pre-existing) source is the Concomitant Medications CRF.
- 2. Concomitant medications that started on or after Day 1 of dosing (study-emergent) source is the Concomitant Medications CRF.
- 3. All concomitant medications, whether pre-existing or study-emergent (merge of ongoing medications from the Prior Study Concomitant Medications CRF and medications that were ongoing on Day 1 of dosing and medications that started on or after Day 1 of dosing from the Concomitant Medications CRF).

Concomitant medications will be summarized by WHO ATC classification level 1 term, ATC level 3 term and Preferred Term (generic name) with frequency and percentage of subjects. At each level of subject summarization, a subject is counted once if he/she reported one or more medications at that level. Each summary will be ordered alphabetically by each level of ATC class and generic drug name within each level of ATC class.

Concomitant medications will be listed with these elements as well as the verbatim drug name. Pre-existing medications, new medications as of the start of this study and medications that are initiated after the last dose of study drug will be flagged.

Prior medications will also be listed (separately). Prior medications are defined as those medications that were either started or ongoing at the end of the prior study participation and were stopped prior to the 020 first dose date.

#### 6. EXTENT OF EXPOSURE

There are four sources of data for determining exposure:

- The date of the first dose is collected on the First Dose of Study Drug CRF.
- The Drug Accountability CRF provides a sequential record of dispensing and return of tablets (including kit ID dispensed and a comment field).
- The Dose Adjustment / Interruption Log CRF provide a record of the start and stop dates of each treatment interruption and dose change (including a comment field).
- The Study Exit Status CRF provides a record of the date of the last dose of study drug.

For each subject, the total duration of exposure, exposure accounting for interruptions, mean and modal daily doses (including a dose of 0 for days not dosed and dose adjustments when applicable), highest daily dose, cumulative dose and dosing compliance, will be summarized descriptively. Notations on the Drug Accountability Log CRF about missed doses are not accounted for programmatically; these will be included in the listing.

Total duration of exposure is defined as the difference between the last dose date and the first dose date, plus 1 day. The total exposure duration defined above includes any periods where the dose is interrupted. A second calculation of exposure duration that excludes dose interruptions will also be performed.

Mean daily dose is calculated as follows:

$$\frac{\sum_{i=1}^{n} Dose_{i}(mg/day) \times Duration(days) \text{ on } Dose_{i}}{Total Duration (days)}$$

The cumulative dose (i.e., the numerator in the above formula) will also be summarized.

Compliance rate over the entire treatment period is calculated using the following formula:

(Total Tablets Dispensed – Total Tablets Returned)

 $\sum_{i=1}^{n} \text{Duration of Dose}_{i} \times \text{Frequency}_{i} - \sum_{j=1}^{m} \text{Duration of Dose Interruption}_{j} \times \text{Frequency of Interrupted Dose}_{j}$ 

#### where

- Duration of Dose<sub>i</sub> is defined as the last dose date the first dose date +1 for the  $i^{th}$  dosing regimen administered.
- Duration of Dose Interruption<sub>j</sub> is defined as the date of dose restart/adjustment the date of the dose interruption for the j<sup>th</sup> dose interruption.
- Frequency<sub>i</sub> is the number of tablets taken daily during the  $i^{th}$  dosing regimen.
- Frequency of Interrupted Dose<sub>j</sub> is the number of tablets taken daily during the dosing regimen that was interrupted.

This analysis will be repeated for subjects who returned an adequate amount of packages to allow for a meaningful calculation.

The frequency and percentage of subjects in the following duration of exposure categories (based on total duration of exposure, inclusive of interruptions) will be presented according to target visit windows defined in Appendix A.

The cumulative number and percentage of subjects across the categories will also be summarized, as well as total subject years of exposure, defined as the sum of exposure in years, will also be presented.

All study drug administration and compliance data will be presented in listings, including chronological dates of administration, number of tablets dispensed and returned with corresponding package ID, treatment duration, mean and modal daily dose, compliance, and any associated comments.

An additional listing will provide a chronological record of study drug administration including the first dose and any subsequent dose increases, reductions, or interruptions, and any associated comments.

#### 7. SAFETY ANALYSES

#### 7.1 Adverse Events

There are two CRFs contributing adverse event data.

- Prior Study Adverse Events CRF: All adverse events as recorded during prior studies 005, 007 and 015 will be automatically uploaded to the Prior Study Adverse Events CRF and and adverse events recorded during the 008 study will be recopied from the 008 records by the site to the Prior Study Adverse Events CRF. The only field that can be modified by the site is the OLEX end date as applicable. Additionally there is a comment field where text can be entered by site.
- Adverse Event CRF: New adverse events or changes to an existing adverse event will be recorded on the Adverse Event CRF.

Adverse events will be coded to SOC and PT using MedDRA (version 16.0). The coding process is described in the Data Management Plan.

AEs are grouped as follows and source(s) of data identified:

- 1. Prior AEs: AEs that were ongoing at the end of the prior study but that resolved before Day 1 of dosing in 020 or that started and resolved during the gap between studies. The source would be both the Prior Study Adverse Events CRF and the (020) Adverse Event CRF.
- 2. Pre-existing AEs: AEs that were ongoing on Day 1 of dosing in 020 source is the Prior Study Adverse Events CRF. The source would be both the Prior Study Adverse Events CRF and the (020) Adverse Event CRF.


- 3. Study-emergent AEs: AEs that started on or after Day 1 of dosing in 020, excluding post-treatment AEs (defined in #5 below). The source would be the (020) Adverse Event CRF.
- 4. All AEs: Whether pre-existing or study-emergent (merge of AEs that were ongoing on Day 1 of dosing) excluding post-treatment AEs. Sources are the Prior Study Adverse Events CRF and the (020) Adverse Event CRF) (note, this is a merge of #2 and 3 above *only*).
- 5. Post-treatment AEs: The study-emergent AEs (3# above) that have an onset more than 14 days after the last dose of study drug or that worsen in intensity or treatment attribution following discontinuation more than 14 days after the last dose of study drug.

The tabular summaries will be provided for AEs, with the number and percentage of subjects reporting each type of event. If a subject reports the same preferred term more than once, it is counted only once within that category. Further, for a given tabulation, the preferred term will only be counted once at its worst severity and strongest relationship to treatment.

After missing date imputation, if the end date and start date of two or more AEs with the same Preferred Term are less than or equal to two days apart, then the AE will be considered to be the same event and will be counted as one event. If the end date is missing for the first AE or the start date for the sequential AE is before the end date for the first AE, then the AEs will be considered one event and will be counted once. In every other case, the events will be counted separately.

The following summaries will be provided for AE categories 2-4 above:

- An overall summary of AEs summarizing the number and percent of subjects, and the number of unique AEs, in the following categories: any AE, severe AE, AE related to study drug, serious AE, related serious AE (serious adverse reaction or SAR), AE with outcome of death, adverse events of special interest (AESIs), AE leading to dose reduction, AE leading to dose interruption, AE leading to withdrawal of study drug, and AE leading to dose reduction, dose interruption, or withdrawal of study drug.
- Number of subjects who experienced AEs and total number of unique AEs by MedDRA SOC and PT.
- Number of subjects who experienced AEs by MedDRA SOC, PT, and worst severity.


- Number of subjects who experienced AEs by MedDRA SOC, PT, and strongest relationship<sup>2</sup> to study drug (Related/Not Related). Events reported as "Possibly Related," or "Related" will be included in the Related category. Events reported as "Unlikely Related" or "Not Related" will be included in the Not Related category. At each level of subject summarization a subject is classified according to the strongest relationship, as determined by the investigator, if the subject reported one or more events. AEs with a missing relationship will be considered related for this summary.
- Number of subjects who experienced serious AEs (SAEs) and total number of unique serious AEs by MedDRA SOC and PT (and subsets for fatal and nonfatal SAEs as well as related SAEs (SARs), as described above).
- Number of subjects who experienced severe AEs and total number of unique severe AEs by MedDRA SOC and PT. AEs with missing severity will be considered severe for inclusion in this summary.
- Number of subjects who experienced AEs leading to change in dose and total number of unique AEs leading to change in dose (dose reduction, dose interruption, and study drug withdrawal, separately and combined) by MedDRA SOC and PT.
- Number of subjects who experienced unique protocol-specified AESIs and total number of unique protocol-specified AESIs by MedDRA SOC and PT.

The above summaries of AEs will also be presented for non-AChEI (acetylcholinesterase inhibitor)/Memantine users. Selected summaries of AEs will also be presented by diagnosis and prior study treatment. Depending on controlled study results, analyses of selected TauRx AE groupings may be undertaken.

A tabular summary of post-treatment adverse events (#5 above) by MedDRA SOC and PT will be provided.

The AE listing will include Prior AEs, All AEs, and Post-treatment AEs (#1, 4, and 5 above). Prior AEs, Pre-existing AEs and Post-treatment AEs will be flagged.

In addition, listings will also be provided for study-emergent or post-treatment SAEs (including subsets for fatal and non-fatal SAEs), study-emergent AEs leading to dose reduction, interruption or study drug withdrawal, and study-emergent or post-treatment AESIs. Post-treatment AEs will be flagged.


<sup>&</sup>lt;sup>2</sup> Relationship is determined by the Investigator

#### 7.2 Clinical Laboratory Evaluation

Central laboratory data are transferred electronically by Covance. The Data Transfer Specification document provides a detailed description of the content and format of the laboratory datasets. Both conventional and SI units are provided and will be summarized in separate tables and listings. The eGFR values will be calculated and included in the tables and listings for clinical chemistry parameters.

Results from local laboratories are entered into the CRF by the site; these will not be included in summary tabulations but will be included in the data listings together with the corresponding normal ranges. Values for local laboratory parameters will be converted to the corresponding alternative units, either conventional or SI, depending on how reported.

For the summary tabulations of laboratory results, Baseline is defined as the last non-missing value prior to first dose of study drug in 020. Laboratory tests obtained on the date of the first dose will be assigned to pre-treatment. For each analyte, Baseline values will be restricted to those subjects in the safety population for whom there is at least one post-Baseline value (either overall or for the corresponding target visit). Any lab result 14 or more days after the last dose will be considered post-treatment.

Visit windows are used when results are presented by target visit (see <u>Appendix A</u>). For each analyte, if a subject has multiple values within a visit window, the "worst" value as defined in <u>Appendix D</u> will be used for that visit window summary.

Results of all continuous laboratory parameters will be summarized using descriptive statistics at baseline and at each post-baseline target visit; the last available on-treatment value and post-treatment results will also be summarized. The baseline data may come from the prior study, if not repeated in 020. For each subsequent target visit, changes from baseline will also be summarized by the number and percentage of subjects and the mean, median, SD, minimum, and maximum values for continuous laboratory parameters. These will also be prepared for subjects categorized by diagnosis and AChEI/Memantine use.

Box and whisker plots will be presented for selected parameters including hemoglobin, reticulocytes (%), neutrophils, and liver function tests. Other parameters may be identified during data review.

Thresholds for potentially clinically significant (PCS) laboratory abnormalities are defined in <u>Appendix B</u> for selected parameters. When there are thresholds provided for low and high values, they will be handled separately. Summaries will include the number and percent of subjects with treatment-emergent PCS values, restricted to those subjects in

whom the values represent a post-baseline worsening (PCST); the number meeting criteria at baseline will also be summarized. A PCST is defined as any PCS event that happened at any post-baseline visit and has a value more out of range than the value for a particular test at baseline (see <u>Appendix D</u> for directionality of worsening).

Listings of laboratory parameter results will be presented. Listings will include all laboratory flags provided by the central laboratory in the data transfer as well as flags for those that meet criteria for being PCS (whether or not a study-emergent worsening); additionally, results evaluated by the investigator as abnormal/clinically significant will be flagged in the listing. A separate listing for samples that could not be analyzed and the corresponding comments will be provided.

Separate listings for each hematology and chemistry parameter will include only subjects with treatment-emergent PCS values and, for these subjects, all laboratory results for the parameter meeting PCS criteria and related parameters (e.g., ALT, AST, bilirubin, neutrophils, WBC, etc.) will be provided.

#### 7.3 Vital Signs

Vital sign measurements will be summarized descriptively by target visit using the visit windows defined in <u>Appendix A</u> and the last available on-treatment visit; baseline will be the last non-missing value prior to the first dose of study drug. The baseline data may come from the prior study, if not repeated in 020. Vital signs include seated blood pressure and pulse, temperature, respiratory rate, and body weight. Change from baseline will also be calculated and summarized. If a subject has multiple values within a visit window, the "worst" value as defined in <u>Appendix D</u> will be used for that visit window summary.

Potentially clinically significant vital sign changes are defined for selected parameters in Appendix C. When there are thresholds provided for low and high values, they will be handled separately. Summaries will include the number and percent of subjects with treatment-emergent PCS values, restricted to those subjects in whom the values represent a post-baseline worsening (PCST). A PCST is defined as any PCS event that happened at any post-baseline visit and has a value more out of range than the value for a particular parameter at baseline (see Appendix D for directionality of worsening).

Listings of vital sign measurements including height at Screening will be presented. Listings will flag results that meet criteria as being PCS (whether or not a treatment emergent worsening).

Separate listings for each vital sign parameter will include only subjects with study-emergent PCS values and, for these subjects, all corresponding vital sign results will be provided.

#### 7.4 Physical and Neurological Examinations and Serotonin Syndrome (Toxicity)

Targeted examinations were optional prior to protocol version 3.0. With version 3.0 or higher, they are to be performed at every visit (or upon early termination), including the 4-week post-treatment follow-up visit if applicable.

The targeted examinations will be focused on, but not limited to, evaluating subjects for potential serotonin toxicity and also as clinically indicated. At a minimum, they are to include assessments for serotonin toxicity, evaluation of deep tendon reflexes, clonus, and muscle rigidity; size and reactivity of pupils; dryness of oral mucosa; intensity of bowel sounds; skin color; and presence or absence of diaphoresis.

Summaries will present the number and percentage of subjects with normal and abnormal observations by body system/parameter evaluated. By-subject listings will detail any abnormalities.

Ratings for signs and symptoms of serotonin syndrome (toxicity), inclusive of the MMSE, were introduced in protocol version 3.0 and will be performed at each visit. A by-subject listing of all responses will be prepared. A separate listing will be provided for the Mini-Mental State Examination (MMSE) scores.

#### 7.5 Electrocardiography

A 12-lead ECG (triplicate recording) was introduced in protocol version 3.0. Measurements are taken approximately every 6 months thereafter (or upon early termination), including the 4-week post-treatment follow-up visit if applicable. Recordings will be evaluated by a centralized ECG reading facility. Interval data (including QT and corrected QT intervals), ventricular rate, and overall interpretation are to be reported for every ECG. The interval data and ventricular rate are to be noted in the CRF as averages of the three readings (with the exception of values that are not evaluable and reported as zero, in which case the average will exclude this zero value and note in the CRF the average of values > 0).

ECG interval and ventricular rate data will be summarized using descriptive statistics. Windows for each target visit will be used (<u>Appendix A</u>). Parameters to be analyzed include heart rate (HR) and PR, QRS, QT, and corrected QT (using Fridericia's and Bazett's corrections), and RR intervals. Counts and percent of subjects in each result

category will be tabulated. Overall interpretations of abnormalities will also be tabulated, with subjects categorized by whether or not they have study-emergent abnormalities.

Subjects are also to be categorized and enumerated on the basis of QTcB/F interval as follows:

- Absolute measurements (in categories of > 450 to  $\le 480$ , > 480 to  $\le 500$ , > 500 msec)
- Change from first 020 measurement (in categories of > 30 to  $\le 60$ , > 60 to < 90,  $\ge 90$  msec)

All HR, interval data, and interpretations will be listed. Any local ECG results (optional prior to version 3.0 of the protocol) will be listed separately.

#### 8. OTHER ASSESSMENTS

#### **8.1 MMSE**

For MMSE in subjects with AD, change from baseline for pooled treatment allocation will be analyzed using a restricted maximum likelihood based repeated measures linear mixed model. The model will include fixed effects for AChEI/Memantine use as randomized in the prior study (Yes and No), time since baseline in the prior study (continuous), AChEI/Memantine use as randomized in the prior study by time interaction and the prior study baseline MMSE, prior study (015 and 005) and region (The Americas and RoW). In addition, the baseline MMSE from the prior study will be included as a covariate An unstructured covariance model will be used. The Kenward and Roger method of calculating the denominator degrees of freedom will be used for the tests of fixed effects. Annualized LS means will be provided. Additionally, observed means according to the visit windowing in Appendix A will be provided.

If more than 20 bvFTD subjects have MMSE values in 020, the above analysis will be repeated for bvFTD subjects.

If more than 10 subjects with AD discontinue AChEI/Memantine in 020, then summary of MMSE at the visits prior to and the visits subsequent to discontinuation will be provided.

#### 8.2 EQ-5D-5L

The EQ-5D-5L is a standardized instrument developed by the EuroQol Group to describe and value health-related quality of life. The EQ-5D-5L will be performed at baseline and approximately every 6 months thereafter (or upon early termination). There will be two

applications of the self-reported EQ-5D-5L at each visit: one version will be completed by the subject and a second copy of this version will be completed by the caregiver.

The instrument comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated by the subject and caregiver on a 5-point scale as having "no problems" (a score of "1"), "slight problems" (a score of "2"), "moderate problems" (a score of "3"), "severe problems" (a score of "4"), and "extreme problems" (a score of "5") based on descriptive examples; the scores are not intended to be summed. Present overall state of health is also to be rated on a vertical visual analogue scale (approximately 20 cm in length) from 0 to 100 (the higher the number the better the quality of life). Each of the five dimensions as well as the overall state of health will be summarized descriptively by visit. Following the 24-Aug-2015 CRF migration, the original EQ-5D-5L eCRF was inactivated and the EQ-5D-5L Patient Rated and EQ-5D-5L Caregiver Rated eCRFs were activated. For subjects under version protocol version 1.1, only the EQ-5D-5L was applied to the subject, who should receive no help from the caregiver. For subjects under protocol version 2.1 or later versions, EQ-5D-5L is to be applied separately to both subject and caregiver. For the purposes of this summary, data obtained from the original EQ-5D-5L eCRF prior to the 24-Aug-2015 CRF migration and data obtained from the EQ-5D-5L Patient Rated eCRF after the 24-Aug-2015 CRF migration will be used.

The EQ-5D-5L health economic and economic modelling, and additional sensitivity analyses will be addressed in a separate external SAP.

#### 8.3 RUD Lite

The RUD Lite assesses both formal and informal resource use, making it possible to calculate costs from a societal perspective. The RUD Lite is administered as an interview with the caregiver. The following dimensions are captured on the subject's part: accommodation/long term care, respite care, hospital care, social service, home nursing care, and work status. In addition, the following aspects are covered from the caregiver perspective: caregiving time for the subject and work status.

Each component of caregiver time will be calculated as the hours of care on a typical day multiplied by days spent on providing these services and summarized descriptively by visit. Caregiver work status, whether the subject was admitted to a hospital, whether the subject received services in a hospital emergency room, whether the subject visited any health care professional, whether the subject received any nursing services as well as caregiver relationship with subject and the subject's living accommodations will also be summarized descriptively by visit.

The RUD Lite unit cost and economic modelling, and additional sensitivity analyses will be addressed in a separate external SAP.

#### 9. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

Any changes will be documented in the Clinical Study Report in Section 9.8.

# **APPENDICES**

# **Appendix A: Post-Dose Visit Windows**

Visit windows are defined in the following table. Unscheduled and early termination visits are included in the windowing algorithm.

| Target Visit | Visit Window | Scheduled Day |
|--------------|-------------------------------|---------------|
| | Time Interval (Study Day*) | |
| Baseline | < 2 | NA |
| Week 2 | 2 to 53 | 15 |
| Week 13 | 54 to 137 | 92 |
| Week 26 | 138 to 228 | 183 |
| Week 39 | 229 to 319 | 274 |
| Week 52 | 320 to 410 | 365 |
| Week 65 | 411 to 501 | 456 |
| Week 78 | 502 to 591 | 546 |
| Week 91 | 592 to 683 | 637 |
| Week 104 | > 683 | 729 |
| Follow-up | First post-treatment value at | |
| | least 14 days after last dose | |

Appendix B: Criteria for Determining Potentially Clinically Significant Values in Laboratory Test Results

| | Criteria | |
|---|---|---|
| Test | System International Units | <b>Conventional Units</b> |
| Hemoglobin | Female: $\leq 95$ g/L; Male: $\leq 115$ | Female: $\leq 9.5 \text{ g/dL}$ ; |
| | g/L | Male: $\leq 11.5 \text{ g/dL}$ |
| | Decrease of $\geq 20\%$ | |
| Hematocrit | Female: $\leq 0.32$ ; Male: $\leq 0.37$ | Female: $\leq 32\%$ ; |
| | 0 | Male: ≤ 37% |
| WBC count | $\leq 2.8 \times 10^9 / L$ | $\leq 2800/\mu L \text{ or } \geq 16000/\mu L$ |
| | $\geq 16 \times 10^9 / L$ | |
| Neutrophils | $\leq 1.0 \times 10^9 / L$ | $\leq 1000/\mu L$ |
| Eosinophils | $\geq 0.7 \times 10^9/L$ | $\geq 700/\mu L$ |
| Platelet count | $\leq 75 \times 10^9/L$ | $\leq 75 \times 10^3 / \mu L$ |
| | $\geq 700 \times 10^9 / L$ | $\geq 700 \times 10^3/\mu$ L |
| Sodium | <130 mmol/L | <130 mEq/L |
| | >150 mmol/L | >150 mEq/L |
| Potassium | < 3.0 mmol/L | < 3.0 mEq/L |
| | > 5.5 mmol/L | > 5.5 mEq/L |
| Calcium | < 1.75 mmol/L | < 7.00 mg/dL |
| | > 3.00 mmol/L | > 12.00 mg/dL |
| Glucose, | < 2.775 mmol/L | < 50 mg/dL |
| fasting/nonfasting/unk | >13.875 mmol/L | > 250 mg/dL |
| nown | | |
| Uric acid | Female: >475.8 μmol/L; Male: | Female: > 8 mg/dL; |
| | >594.8 µmol/L | Male: >10 mg/dL |
| Albumin | <25 g/L | <2.5 g/dL |
| Total bilirubin | $\geq$ 34.2 $\mu$ mol/L | $\geq 2 \text{ mg/dL}$ |
| ALT | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| AST | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| Alkaline phosphatase | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| Urea (nitrogen) | > 17.85 mmol/L | > 50 mg/dL |
| Creatinine | $\geq 177 \; \mu \text{mol/L}$ | $\geq$ 2 mg/dL |
| CK | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| GGT | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| LDH | $\geq$ 3 × ULN | $\geq$ 3 × ULN |
| Phosphorus | < 0.646 mmol/L | Low: <2.0 mg/dL |
| | > 1.777 mmol/L | High: >5.5 mg/dL |

ULN = Upper Limit of Normal

# **Appendix C: Criteria for Determining Potentially Clinically Significant Values in Vital Signs**

| Test | Criteria |
|---|---|
| Systolic Blood Pressure | Increase of ≥ 20 mmHg from baseline and ≥ 180 mmHg |
| (SBP) – Seated (mmHg) | ≤ 90 mmHg |
| | Decrease of ≥ 20 mmHg from baseline and ≤ 90 mmHg |
| Diastolic Blood Pressure | Increase of ≥ 15 mmHg from baseline and ≥ 105 mmHg |
| (DBP) – Seated (mmHg) | ≤50 mmHg |
| Pulse – Seated (beats/min) | Increase of ≥ 15 beats/min from baseline and > 120 beats/min |
| | Decrease of ≥ 15 beats/min from baseline and ≤ 50 beats/min |
| Temperature | Increase of ≥ 2.0°C from baseline and ≥ 38.0°C |
| | Decrease of ≥ 2.0°C from baseline and ≤ 36.0°C |
| Weight | Decrease of ≥ 7% from baseline |
| | Decrease of $\geq 10\%$ from baseline |
| | Increase of ≥ 7% from baseline |
| | Increase of $\geq 10\%$ from baseline |

# Appendix D: Rules for Determining "Worst" Value

# "Worst" Clinical Laboratory Value

| Rule | Parameters |
|---|---|
| Highest value | Hematology: eosinophils, basophils, monocytes, reticulocytes |
| | Serum chemistry: ALT, AST, ALK-P, creatinine, total bilirubin, urea (nitrogen), uric acid, LDH, creatine kinase, GGT |
| Lowest value | Hematology: neutrophils, RBC count, HCT, hemoglobin, platelets |
| | Serum chemistry: albumin, creatinine clearance total protein |
| Farthest from | Hematology: WBC count, lymphocytes, MCV, MCH, MCHC |
| normal range<br>midpoint | Serum chemistry: glucose (random), Na, K, phosphate, calcium, chloride |

# "Worst" Vital Sign and Weight Measurement

| Parameter | Criterion for "Worst" Vital Sign |
|--------------------------|-----------------------------------------|
| Systolic blood pressure | Value farthest from 125 mmHg |
| Diastolic blood pressure | Value farthest from 75 mmHg |
| Pulse | Value farthest from 75 beats per minute |
| Temperature | Highest |
| Respiratory Rate | Highest |
| Weight | Greatest weight loss from baseline |

# "Worst" ECG Measurement

| 11 0100 = 0 0 110000 = 0 0 1 | |
|------------------------------|----------------------------------------------|
| Parameter | Criterion for "Worst" ECG |
| PR | Highest |
| QT (QTcF and QTcB) | Highest |
| QRS | Value farthest from midpoint of normal range |
| Heart Rate | Value farthest from midpoint of normal range |
#### **Appendix E: Rules for Scoring the MMSE**

The MMSE score ranges from 0 to 30, and is defined as the sum of 11 items as listed in the following table.

| Item | Maximum<br>Score |
|---|---|
| Orientation – Time (including questions about year, season, month, week, date) | 5 |
| Orientation – Place (including questions about state, county, city/town, building and floor) | 5 |
| Memory – Registration (including registration word 1-3) | 3 |
| Attention and Concentration (including five "what is 100 taken away 7" questions) | 5 |
| Memory – Recall (including questions of "Recall Word" 1-3) | 3 |
| Language – Naming (including questions about pencil/pen and watch) | 2 |
| Language – Repetition ("Repeat what I say") | 1 |
| Language – Reading Comprehension ("Close your eyes") | 1 |
| Praxis – Ideational (Including questions of "Take in right hand" "Fold in Half" "Put on Floor"). | 3 |
| Language – Writing Spontaneous ("Please Write a Sentence") | 1 |
| Praxis – Coping Drawing ("Please copy this design") | 1 |
| Total | 30 |

## Appendix F: List of Tables, Figures and Listings

## **List of Tables**

| Table | |
|---|---|
| Number | Table Description |
| 14.1.1.1 | Subject Disposition (All Subjects) |
| 14.1.1.2 | Subject Disposition by Region (All Subjects) |
| 14.1.1.3 | Subject Disposition by Country and Site (All Subjects) |
| 14.1.1.4 | Subject Disposition – Non-AChEI/Memantine Users (All Subjects) |
| 14.1.2.1 | Study Discontinuation by Time Period (Safety Population) |
| 14.1.2.2 | Study Discontinuation by Time Period – Non-AChEI/Memantine |
| | Users (Safety Population) |
| 14.1.2.3 | Study Discontinuation by Time Period and by Region (Safety |
| | Population) |
| 14.1.3.1 | Protocol Deviations (Safety Population) |
| 14.1.3.2 | Protocol Deviations by Critical, Major and Minor Categories (Safety |
| | Population) |
| 14.1.4.1 | Demographic and Baseline Characteristics (Safety Population) |
| 14.1.4.2 | Demographic and Baseline Characteristics – Non-AChEI/Memantine |
| | Users (Safety Population) |
| 14.1.5.1 | Medical History (Safety Population) |
| 14.1.5.2 | Medical History – Non-AChEI/Memantine Users (Safety Population) |
| 14.1.6.1.1 | Concomitant Medications Ongoing On Day 1 of Dosing (Pre-existing |
| | Medications) (Safety Population) |
| 14.1.6.1.2 | Concomitant Medications Ongoing On Day 1 of Dosing (Pre-existing |
| | Medications) – Non-AChEI/Memantine Users (Safety Population) |
| 14.1.6.2.1 | Concomitant Medications that Started On or After Day 1 of Dosing |
| | (Study-emergent Medications) (Safety Population) |
| 14.1.6.2.2 | Concomitant Medications that Started On or After Day 1 of Dosing |
| | (Study-emergent Medications) – Non-AChEI/Memantine Users |
| | (Safety Population) |
| 14.1.6.3.1 | Concomitant Medications (Pre-existing and Study-emergent |
| | Medications) (Safety Population) |
| 14.1.6.3.2 | Concomitant Medications (Pre-existing and Study-emergent |
| | Medications) – Non-AChEI/Memantine Users (Safety Population) |
| 14.2.1.1 | MMSE (Safety Population: Subjects with AD) |

020 SAP 30MAR17.docxPage 38 of 169CONFIDENTIAL

| Table | |
|---|---|
| Number | Table Description |
| 14.2.1.2 | MMSE Annualized LS Means (Safety Population: Subjects with AD) |
| 14.2.2 | RUD Lite (Safety Population: Subjects with at Least One Post-Baseline |
| | RUD Lite Questionnaire) |
| 14.2.3 | EQ-5D-5L (Safety Population: Subjects with at Least One |
| | Post-Baseline EQ-5D-5L Questionnaire) |
| 14.3.1.1 | Study Drug Exposure and Compliance (Safety Population) |
| 14.3.1.2 | Study Drug Exposure and Compliance – Non-AChEI/Memantine |
| | Users (Safety Population) |
| 14.3.2.1.1.1 | Overall Summary of Adverse Events Ongoing On Day 1 of Dosing |
| | (Pre-existing Adverse Events) (Safety Population) |
| 14.3.2.1.1.2 | Overall Summary of Adverse Events Ongoing On Day 1 of Dosing |
| | (Pre-existing Adverse Events) – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.2.1.2.1 | Overall Summary of Adverse Events that Started On or After Day 1 of |
| | Dosing (Study-emergent Adverse Events) (Safety Population) |
| 14.3.2.1.2.2 | Overall Summary of Adverse Events that Started On or After Day 1 of |
| | Dosing (Study-emergent Adverse Events) – Non-AChEI/Memantine |
| | Users (Safety Population) |
| 14.3.2.1.3.1 | Overall Summary of Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) (Safety Population) |
| 14.3.2.1.3.2 | Overall Summary of Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) – Non-AChEI/Memantine Users |
| | (Safety Population) |
| 14.3.2.1.3.3 | Overall Summary of Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by Diagnosis and Prior Study |
| | Treatment (Safety Population) |
| 14.3.2.2.1.1 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse |
| | Events) by System Organ Class and Preferred Term (Safety |
| 1122212 | Population) |
| 14.3.2.2.1.2 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse |
| | Events) by System Organ Class and Preferred Term – |
| 142221 | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.2.2.1 | Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.2.2.2 | Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.2.3.1 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by System Organ Class and Preferred Term (Safety |
| | Population) |
| 14.3.2.2.3.2 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by System Organ Class and Preferred Term – |
| | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.2.3.3 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by Diagnosis, Prior Study Treatment, System Organ |
| | Class and Preferred Term (Safety Population) |
| 14.3.2.3.1.1 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse |
| | Events) by System Organ Class, Preferred Term and Severity (Safety |
| | Population) |
| 14.3.2.3.1.2 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse |
| | Events) by System Organ Class, Preferred Term and Severity – |
| | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.3.2.1 | Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class, Preferred |
| | Term and Severity (Safety Population) |
| 14.3.2.3.2.2 | Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class, Preferred |
| | Term and Severity – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.2.3.3.1 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by System Organ Class, Preferred Term and Severity |
| | (Safety Population) |
| 14.3.2.3.3.2 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by System Organ Class, Preferred Term and Severity |
| | - Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.4.1.1 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse |
| | Events) by System Organ Class, Preferred Term and Relationship |
| | (Safety Population) |
| 14.3.2.4.1.2 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse |
| | Events) by System Organ Class, Preferred Term and Relationship – |
| | Non-AChEI/Memantine Users (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.4.2.1 | Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class, Preferred |
| | Term and Relationship (Safety Population) |
| 14.3.2.4.2.2 | Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class, Preferred |
| | Term and Relationship – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.2.4.3.1 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by System Organ Class, Preferred Term and |
| | Relationship (Safety Population) |
| 14.3.2.4.3.2 | Adverse Events (Pre-existing Adverse Events and Study-emergent |
| | Adverse Events) by System Organ Class, Preferred Term and |
| | Relationship – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.5.1.1 | Serious Adverse Events Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term (Safety |
| | Population) |
| 14.3.2.5.1.2 | Serious Adverse Events Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term – |
| | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.5.2.1 | Serious Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.5.2.2 | Serious Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.5.3.1 | Serious Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.5.3.2 | Serious Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.6.1.1 | Fatal Adverse Events Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term (Safety |
| | Population) |
| 14.3.2.6.1.2 | Fatal Adverse Events Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term – |
| | Non-AChEI/Memantine Users (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.6.2.1 | Fatal Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.6.2.2 | Fatal Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.6.3.1 | Fatal Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.6.3.2 | Fatal Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.7.1.1 | Non-Fatal Serious Adverse Events Ongoing On Day 1 of Dosing |
| | (Pre-existing Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.7.1.2 | Non-Fatal Serious Adverse Events Ongoing On Day 1 of Dosing |
| | (Pre-existing Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.7.2.1 | Non-Fatal Serious Adverse Events that Started On or After Day 1 of |
| | Dosing (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.7.2.2 | Non-Fatal Serious Adverse Events that Started On or After Day 1 of |
| | Dosing (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.7.3.1 | Non-Fatal Serious Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.7.3.2 | Non-Fatal Serious Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.8.1.1 | Serious Adverse Reactions Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term (Safety |
| | Population) |
| 14.3.2.8.1.2 | Serious Adverse Reactions Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term – |
| | Non-AChEI/Memantine Users (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.8.2.1 | Serious Adverse Reactions that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.8.2.2 | Serious Adverse Reactions that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.8.3.1 | Serious Adverse Reactions (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.8.3.2 | Serious Adverse Reactions (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.9.1.1 | Severe Adverse Events Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term (Safety |
| | Population) |
| 14.3.2.9.1.2 | Severe Adverse Events Ongoing On Day 1 of Dosing (Pre-existing |
| | Adverse Events) by System Organ Class and Preferred Term – |
| | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.9.2.1 | Severe Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.9.2.2 | Severe Adverse Events that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.9.3.1 | Severe Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.9.3.2 | Severe Adverse Events (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.10.1.1 | Adverse Events Leading to Dose Reduction that were Ongoing On Day |
| | 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.10.1.2 | Adverse Events Leading to Dose Reduction that were Ongoing On Day |
| | 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.10.2.1 | Adverse Events Leading to Dose Reduction that Started On or After |
| | Day 1 of Dosing (Study-emergent Adverse Events) by System Organ |
| 11221022 | Class and Preferred Term (Safety Population) |
| 14.3.2.10.2.2 | Adverse Events Leading to Dose Reduction that Started On or After |
| | Day 1 of Dosing (Study-emergent Adverse Events) by System Organ |
| | Class and Preferred Term – Non-AChEI/Memantine Users (Safety |
| 14221021 | Population) |
| 14.3.2.10.3.1 | Adverse Events Leading to Dose Reduction (Pre-existing Adverse |
| | Events and Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term (Safety Population) |
| 14.3.2.10.3.2 | Adverse Events Leading to Dose Reduction (Pre-existing Adverse |
| | Events and Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.2.10.3.3 | Adverse Events Leading to Dose Reduction (Pre-existing Adverse |
| | Events and Study-emergent Adverse Events) by Diagnosis, Prior Study |
| | Treatment, System Organ Class and Preferred Term (Safety |
| | Population) |
| 14.3.2.11.1.1 | Adverse Events Leading to Dose Interruption that were Ongoing On |
| | Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class |
| | and Preferred Term (Safety Population) |
| 14.3.2.11.1.2 | Adverse Events Leading to Dose Interruption that were Ongoing On |
| | Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class |
| | and Preferred Term – Non-AChEI/Memantine Users (Safety |
| 14221121 | Population) |
| 14.3.2.11.2.1 | Adverse Events Leading to Dose Interruption that Started On or After |
| | Day 1 of Dosing (Study-emergent Adverse Events) by System Organ |
| 14221122 | Class and Preferred Term (Safety Population) |
| 14.3.2.11.2.2 | Adverse Events Leading to Dose Interruption that Started On or After |
| | Day 1 of Dosing (Study-emergent Adverse Events) by System Organ |
| | Class and Preferred Term – Non-AChEI/Memantine Users (Safety |
| 14221121 | Population) |
| 14.3.2.11.3.1 | Adverse Events Leading to Dose Interruption (Pre-existing Adverse |
| | Events and Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.11.3.2 | Adverse Events Leading to Dose Interruption (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.11.3.3 | Adverse Events Leading to Dose Interruption (Pre-existing Adverse Events and Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term (Safety Population) |
| 14.3.2.12.1.1 | Adverse Events Leading to Study Drug Withdrawal that were Ongoing<br>On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ<br>Class and Preferred Term (Safety Population) |
| 14.3.2.12.1.2 | Adverse Events Leading to Study Drug Withdrawal that were Ongoing<br>On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ<br>Class and Preferred Term – Non-AChEI/Memantine Users (Safety<br>Population) |
| 14.3.2.12.2.1 | Adverse Events Leading to Study Drug Withdrawal that Started On or<br>After Day 1 of Dosing (Study-emergent Adverse Events) by System<br>Organ Class and Preferred Term (Safety Population) |
| 14.3.2.12.2.2 | Adverse Events Leading to Study Drug Withdrawal that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.12.3.1 | Adverse Events Leading to Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) |
| 14.3.2.12.3.2 | Adverse Events Leading to Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.12.3.3 | Adverse Events Leading to Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term (Safety Population) |
| 14.3.2.13.1.1 | Adverse Events Leading to Dose Reduction, Dose Interruption or<br>Study Drug Withdrawal that were Ongoing On Day 1 of Dosing<br>(Pre-existing Adverse Events) by System Organ Class and Preferred<br>Term (Safety Population) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.13.1.2 | Adverse Events Leading to Dose Reduction, Dose Interruption or |
| | Study Drug Withdrawal that were Ongoing On Day 1 of Dosing |
| | (Pre-existing Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.13.2.1 | Adverse Events Leading to Dose Reduction, Dose Interruption or |
| | Study Drug Withdrawal that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term (Safety Population) |
| 14.3.2.13.2.2 | Adverse Events Leading to Dose Reduction, Dose Interruption or |
| | Study Drug Withdrawal that Started On or After Day 1 of Dosing |
| | (Study-emergent Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.13.3.1 | Adverse Events Leading to Dose Reduction, Dose Interruption or |
| | Study Drug Withdrawal (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.13.3.2 | Adverse Events Leading to Dose Reduction, Dose Interruption or |
| | Study Drug Withdrawal (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.13.3.3 | Adverse Events Leading to Dose Reduction, Dose Interruption or |
| | Study Drug Withdrawal (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, |
| 14221411 | System Organ Class and Preferred Term (Safety Population) |
| 14.3.2.14.1.1 | Adverse Events of Special Interest (AESI) Ongoing On Day 1 of |
| | Dosing (Pre-existing Adverse Events) by System Organ Class and |
| 14221412 | Preferred Term (Safety Population) |
| 14.3.2.14.1.2 | Adverse Events of Special Interest (AESI) Ongoing On Day 1 of |
| | Dosing (Pre-existing Adverse Events) by System Organ Class and |
| 14221421 | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.2.14.2.1 | Adverse Events of Special Interest (AESI) that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term (Safety Population) |
| 14.3.2.14.2.2 | Adverse Events of Special Interest (AESI) that Started On or After Day |
| 17.3.2.17.2.2 | 1 of Dosing (Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term – Non-AChEI/Memantine Users (Safety |
| | Population) |
| | 1 opulation) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.2.14.3.1 | Adverse Events of Special Interest (AESI) (Pre-existing Adverse |
| | Events and Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term (Safety Population) |
| 14.3.2.14.3.2 | Adverse Events of Special Interest (AESI) (Pre-existing Adverse |
| | Events and Study-emergent Adverse Events) by System Organ Class |
| | and Preferred Term – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.2.15.1 | Post-Treatment Adverse Events by System Organ Class and Preferred |
| | Term (Safety Population) |
| 14.3.2.15.2 | Post-Treatment Adverse Events by System Organ Class and Preferred |
| | Term – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.3.1.1.1 | Hematology Values and Changes from Baseline at All Visits – |
| | Conventional Units (Safety Population) |
| 14.3.3.1.1.2 | Hematology Values and Changes from Baseline at All Visits – |
| | Conventional Units – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.3.1.2.1 | Hematology Values and Changes from Baseline at All Visits – SI Units |
| | (Safety Population) |
| 14.3.3.1.2.2 | Hematology Values and Changes from Baseline at All Visits – SI Units |
| | - Non-AChEI/Memantine Users (Safety Population) |
| 14.3.3.2.1.1 | Serum Chemistry Values and Changes from Baseline at All Visits – |
| | Conventional Units (Safety Population) |
| 14.3.3.2.1.2 | Serum Chemistry Values and Changes from Baseline at All Visits – |
| | Conventional Units – Non-AChEI/Memantine Users (Safety |
| 142221 | Population) |
| 14.3.3.2.2.1 | Serum Chemistry Values and Changes from Baseline at All Visits – SI |
| 142222 | Units (Safety Population) |
| 14.3.3.2.2.2 | Serum Chemistry Values and Changes from Baseline at All Visits – SI |
| 142221 | Units – Non-AChEl/Memantine Users (Safety Population) |
| 14.3.3.3.1 | Incidence of Potentially Clinically Significant Hematology and Serum |
| 14.3.3.3.2 | Biochemistry Results (Safety Population) Incidence of Potentially Clinically Significant Hematology and Serum |
| 14.3.3.3.4 | Biochemistry Results – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.4.1.1.1 | Vital Signs (Safety Population) |
| 14.3.4.1.1.2 | Vital Signs – Non-AChEI/Memantine Users (Safety Population) |
| 14.3.4.1.2.1 | Weight Directional Changes (Safety Population) |
| 17.3.7.1.4.1 | Weight Directional Changes (Safety 1 optilation) |

| Table | |
|---|---|
| Number | Table Description |
| 14.3.4.1.2.2 | Weight Directional Changes – Non-AChEI/Memantine Users (Safety |
| | Population) |
| 14.3.4.1.3.1 | Incidence of Potentially Clinically Significant Vital Sign Results |
| | (Safety Population) |
| 14.3.4.1.3.2 | Incidence of Potentially Clinically Significant Vital Sign Results – |
| | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.4.2 | Physical Examination by Visit (Safety Population) |
| 14.3.4.3 | Neurological Examination by Visit (Safety Population) |
| 14.3.4.4.1 | Serotonin Toxicity (Syndrome) Ratings by Visit (Safety Population) |
| 14.3.4.4.2 | Serotonin Toxicity (Syndrome) Ratings by Visit – |
| | Non-AChEI/Memantine Users (Safety Population) |
| 14.3.4.5.1 | Central ECG Data by Visit (Safety Population) |
| 14.3.4.5.2 | Central ECG Data – Change from Baseline in Investigator's Overall |
| | Interpretation of Clinical Significance by Visit (Safety Population) |
| 14.3.4.5.3 | Central ECG Data – QTc Abnormalities (Safety Population) |

# **List of Figures**

| Figure | |
|---|---|
| Number | Figure Description |
| 14.2.4.1 | Observed Mean MMSE by Visit (Safety Population) |
| Annualized Mean Change from Baseline in MMSE (Safety | |
| 14.2.4.2 | Population) |
| 14.3.5.1.1 | Box Plots of Hemoglobin by Visit – Conventional Units (Safety |
| | Population) |
| 14.3.5.1.2 | Box Plots of Hemoglobin Change from Baseline by Visit – |
| | Conventional Units (Safety Population) |
| 14.3.5.1.3 | Box Plots of Hemoglobin by Visit – SI Units (Safety Population) |
| 14.3.5.1.4 | Box Plots of Hemoglobin Change from Baseline by Visit – SI Units |
| | (Safety Population) |
| 14.3.5.2.1 | Box Plots of Reticulocytes by Visit – Conventional Units (Safety |
| | Population) |
| 14.3.5.2.2 | Box Plots of Reticulocytes Change from Baseline by Visit – |
| | Conventional Units (Safety Population) |
| 14.3.5.2.3 | Box Plots of Reticulocytes by Visit – SI Units (Safety Population) |
| 14.3.5.2.4 | Box Plots of Reticulocytes Change from Baseline by Visit – SI Units |
| | (Safety Population) |
| 14.3.5.3.1 | Box Plots of Neutrophils by Visit (Safety Population) |
| 14.3.5.3.2 | Box Plots of Neutrophils Change from Baseline by Visit (Safety |
| | Population) |
| 14.3.5.4.1 | Box Plots of Albumin by Visit – Conventional Units (Safety |
| | Population) |
| 14.3.5.4.2 | Box Plots of Albumin Change from Baseline by Visit – Conventional |
| | Units (Safety Population) |
| 14.3.5.4.3 | Box Plots of Albumin by Visit – SI Units (Safety Population) |
| 14.3.3.4.4 | Box Plots of Albumin Change from Baseline by Visit – SI Units |
| | (Safety Population) |
| 14.3.5.5.1 | Box Plots of ALT by Visit (Safety Population) |
| 14.3.5.5.2 | Box Plots of ALT Change from Baseline by Visit (Safety Population) |
| 14.3.5.6.1 | Box Plots of AST by Visit (Safety Population) |
| 14.3.5.6.2 | Box Plots of AST Change from Baseline by Visit (Safety Population) |
| 14.3.5.7.1 | Box Plots of Alkaline Phosphatase by Visit (Safety Population) |
| 14.3.5.7.2 | Box Plots of Alkaline Phosphatase Change from Baseline by Visit |
| | (Safety Population) |

| Figure | |
|---|---|
| Number | Figure Description |
| 14.3.5.8.1 | Box Plots of Total Bilirubin by Visit – Conventional Units (Safety |
| | Population) |
| 14.3.5.8.2 | Box Plots of Total Bilirubin Change from Baseline by Visit – |
| | Conventional Units (Safety Population) |
| 14.3.5.8.3 | Box Plots of Total Bilirubin by Visit – SI Units (Safety Population) |
| 14.3.5.8.4 | Box Plots of Total Bilirubin Change from Baseline by Visit – SI Units |
| | (Safety Population) |
| 14.3.5.9.1 | Box Plots of Direct Bilirubin by Visit – Conventional Units (Safety |
| | Population) |
| 14.3.5.9.2 | Box Plots of Direct Bilirubin Change from Baseline by Visit – |
| | Conventional Units (Safety Population) |
| 14.3.5.9.3 | Box Plots of Direct Bilirubin by Visit – SI Units (Safety Population) |
| 14.3.5.9.4 | Box Plots of Direct Bilirubin Change from Baseline by Visit – SI |
| | Units (Safety Population) |

# **List of Listings**

| Listing | |
|---|---|
| Number | Listing Description |
| 16.2.1.1.1 | Subjects Who Entered the Study (All Enrolled) |
| 16.2.1.1.2 | Informed Consent (All Enrolled) |
| 16.2.1.1.3 | Reconsent for Additional 12-Month Treatment Extension (All Enrolled) |
| 16.2.1.2 | Subject Disposition (All Enrolled) |
| 16.2.1.3 | Subject Visit Dates (All Enrolled) |
| 16.2.2.1 | Protocol Deviations (Safety Population) |
| 16.2.2.2 | Withdrawal of Consent (Safety Population) |
| 16.2.2.3 | Inclusion/Exclusion Criteria (Safety Population) |
| 16.2.4.1 | Demographics and Baseline Characteristics (Safety Population) |
| 16.2.4.2 | Medical History at Study Entry (Safety Population) |
| 16.2.4.3.1 | Prior Medications (Safety Population) |
| 16.2.4.3.2 | Concomitant Medications (Safety Population) |
| 16.2.4.4 | Procedures and Therapies (Safety Population) |
| 16.2.5.1 | Drug Accountability and Compliance (Safety Population) |
| 16.2.5.2 | By-Subject Summary of Overall Exposure (Safety Population) |
| 16.2.5.3 | Chronological Study Drug Administration Including Dose Interruption |
| | and Adjustment (Safety Population) |
| 16.2.6.1 | RUD Lite (Safety Population) |
| 16.2.6.2.1 | EQ-5D-5L (Safety Population) |
| 16.2.6.2.2 | EQ-5D-5L, Patient Rated (Safety Population) |
| 16.2.6.2.3 | EQ-5D-5L, Caregiver Rated (Safety Population) |
| 16.2.7.1 | Adverse Events (Safety Population) |
| 16.2.7.2.1 | Serious Adverse Events (Safety Population) |
| 16.2.7.2.2 | Fatal Adverse Events (Safety Population) |
| 16.2.7.2.3 | Non-Fatal Serious Adverse Events (Safety Population) |
| 16.2.7.2.4 | Serious Adverse Events (Additional Information About the SAE |
| | Collected on the AE CRF) |
| 16.2.7.2.5 | Serious Adverse Events (Collected on the SAE CRF) |
| 16.2.7.3.1 | Adverse Events Leading to Dose Reduction, Interruption or Study Drug |
| | Withdrawal (Safety Population) |
| 16.2.7.3.2 | All AEs for Subjects with Adverse Events Leading to Dose Reduction, |
| | Interruption or Study Drug Withdrawal (Safety Population) |
| 16.2.7.4 | Adverse Events of Special Interest (Safety Population) |
| 16.2.8.1.1 | Central Laboratory Normal Ranges (Safety Population) |

| Listing | |
|---|---|
| Number | Listing Description |
| 16.2.8.1.2 | Central Laboratory – Comments on Samples Not Analyzed (Safety |
| | Population) |
| 16.2.8.2.1 | Central Lab - Hematology – Conventional Units (Safety Population) |
| 16.2.8.2.2 | Central Lab - Hematology – SI Units (Safety Population) |
| 16.2.8.2.3 | Local Lab - Hematology – Conventional Units (Safety Population) |
| 16.2.8.2.4 | Local Lab - Hematology – SI Units (Safety Population) |
| 16.2.8.3.1 | Central Lab - Serum Chemistry – Conventional Units (Safety Population) |
| 16.2.8.3.2 | Central Lab - Serum Chemistry – SI Units (Safety Population) |
| 16.2.8.3.3 | Local Lab - Serum Chemistry – Conventional Units (Safety Population) |
| 16.2.8.3.4 | Local Lab - Serum Chemistry – SI Units (Safety Population) |
| 16.2.8.4.1 | Local Lab - Urinalysis – Conventional Units (Safety Population) |
| 16.2.8.4.2 | Local Lab - Urinalysis – SI Units (Safety Population) |
| 16.2.8.5.1 | Hematology Results of Potential Clinical Significance – Conventional |
| | Units (Safety Population) |
| 16.2.8.5.2 | Hematology Results of Potential Clinical Significance – SI Units (Safety |
| | Population) |
| 16.2.8.5.3 | Hematology Results of Potential Clinical Significance – Includes Only |
| | Hgb and Hct Reticulocy (Safety Population) |
| 16.2.8.5.4 | Hematology Results of Potential Clinical Significance – WBCs and |
| | Neutrophils (Safety Population) |
| 16.2.8.5.5 | Hematology Results of Potential Clinical Significance – Eosinophils |
| | (Safety Population) |
| 16.2.8.5.6 | Hematology Results of Potential Clinical Significance – Platelets (Safety |
| | Population) |
| 16.2.8.6.1 | Serum Chemistry Results of Potential Clinical Significance – |
| 162062 | Conventional Units (Safety Population) |
| 16.2.8.6.2 | Serum Chemistry Results of Potential Clinical Significance – SI Units |
| 162962 | (Safety Population) |
| 16.2.8.6.3 | Serum Chemistry Results of Potential Clinical Significance – Urea |
| 162964 | (Nitrogen) or Creatinine (Safety Population) |
| 16.2.8.6.4 | Serum Chemistry Results of Potential Clinical Significance – ALT, AST, |
| 16 2 0 1 | GGT, Bilirubin or Alkaline Phosphatase (Safety Population) |
| 16.2.9.1 | Vital Signs (Safety Population) Vital Sign Results of Potential Clinical Significance (Safety Population) |
| 16.2.9.2.1<br>16.2.9.2.2 | Subjects with Potentially Clinically Significant Vital Sign Results (Safety |
| 10.2.7.2.2 | Population) |
| 16.2.9.2.3 | Respiratory Rate (Safety Population) |
| 10.2.7.2.3 | Respiratory Rate (Surety 1 Sparation) |

| Listing | |
|------------|----------------------------------------------------------|
| Number | Listing Description |
| 16.2.9.3 | Pregnancy (Safety Population) |
| 16.2.9.4 | Physical Examination (Safety Population) |
| 16.2.9.5 | Neurological Examination (Safety Population) |
| 16.2.9.6 | Serotonin Toxicity Assessment (Safety Population) |
| 16.2.9.7 | Mini-Mental State Examination (MMSE) (Safety Population) |
| 16.2.9.8.1 | Central Electrocardiogram (Safety Population) |
| 16.2.9.8.2 | Local Electrocardiogram (Safety Population) |

**Appendix G: Table Layouts** 


Table 14.1.1.1 Subject Disposition All Subjects

| | AD | bvFTD | All Subjects |
|---|---|---|---|
| Subjects Enrolled | n | n | n |
| Safety Population [1] | n (%) | n (%) | n (%) |
| Completed<br>Discontinued | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| All Reasons for Study Discontinuation <sup>[2]</sup><br>Reason 1<br>Reason 2 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| Primary Reason for Study Discontinuation <sup>[2]</sup> Reason 1 Reason 2 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |

<sup>[1]</sup>All enrolled subjects who take at least one dose of study drug.

Programming Note: Repeat table for Table 14.1.1.4 Subject Disposition - Non-AChEI/Memantine Users (All Subjects)

<sup>[2]</sup> Subjects may be counted for more than one reason for study discontinuation but are counted only once for primary reason for discontinuation. Note: The following xx subjects vvv, www, xxx, yyy, zzz were enrolled but not dosed. (programming note: List the subject IDs)

**Table 14.1.1.2 Subject Disposition by Region** All Subjects

| | AD | bvFTD | All Subjects |
|---|---|---|---|
| Subjects Enrolled | n | n | n |
| Safety Population [1] | n (%) | n (%) | n (%) |
| Completed Discontinued | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| All Reasons for Study Discontinuation [2] | | | |
| Reason 1 | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) |
| Primary Reason for Study Discontinuation <sup>[2]</sup> | | | |
| Reason 1 | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) |
| Reason 1 | \ / | ( ) | ( / |

<sup>[1]</sup> All enrolled subjects who take at least one dose of study drug.
[2] Subjects may be counted for more than one reason for study discontinuation but are counted only once for primary reason for discontinuation.

Note: The following xx subjects vvv, www, xxx, yyy, zzz were enrolled but not dosed. (programming note: List the subject IDs)

**Table 14.1.1.3** Subject Disposition by Country and Site All Subjects

| Country | Site | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| Country 1 | All Sites Subjects Enrolled | n | n | n |
| | Safety Population [1] | n (%) | n (%) | n (%) |
| | Completed | n (%) | n (%) | n (%) |
| | Discontinued | n (%) | n (%) | n (%) |
| | All Reasons for Study Discontinuation [2] | | | |
| | Reason 1 | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) |
| | Primary Reason for Study Discontinuation [2] | | | |
| | Reason 1 | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) |
| | • • • | | | |
| | Site 1 | | | |
| | ••• | | | |

Programmer note: Start each site on a new page. Group sites within country within region.

<sup>[1]</sup> All enrolled subjects who take at least one dose of study drug.
[2] Subjects may be counted for more than one reason for study discontinuation but are counted only once for primary reason for discontinuation. Note: The following xx subjects vvv, www, xxx, yyy, zzz were enrolled but not dosed. (programming note: List the subject IDs)

Table 14.1.2.1 Study Discontinuation by Time Period Safety Population

| | AD<br>(N= ) | bvFTD | All Subjects |
|-----------------------|-------------|-------|--------------|
| | (N- ) | (N= ) | (N= ) |
| Study Discontinuation | n (%) | n (%) | n (%) |
| Study Discontinuation | n (%) | n (%) | n (%) |
| on Day 1 | | | |
| Reason 1 | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) |
| Study Discontinuation | n (%) | n (%) | n (%) |
| During Days 2- | - (. 5) | () | (, , |
| Reason 1 | n (%) | n (%) | n (%) |
| Reason 2 | n (%) | n (%) | n (%) |
| | . , | . , | |

Repeat for other period categories

. . .

Note: Percentages are based on the number of subjects in the Safety Population.

Programming Note: Repeat table for Table 14.1.2.2 Study Discontinuation by Time Period - Non-AChEI/Memantine Users (Safety Population)

Table 14.1.2.3
Study Discontinuation by Time Period and by Region
Safety Population

| Country | | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects (N= ) |
|---|---|---|---|---|
| Country 1 | Study Discontinuation | n (%) | n (%) | n (%) |
| | Study Discontinuation on Day 1 | n (%) | n (%) | n (%) |
| | Reason 1 | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) |
| | Study Discontinuation<br>During Days 2- | n (%) | n (%) | n (%) |
| | Reason 1 | n (%) | n (%) | n (%) |
| | Reason 2 | n (%) | n (%) | n (%) |
| | Repeat for other period categories | | | |

Note: Percentages are based on the number of subjects in the Safety Population.

TauRx Therapeutics Ltd TRx-237-020

**Table 14.1.3.1 Protocol Deviations Safety Population** 

| | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects (N= ) |
|--------------------------|-------------|----------------|--------------------|
| All Deviations Types | n (%) | n (%) | n (%) |
| Informed consent | n (%) | n (%) | n (%) |
| Safety | n (%) | n (%) | n (%) |
| IP / Treatment Deviation | n (%) | n (%) | n (%) |
| Other Deviations | n (%) | n (%) | n (%) |

Note: IP = investigational product

path\t\_program.sas date time

Table 14.1.3.2
Protocol Deviations by Critical, Major and Minor Categories
Safety Population

| | AD | bvFTD | All Subjects |
|--------------------------|-------|-------|--------------|
| | (N= ) | (N= ) | (N= ) |
| Critical Deviation | n (%) | n (%) | n (%) |
| Informed consent | n (%) | n (%) | n (%) |
| Safety | n (%) | n (%) | n (%) |
| IP / Treatment Deviation | n (%) | n (%) | n (%) |
| Other Deviations | n (%) | n (%) | n (%) |
| Major Deviation | n (%) | n (%) | n (%) |
| Informed consent | n (%) | n (%) | n (%) |
| ••• | n (%) | n (%) | n (%) |
| Minor Deviation | n (%) | n (%) | n (%) |
| Informed consent | n (%) | n (%) | n (%) |
| | n (%) | n (%) | n (%) |

Note: IP = investigational product

path\t\_program.sas date time

Table 14.1.4.1 Demographic and Baseline Characteristics Safety Population

| | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects (N= ) |
|---|---|---|---|
| | (2. | (2.1 | (11) |
| Age at Informed Consent to Prior Study (years) | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| < 75 years | n (%) | n (%) | n (%) |
| ≥75 years | n (%) | n (%) | n (%) |
| Gender | | | |
| Male | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) |
| Ethnicity | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) |
| Race | | | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) |
| Black or African American | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Multiple Races Checked | n (%) | n (%) | n (%) |
| Geographic Region | | | |
| The Americas | n (%) | n (%) | n (%) |
| Europe | n (%) | n (%) | n (%) |
| Rest of World | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Table 14.1.4.1 Demographic and Baseline Characteristics Safety Population

| | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects<br>(N= ) |
|---|---|---|---|
| Height (cm) | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Weight (kg) | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| BMI (kg/m²) | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| Subject's Living Accommodation | | | |
| Own Home (owner occupied or rented) | n (%) | n (%) | n (%) |
| Intermediate Forms of Accommodation (not dementia-specific) | n (%) | n (%) | n (%) |
| Dementia-specific Residential Accommodation | n (%) | n (%) | n (%) |
| Long-term Institutional Care | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Not Available | n (%) | n (%) | n (%) |
| Who Does the Subject Live With? | | | |
| Alone | n (%) | n (%) | n (%) |
| Spouse | n (%) | n (%) | n (%) |
| Sibling | n (%) | n (%) | n (%) |
| Child | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) |
| Not Available | n (%) | n (%) | n (%) |

path\t program.sas date time

Programming Note: Repeat table for Table 14.1.4.2 Demographic and Baseline Characteristics - Non-AChEI/Memantine Users (Safety Population)

Table 14.1.5.1 Medical History Safety Population

MedDRA System Organ Class High Level Term

| High Level Term<br>Preferred Term | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects<br>(N= ) |
|---|---|---|---|
| 5001 | n (0/) | n (0/) | n (0/) |
| SOC1 | n (%) | n (%) | n (%) |
| High Level Term 1 | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) |
| Etc | n (%) | n (%) | n (%) |
| High Level Term 2 | n (%) | n (%) | n (%) |
| SOC1 | n (%) | n (%) | n (%) |
| etc. | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Programmer note: Sort table based on SOC order alphabetically

Programming Note: Repeat table for Table 14.1.5.2 Medical History - Non-AChEI/Memantine Users (Safety Population)

Table 14.1.6.1.1 Concomitant Medications Ongoing On Day 1 of Dosing (Pre-existing Medications) **Safety Population** 

| ATC Class (Level 1) / | | | |
|---|---|---|---|
| ATC Class (Level 3)/ | AD | bvFTD | All Subjects |
| Generic Drug Name | (N= ) | (N= ) | (N= ) |
| Subjects Receiving Concomitant <sup>[1]</sup> Medications | n (%) | n (%) | n (%) |
| ATC Class (Level 1) 1 | n (%) | n (%) | n (%) |
| ATC Class (Level 3) 1 | n (%) | n (%) | n (%) |
| Generic Drug Name 1 | n (%) | n (%) | n (%) |
| Generic Drug Name 2 | n (%) | n (%) | n (%) |
| • | | | |
| ATC Class (Level 3) 2 | n (%) | n (%) | n (%) |
| Generic Drug Name 1 | n (%) | n (%) | n (%) |
| Generic Drug Name 2 | n (%) | n (%) | n (%) |
| ATC Class (Level 1) 2 | n (%) | n (%) | n (%) |
| ATC Class (Level 3) 1 | n (%) | n (%) | n (%) |
| Generic Drug Name 1 | n (%) | n (%) | n (%) |
| Generic Drug Name 2 | n (%) | n (%) | n (%) |

Note: At each level of summation (overall, ATC classes, generic drug name), subjects reporting more than one medication are counted only once. Each summary is ordered alphabetically by ATC class and generic drug name within each ATC class.

path\t program.sas date time

Programming Note: Repeat table for the tables listed below

| Table 14.1.6.1.2 | Concomitant Medications Ongoing On Day 1 of Dosing (Pre-existing Medications) – Non-AChEI/Memantine Users (Safety |
|---|---|
| | Population) |
| Table 14.1.6.2.1 | Concomitant Medications that Started On or After Day 1 of Dosing (Study-emergent Medications) (Safety Population) |
| Table 14.1.6.2.2 | Concomitant Medications that Started On or After Day 1 of Dosing (Study-emergent Medications) - Non-AChEI/Memantine Users |
| | (Safety Population) |
| Table 14.1.6.3.1 | Concomitant Medications (Pre-existing and Study-emergent Medications) (Safety Population) |
| Table 14.1.6.3.2 | Concomitant Medications (Pre-existing and Study-emergent Medications) – Non-AChEI/Memantine Users (Safety Population) |

<sup>[1]</sup> Pre-existing concomitant medications are those medications that were ongoing on Day 1 of dosing.

Table 14.2.1.1 MMSE Safety Population

| Median Min, Max Week 26 n Mean (SD) Median Min, Max Change from Baseline to Week 26 n | | AD |
|---|---|---|
| n Mean (SD) Median Min, Max Week 26 n Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | Time Point | (N= ) |
| Mean (SD) Median Min, Max Week 26 n Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | Baseline [1] | |
| Median Min, Max Week 26 n Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | n | n |
| Median Min, Max Week 26 n Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | Mean (SD) | xx.x (xx.xx) |
| Week 26 n Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | | XX.X |
| n Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | Min, Max | xx, xx |
| Mean (SD) Median Min, Max Change from Baseline to Week 26 n Mean (SD) | Week 26 | |
| Median Min, Max Change from Baseline to Week 26 n Mean (SD) | n | n |
| Min, Max Change from Baseline to Week 26 n Mean (SD) | Mean (SD) | xx.x (xx.xx) |
| Change from Baseline to Week 26<br>n<br>Mean (SD) | Median | XX.X |
| n<br>Mean (SD) | Min, Max | xx, xx |
| Mean (SD) | Change from Baseline to Week 26 | |
| | n | n |
| Median | Mean (SD) | xx.x (xx.xx) |
| | Median | XX.X |
| Min, Max | Min, Max | XX, XX |
| | • | |
| | • | |
| · | • | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug in 020.

path\t\_program.sas date time

#### **Table 14.2.1.2 MMSE Annualized LS Means Safety Population**

| | AD |
|---|---|
| Time Point | (N= ) |
| 513 | |
| Baseline [1] | |
| n | n |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| Min, Max | XX, XX |
| 52 Weeks<br>LS Mean <sup>[2]</sup><br>95% CI <sup>[2]</sup> | $\begin{array}{c} xx.x \\ (xx, xx) \end{array}$ |
| 104 Weeks<br>LS Mean <sup>[2]</sup><br>95% CI <sup>[2]</sup> | xx.x<br>(xx, xx) |
| ·<br>· | |

Baseline is defined as the last non-missing value prior to first dose of study drug in the prior study.

[2] LS means and 95% CIs are from a restricted maximum likelihood based repeated measures linear mixed model with fixed effects for AChEI/Memantine use as randomized in the prior study (Yes and No), time since baseline in the prior study (continuous), AChEI/Memantine use as randomized in the prior study by time interaction and the prior study baseline MMSE, prior study (015 and 005) and region (The Americas and RoW). In addition, the baseline MMSE was included as a covariate. An unstructured covariance model was used.

Table 14.2.2
RUD Lite
Safety Population: Subjects with at Least One Post-Baseline RUD Lite Questionnaire

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| RUD Lite Items | Time Point | (N= ) | (N= ) | (N= ) |
| | | | · | |
| Caregiver Time Spent on Toilet visit, etc. in Last 30 | Baseline [1] | | | |
| Days | | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Week 26 | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Change from Baseline to Week 26 | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |

Caregiver Time Spent on Shopping, etc.in Last 30 Days

-

Caregiver Time Spent on Supervising in Last 30 Days

. . .

path\t\_program.sas date time

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Table 14.2.2
RUD Lite
Safety Population: Subjects with at Least One Post-Baseline RUD Lite Questionnaire

| RUD Lite Items | Time Point | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects<br>(N= ) |
|---|---|---|---|---|
| Missed Any Whole Days of Work in Last 30 Days | Baseline <sup>[1]</sup> | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missed Any Part of Days of Work in Last 30 Days | Baseline <sup>[1]</sup> | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

...

path\t\_program.sas date time

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Table 14.2.2
RUD Lite
Safety Population: Subjects with at Least One Post-Baseline RUD Lite Questionnaire

| | Time Point | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects (N= ) |
|---|---|---|---|---|
| | Time Point | (N- ) | (IN- ) | (IN- ) |
| Patient Current Living Accommodation | Baseline [1] | n= | n= | n= |
| č | Own Home | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Intermediate Forms of Accommodation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Dementia-specific Residential Accommodation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Long-term Institutional Care | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Any permanent changes since last visit | Week 26<br>Yes | n= | n= | n= |
| Whom Patient Lives with | Baseline [1] | n= | n= | n= |
| | Alone | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Spouse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Sibling | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Child | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not Applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| Temporary Living Accommodation in Last Days | 30 Baseline [1] | n= | n= | n= |
| 2.0,0 | Own Home | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Intermediate Forms of Accommodation | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | Dementia-specific Residential Accommodation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Long-term Institutional Care | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug. path\t\_program.sas date time

Table 14.2.2
RUD Lite
Safety Population: Subjects with at Least One Post-Baseline RUD Lite Questionnaire

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| | Time Point | (N= ) | (N= ) | (N= ) |
| A1 20 10 H 2012 L 2015 | D 1: [1] | | | |
| Admitted to a Hospital in Last 30 Days | Baseline [1] | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | , | , | , |
| Ward if Admitted to a Hospital in Last 30 | ) Baseline [1] | n= | n= | n= |
| Days | Geriatric | (0/) | (0/) | (0/) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Psychiatric | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Internal Medicine | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Surgery | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Neurology | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | General Ward | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Other | | | |
| | Week 26 | n= | n= | n= |

path\t\_program.sas date time

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Table 14.2.2
RUD Lite
Safety Population: Subjects with at Least One Post-Baseline RUD Lite Questionnaire

| • • | - | AD | bvFTD | All Subject |
|---|---|---|---|---|
| | Time Point | (N= ) | (N= ) | (N= ) |
| Received Care in a Hospital Emergency Room in | LastBaseline [1] | n= | n= | n= |
| 0 Days | | | | |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| D 4 17 7 1 4 10 D | <br>D. 1: []] | | | |
| ny Doctor Visits in Last 30 Days | Baseline [1] | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Type of Care if Any Doctor Visits in Last 30 Da | ys Baseline <sup>[1]</sup> | n= | n= | n= |
| ype of care if they boctor visits in East 50 Ba | General Practitioner | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Geriatrician | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Neurologist | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Psychiatrist | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Physiotherapist | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Occupational Therapist | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Social Worker | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Psychologist | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug. path\t\_program.sas date time

Table continues on next page.
**Table 14.2.2 RUD** Lite Safety Population: Subjects with at Least One Post-Baseline RUD Lite Questionnaire

| | T' D' | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| | Time Point | (N= ) | (N= ) | (N= ) |
| Received Any Nursing Service in Last 30 Days | Baseline [1] | n= | n= | n= |
| , , | Yes | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Type of Care if Received Any Nursing Service in I 30 Days | <br>astBaseline <sup>[1]</sup> | n= | n= | n= |
| 30 Bajs | District Nurse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Home Help/Healthcare Assistant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Meals on Wheels | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Day Care | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Transportation (care related) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | | | |

path\t\_program.sas date

time

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Table 14.2.3 EQ-5D-5L Safety Population: Subjects with at Least One Post-Baseline EQ-5D-5L Questionnaire

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| | Time Point | (N= ) | (N= ) | (N= ) |
| Mobility | Baseline [1] | n= | n= | n= |
| J | I have no problems in walking about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | I have slight problems in walking about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | I have moderate problems in walking about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | I have severe problems in walking about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | I am unable to walk about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Week 26 | n= | n= | n= |
| | I have no problems in walking about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | I have slight problems in walking about | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Self-care | Baseline [1] | n= | n= | n= |
| 2011 00110 | I have no problems washing or dressing myself | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | I have slight problems washing or dressing myself | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | *** 1.00 | | | |
| | Week 26 | | | |
| ••• | | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

Note: Following the 24-Aug-2015 CRF migration, the original EQ-5D-5L eCRF was inactivated and the EQ-5D-5L Patient Rated and EQ-5D-5L Caregiver Rated eCRFs were activated. For the purposes of this summary, data obtained from the original EQ-5D-5L eCRF prior to the 24-Aug-2015 CRF migration and data obtained from the EQ-5D-5L Patient Rated eCRF after the 24-Aug-2015 CRF migration are used.

path\t program.sas date time

**Table 14.3.1.1 Study Drug Exposure and Compliance** Safety Population

| | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects (N= ) |
|---|---|---|---|
| Total Duration of Exposure (days) <sup>[1]</sup> | | | |
| n<br>M (GD) | n | n | n |
| Mean (SD) | xx.x(xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Total Duration Category (days) [2] | | | |
| 1 | n (%) [n (%)] | n (%) [n (%)] | n (%) [n (%)] |
| 2- | ( / [ ( / ] | n (%) [n (%)] | ( / [ ( / ] |
| etc. (refer to Section 5.2) | ( · -) [ ( · -)] | ( · - / [ ( · - /)] | ( ) [ ( )] |
| Duration of the Exposure Accounting for Interruptions (days) [3] | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Mean Daily Dose (mg) [4] | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX |

<sup>[1]</sup> Total duration of exposure in days is defined as the difference between the last dose date recorded on the study exit CRF page and the first dose date, plus 1 day.

<sup>[2]</sup> Number (%) of subjects in each category followed by [cumulative number (%) of subjects].
[3] Defined as the difference between the last dose date recorded on the study exit CRF page and the first dose date, minus the duration of dose interruption(s), plus 1 day.

<sup>[4]</sup> Defined as the total dose received divided by total duration of exposure.
[5] Defined as 100 x (Total Tablets Dispensed – Total Tablets Returned) / (Expected Number of Tablets).

Table 14.3.1.1 Study Drug Exposure and Compliance Safety Population

| | AD | bvFTD | All Subjects |
|---------------------------------|--------------|--------------|--------------|
| | (N= ) | (N= ) | (N= ) |
| Total Subject Years of Exposure | XXX.X | XXX.X | XXX.X |
| Cumulative Dose (mg) | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Modal Daily Dose (mg) | | | |
| Dose 1 | n (%) | n (%) | n (%) |
| Dose 2 | n (%) | n (%) | n (%) |
| Dose 3 | n (%) | n (%) | n (%) |
| etc | | | |
| Highest Daily Dose (mg) | | | |
| Dose 1 | n (%) | n (%) | n (%) |
| Dose 2 | n (%) | n (%) | n (%) |
| Dose 3 | n (%) | n (%) | n (%) |
| etc | | | |
| Compliance (%) [5] | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |

<sup>[1]</sup> Total duration of exposure in days is defined as the difference between the last dose date recorded on the study exit CRF page and the first dose date, plus 1 day.

Programming Note: Repeat table for Table 14.3.1.2 Study Drug Exposure and Compliance - Non-AChEI/Memantine Users (Safety Population)

<sup>[2]</sup> Number (%) of subjects in each category followed by [cumulative number (%) of subjects].

<sup>[3]</sup> Defined as the difference between the last dose date recorded on the study exit CRF page and the first dose date, minus the duration of dose interruption(s), plus 1 day.

<sup>[4]</sup> Defined as the total dose received divided by total duration of exposure.

<sup>[5]</sup> Defined as 100 x (Total Tablets Dispensed – Total Tablets Returned) / (Expected Number of Tablets).

Table 14.3.2.1.1.1 Overall Summary of Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) Safety Population

| | AD | bvFTD | All Subjects |
|---|---|---|---|
| | (N= ) | (N= ) | (N= ) |
| | (a.c.[2] | (0.1) | (2.1) |
| Subjects with any AE | n (%) <sup>[2]</sup> | n (%) | n (%) |
| Subjects with any Severe AE | n (%) | n (%) | n (%) |
| Subjects with any AE Related to Study Drug [1] | n (%) | n (%) | n (%) |
| Subjects with any Serious AE | n (%) | n (%) | n (%) |
| Subjects with any Serious AE Related to Study Drug [1] | n (%) | n (%) | n (%) |
| Subjects with any AE with Outcome of Death | n (%) | n (%) | n (%) |
| Subjects with any AESI | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Dose Reduction | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Dose Interruption | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Study Drug Withdrawal | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Dose Reduction, Interruption, or | n (%) | n (%) | n (%) |
| Withdrawal | . , | | . , |
| Total Number of AEs | n | n | n |
| Total Number of Severe AEs | n | n | n |
| Total Number of AEs Related to Study Drug [1] | n | n | n |
| Total Number of Serious AEs | n | n | n |
| Total Number of Serious AEs Related to Study Drug [1] | n | n | n |
| Total Number of AEs with Outcome of Death | n | n | n |
| Total Number of AESIs | n | n | n |
| Total Number of AEs Leading to Dose Reduction | n | n | n |
| Total Number of AEs Leading to Dose Interruption | n | n | n |
| Total Number of AEs Leading to Study Drug Withdrawal | n | n | n |
| Total Number of AEs Leading to Dose Reduction, Interruption, or | n | n | n |
| Withdrawal | | | •• |

<sup>[1]</sup> Includes all events reported as "Possibly Related" or "Related" to study drug.

Programming Note: Repeat table for the tables listed below

Table 14.3.2.1.1.2 Overall Summary of Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) – Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.1.2.1 Overall Summary of Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) (Safety Population)

Table 14.3.2.1.2.2 Overall Summary of Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) – Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.1.3.1 Overall Summary of Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) (Safety Population)

Table 14.3.2.1.3.2 Overall Summary of Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) – Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.1.3.3

Overall Summary of Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by Diagnosis and Prior Study Treatment Safety Population

| | | A | D | | bvFTD | |
|---|---|---|---|---|---|---|
| - | LMTM | LMTM | LMTM | LMTM | LMTM | LMTM |
| | 8 mg/day | 150 mg/day | 200 mg/day | 250 mg/day | 8 mg/day | 200 mg/day |
| | (N= ) | (N= ) | (N= ) | (N= ) | (N= ) | (N= ) |
| Subjects with any AE | n (%) <sup>[2]</sup> | n (%) | n (%) | n (%) <sup>[2]</sup> | n (%) | n (%) |
| Subjects with any Severe AE | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE Related to Study Drug [1] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any Serious AE | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any Serious AE Related to Study Drug [1] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE with Outcome of Death | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AESI | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Dose Reduction | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Dose Interruption | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Study Drug Withdrawal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with any AE Leading to Dose Reduction, Interruption, or Withdrawal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total Number of AEs | n | n | n | n | n | n |
| Total Number of Severe AEs | n | n | n | n | n | n |
| Total Number of AEs Related to Study Drug [1] | n | n | n | n | n | n |
| Total Number of Serious AEs | n | n | n | n | n | n |
| Total Number of AEs with Outcome of Death | n | n | n | n | n | n |
| Total Number of AESIs | n | n | n | n | n | n |
| Total Number of AEs Leading to Dose Reduction | n | n | n | n | n | n |
| Total Number of AEs Leading to Dose Interruption | n | n | n | n | n | n |
| Total Number of AEs Leading to Study Drug Withdrawal | n | n | n | n | n | n |
| Total Number of AEs Leading to Dose Reduction, Interruption, or | n | n | n | n | n | n |
| Withdrawal | | | | | | |

<sup>[1]</sup> Includes all events reported as "Possibly Related" or "Related" to study drug.

Table 14.3.2.2.1.1

Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term Safety Population

| System Organ Class / | AD<br>(N= ) | | bvFT<br>(N= | | (N= | All Subjects<br>(N= ) |
|---|---|---|---|---|---|---|
| Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at<br>Least One Adverse<br>Event | n (%) | n | n (%) | n | n (%) | n (%) |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n (%) |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n (%) |

Programming Note: Repeat table for the tables listed below

- Table 14.3.2.2.1.2 Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term Non-AChEI/Memantine Users (Safety Population)
- Table 14.3.2.2.2.1 Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population)
- Table 14.3.2.2.2.2 Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term

   Non-AChEI/Memantine Users (Safety Population)
- Table 14.3.2.2.3.1 Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population)
- Table 14.3.2.2.3.2 Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term Non-AChEI/Memantine Users (Safety Population)

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

Table 14.3.2.2.3.3

Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term
Safety Population

| AD | | | | | | | | bvFTD | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ | | | LMT | | LMT | | LMT | | LMT | | LMT | |
| Class / | 8 mg/c | lay | 150 mg/ | /day | 200 mg/ | 'day | 250 mg | /day | 8 mg/c | lay | 200 mg | g/day |
| Preferred | (N= | | (N= | ) | (N= | ) | (N= | ) | (N= | | (N= | ) |
| Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects<br>Reporting at<br>Least One<br>Adverse Event | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |
| System Organ<br>Class 1 | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred<br>Term 2 | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |
| System Organ<br>Class 2 | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred<br>Term 1 | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |
| Preferred<br>Term 2 | n (%) | n | n (%) | n | n (%) | n (%) | n (%) | n | n (%) | n | n (%) | n (%) |

Programming Note: Repeat table for the tables listed below

Table 14.3.2.10.3.3 Adverse Events Leading to Dose Reduction (Pre-existing Adverse Events and Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term (Safety Population)

Table 14.3.2.11.3.3 Adverse Events Leading to Dose Interruption (Pre-existing Adverse Events and Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term (Safety Population)

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

| Table 14.3.2.12.3.3 | Adverse Events Leading to Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by |
|---|---|
| | Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.13.3.3 | Adverse Events Leading to Dose Reduction, Dose Interruption or Study Drug Withdrawal (Pre-existing Adverse Events and |
| | Study-emergent Adverse Events) by Diagnosis, Prior Study Treatment, System Organ Class and Preferred Term (Safety |
| | Population) |

Table 14.3.2.3.1.1

Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class, Preferred Term and Severity Safety Population

| System Organ Class / | AD<br>(N= ) | | | bvFTD<br>(N= ) | | | All Subjects (N= ) | | |
|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Subjects Reporting at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the worst severity.

path\t\_program.sas date time

Programming Note: Repeat table for the tables listed below

| Table 14.3.2.3.1.2 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class, Preferred Term and Severity – |
|---|---|
| | Non-AChEI/Memantine Users (Safety Population) |

- Table 14.3.2.3.2.1 Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class, Preferred Term and Severity (Safety Population)
- Table 14.3.2.3.2.2 Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class, Preferred Term and Severity Non-AChEI/Memantine Users (Safety Population)
- Table 14.3.2.3.3.1 Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class, Preferred Term and Severity (Safety Population)
- Table 14.3.2.3.3.2 Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class, Preferred Term and Severity Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.4.1.1

Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class, Preferred Term and Relationship Safety Population

| System Organ Class / | O | AD<br>N= ) | | vFTD<br>N= ) | All Subjects (N= ) | |
|---|---|---|---|---|---|---|
| Preferred Term | Related [1] | Not Related [2] | Related [1] | Not Related [2] | Related [1] | Not Related [2] |
| Subjects Reporting at Least One<br>Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2<br>Preferred Term 1<br>Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the strongest relationship to study drug.

path\t program.sas date time

Programming Note: Repeat table for the tables listed below

| Table 14.3.2.4.1.2 | Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class, Preferred Term and Relationship |
|---|---|
| | - Non-AChEI/Memantine Users (Safety Population) |

Table 14.3.2.4.2.1 Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class, Preferred Term and Relationship (Safety Population)

Table 14.3.2.4.3.2 Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class, Preferred Term and Relationship – Non-AChEI/Memantine Users (Safety Population)

<sup>[1]</sup> Includes all events reported by the Investigator as "Possibly Related," or "Related" to study drug.

<sup>[2]</sup> Includes all events reported by the Investigator as "Unlikely Related" or "Not Related" to study drug.

Table 14.3.2.4.2.2 Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class, Preferred Term and Relationship – Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.4.3.1 Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class, Preferred Term and Relationship (Safety Population)

Table 14.3.2.5.1.1
Serious Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term
Safety Population

| System Organ Class / | AD<br>(N= ) | | bvFTD<br>(N= ) | | All Subjects (N= ) | |
|---|---|---|---|---|---|---|
| Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse<br>Event | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |
| • | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |

Programming Note: Repeat table for the tables listed below

| Table 14.3.2.5.1.2 | Serious Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
|---|---|
| Table 14.3.2.5.2.1 | Serious Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and<br>Preferred Term (Safety Population) |
| Table 14.3.2.5.2.2 | Serious Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| Table 14.3.2.5.3.1 | Serious Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and<br>Preferred Term (Safety Population) |
| Table 14.3.2.5.3.2 | Serious Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and<br>Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| Table 14.3.2.6.1.1 | Fatal Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.6.1.2 | Fatal Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

Table 14.3.2.6.2.1 Fatal Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.6.2.2 Fatal Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.6.3.1 Fatal Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.6.3.2 Fatal Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.7.1.1 Non-Fatal Serious Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.7.1.2 Non-Fatal Serious Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term-Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.7.2.1 Non-Fatal Serious Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.7.2.2 Non-Fatal Serious Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.7.3.1 Non-Fatal Serious Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.7.3.2 Non-Fatal Serious Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.8.1.1 Serious Adverse Reactions Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.8.1.2 Serious Adverse Reactions Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.8.2.1 Serious Adverse Reactions that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.8.2.2 Serious Adverse Reactions that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.8.3.1 Serious Adverse Reactions (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.8.3.2 Serious Adverse Reactions (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.9.1.1 Severe Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.9.1.2 Severe Adverse Events Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population) Severe Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Table 14.3.2.9.2.1 Preferred Term (Safety Population) Table 14.3.2.9.2.2 Severe Adverse Events that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.9.3.1 Severe Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.9.3.2 Severe Adverse Events (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.10.1.1 Adverse Events Leading to Dose Reduction that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population)

Table 14.3.2.10.1.2 Adverse Events Leading to Dose Reduction that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.10.2.1 Adverse Events Leading to Dose Reduction that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.10.2.2 Adverse Events Leading to Dose Reduction that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.10.3.1 Adverse Events Leading to Dose Reduction (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.10.3.2 Adverse Events Leading to Dose Reduction (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.11.1.1 Adverse Events Leading to Dose Interruption that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.11.1.2 Adverse Events Leading to Dose Interruption that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.11.2.1 Adverse Events Leading to Dose Interruption that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.11.2.2 Adverse Events Leading to Dose Interruption that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.11.3.1 Adverse Events Leading to Dose Interruption (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.11.3.2 Adverse Events Leading to Dose Interruption (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.12.1.1 Adverse Events Leading to Study Drug Withdrawal that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.12.1.2 Adverse Events Leading to Study Drug Withdrawal that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Adverse Events Leading to Study Drug Withdrawal that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) Table 14.3.2.12.2.1 by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.12.2.2 Adverse Events Leading to Study Drug Withdrawal that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.12.3.1 Adverse Events Leading to Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.12.3.2 Adverse Events Leading to Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.13.1.1 Adverse Events Leading to Dose Reduction, Dose Interruption or Study Drug Withdrawal that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.13.1.2 Adverse Events Leading to Dose Reduction, Dose Interruptio, or Study Drug Withdrawal that were Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.13.2.1 Adverse Events Leading to Dose Reduction, Dose Interruption or Study Drug Withdrawal that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population) Table 14.3.2.13.2.2 Adverse Events Leading to Dose Reduction, Dose Interruption or Study Drug Withdrawal that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) Table 14.3.2.13.3.1 Adverse Events Leading to Dose Reduction, Dose Interruption or Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term (Safety Population)

Table 14.3.2.13.3.2 Adverse Events Leading to Dose Reduction, Dose Interruption or Study Drug Withdrawal (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.14.1.1 Adverse Events of Special Interest (AESI) Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and Preferred Term **Safety Population** 

| System Organ Class /<br>Preferred Term | AD<br>(N=<br>Subjects [1] | )<br>Events | bvFTI<br>(N=<br>Subjects [1] | D<br>)<br>Events | All Subj<br>(N=<br>Subjects [1] | jects ) Events |
|---|---|---|---|---|---|---|
| Subjects Reporting at Least One<br>AESI | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |
| | n (%) | n | n (%) | n | n (%) | n |
| | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |
| | n (%) | n | n (%) | n | n (%) | n |
| | n (%) | n | n (%) | n | n (%) | n |

<sup>[1]</sup> At each level of summation (any AESI, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

path\t\_program.sas date

ramming Note: Pengat table for the tables listed hele

| Programming Note: I | Repeat table for the tables listed below |
|---|---|
| Table 14.3.2.14.1.2 | Adverse Events of Special Interest (AESI) Ongoing On Day 1 of Dosing (Pre-existing Adverse Events) by System Organ Class and |
| | Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| Table 14.3.2.14.2.1 | Adverse Events of Special Interest (AESI) that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System |
| | Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.14.2.2 | Adverse Events of Special Interest (AESI) that Started On or After Day 1 of Dosing (Study-emergent Adverse Events) by System |
| | Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population) |
| Table 14.3.2.14.3.1 | Adverse Events of Special Interest (AESI) (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ |
| | Class and Preferred Term (Safety Population) |
| - 11 | |

Table 14.3.2.14.3.2 Adverse Events of Special Interest (AESI) (Pre-existing Adverse Events and Study-emergent Adverse Events) by System Organ Class and Preferred Term - Non-AChEI/Memantine Users (Safety Population)

Table 14.3.2.15.1

Post-Treatment Adverse Events by System Organ Class and Preferred Term
Safety Population

| | AΓ | ) | bvFT | D | All Sub | jects |
|---|---|---|---|---|---|---|
| System Organ Class / | (N= | ) | (N= | ) | (N= | ) |
| Preferred Term | Subjects [1] | Events | Subjects [1] | Events | Subjects [1] | Events |
| Subjects Reporting at Least One Adverse<br>Event | n (%) | n | n (%) | n | n (%) | n |
| System Organ Class 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |
| ·<br>· | | | | | | |
| System Organ Class 2 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 1 | n (%) | n | n (%) | n | n (%) | n |
| Preferred Term 2 | n (%) | n | n (%) | n | n (%) | n |

Note: Post-treatment adverse events are defined as TEAEs that have an onset more than 14 days after the last dose of study drug.

path\t program.sas date time

Programming Note: Repeat table for Table 14.3.2.15.2 Post-Treatment Adverse Events by System Organ Class and Preferred Term – Non-AChEI/Memantine Users (Safety Population)


<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once.

TRx-237-020

Table 14.3.3.1.1.1 Hematology Values and Changes from Baseline at All Visits - Conventional Units Safety Population

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| Laboratory Parameter | Target Visit | (N= ) | (N= ) | (N= ) |
| Hematocrit (%) | Baseline [1] | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx |
| | By-visit Baseline for Week 2 Visit <sup>[2]</sup> | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx |
| | Week 2 | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| | Change from Baseline to Week 2 | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |

Hemoglobin (g/dL)

path\t program.sas date

Programming note: Table will include all hematology parameters collected from Central Laboratory, and all target visits and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Programming Note: Repeat table for the tables listed below

Table 14.3.3.1.1.2 Hematology Values and Changes from Baseline at All Visits -

Conventional Units - Non-AChEI/Memantine Users (Safety Population)

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

<sup>[2]</sup> By-visit Baseline is defined as the baseline assessments from subjects with a non-missing assessment at that visit.

| Table 14.3.3.1.2.1 | Hematology Values and Changes from Baseline at All Visits – SI Units |
|---|---|
| | (Safety Population) |
| Table 14.3.3.1.2.2 | Hematology Values and Changes from Baseline at All Visits - SI Units - |
| | Non-AChEI/Memantine Users (Safety Population) |

Table 14.3.3.2.1.1 Serum Chemistry Values and Changes from Baseline at All Visits – Conventional Units Safety Population

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| Laboratory Parameter | Target Visit | (N= ) | (N= ) | (N= ) |
| • | | | | |
| Sodium (mEq/L) | Baseline [1] | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | By-visit Baseline for Week 2 Visit <sup>[2]</sup> | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Week 2 | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Change from Baseline to Week 2 | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| Poatassium (mEq/L) | | | | |

Poatassium (mEq/L)

.

path\t\_program.sas date time

Programming note: Table will include all serum chemistry parameters collected from Central Laboratory, and all target visits and for Last Available On-Treatment Value. Please see Appendix A for visit windows.

Programming Note: Repeat table for the tables listed below

Table 14.3.3.2.1.2 Serum Chemistry Values and Changes from Baseline at All Visits – Conventional Units – Non-AChEI/Memantine Users (Safety Population)

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

<sup>[2]</sup> By-visit Baseline is defined as the baseline assessments from subjects with a non-missing assessment at that visit.

Table 14.3.3.2.2.1 Serum Chemistry Values and Changes from Baseline at All Visits – SI Units (Safety Population)

Table 14.3.3.2.2.2 Serum Chemistry Values and Changes from Baseline at All Visits – SI Units –

Non-AChEI/Memantine Users (Safety Population)

Table 14.3.3.3.1 Incidence of Potentially Clinically Significant Hematology and Serum Biochemistry Results Safety Population

| | | | AD<br>m/n (%) <sup>[1]</sup> | bvFTD<br>m/n (%) <sup>[1]</sup> | All Subjects<br>m/n (%) <sup>[1]</sup> |
|---|---|---|---|---|---|
| Laboratory Parameter | Potentially Clinically<br>Significant Criteria | Target Visit | (N= ) | (N= ) | (N= ) |
| Hematology | | | | | |
| Hemoglobin | Criteria | Baseline | m/n (%) | m/n (%) | m/n (%) |
| | | Any Post-Baseline PCS | m/n (%) | m/n (%) | m/n (%) |
| | | Any Post-Baseline | m/n (%) | m/n (%) | m/n (%) |
| | | Worsening | . , | | |
| | | Week 2 | m/n (%) | m/n (%) | m/n (%) |
| | | Week 13 | m/n (%) | m/n (%) | m/n (%) |
| Serum Chemistry | | | | | |
| Sodium | Criteria | Baseline | m/n (%) | m/n (%) | m/n (%) |
| | | Any Post-Baseline PCS | m/n (%) | m/n (%) | m/n (%) |
| | | Any Post-Baseline | m/n (%) | m/n (%) | m/n (%) |
| | | Worsening | | | |
| | | Week 2 | m/n (%) | m/n (%) | m/n (%) |
| | | Week 13 | m/n (%) | m/n (%) | m/n (%) |

Note: ULN = Upper Limit of Normal.

Note: For the post-Baseline visits, only subjects in whom the values represent a treatment-emergent worsening from Baseline (i.e. more out of range) are summarized.

path\t\_program.sas date time

Programming note: Table will include all parameters with defined potentially clinically significant ranges at each post-Baseline visit and for Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows. Ensure that criteria indicating an increase or a decrease are presented separately.

Programming Note: Repeat table for Table 14.3.3.3.2 Incidence of Potentially Clinically Significant Hematology and Serum Biochemistry Results – Non-AChEI/Memantine Users (Safety Population)

<sup>[1]</sup> m: number of subjects with at least one potentially clinically significant result at corresponding visit; n: number of subjects with at least one non-missing result at corresponding visit.

## Table 14.3.4.1.1.1 Vital Signs Safety Population

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| Vital Sign | Target Visit | (N= ) | (N= ) | (N= ) |
| Systolic BP (mmHg) | Baseline | | | |
| | n | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Baseline [1] | | | |
| | Week 2 | | | |
| | Change from Baseline to Week 2 | | | |

<sup>[1]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t\_program.sas date time

Programming note: Table will include the following vital signs: systolic BP (mmHg), diastolic BP (mmHg), heart rate (bpm), oral temperature (°C), respiratory rate (bpm) and weight (kg) for all target visits and for Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows.

Programming Note: Repeat table for Table 14.3.4.1.1.2 Vital Signs - Non-AChEI/Memantine Users (Safety Population)

## Table 14.3.4.1.2.1 Weight Directional Changes Safety Population

| Direction of Change | Target Visit | Category | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects<br>(N= ) |
|---|---|---|---|---|---|
| Increase | Baseline | 0-5 kg<br>>5 - 10 kg<br>>10 - 15 kg | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| | | etc | | | |
| Decrease | | 0-5 kg<br>>5 - 10 kg<br>>10 - 15 kg | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| | etc | etc | | | |
| path\t_program.sas date | time | | | | |

Programming note: Table will include all target visits and Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows..

Programming Note: Repeat table for Table 14.3.4.1.2.2 Weight Directional Changes - Non-AChEI/Memantine Users (Safety Population)

Table 14.3.4.1.3.1 Incidence of Potentially Clinically Significant Vital Sign Results Safety Population

| Any Post-Baseline<br>Clinically Significant Abnormalities | Potentially Clinically<br>Significant Criteria | Target Visit | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects (N= ) |
|---|---|---|---|---|---|
| Systolic Blood Pressure | Criteria | Baseline<br>Any Post-Baseline<br>Visit | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| | | Day 1 Post-Dose<br>Week 2 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| Diastolic Blood Pressure | Criteria | Baseline<br>Any Post-Baseline<br>Visit | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| | | Day 1 Post-Dose<br>Week 2 | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |

path\t\_program.sas date time

Programming note: Table will include all parameters (systolic BP (mmHg), diastolic BP (mmHg), pulse (bpm), temperature (°C), and weight (kg)) with defined potentially clinically significant ranges at each post-Baseline visit. Table will include all target visits and Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows

Programming Note: Repeat table for Table 14.3.4.1.3.2 Incidence of Potentially Clinically Significant Vital Sign Results – Non-AChEI/Memantine Users (Safety Population)

**Table 14.3.4.2 Physical Examination by Visit Safety Population** 

| | | AD | bvFTD | All Subjects |
|-------------|--------------|-------|-------|--------------|
| Body System | Time Point | (N= ) | (N= ) | (N= ) |
| Skin | Baseline [1] | (n=) | (n=) | (n=) |
| | Normal | n (%) | n (%) | n (%) |
| | Abnormal NCS | n (%) | n (%) | n (%) |
| | Abnormal CS | n (%) | n (%) | n (%) |
| | Week 2 | (n=) | (n=) | (n=) |
| | Normal | n (%) | n (%) | n (%) |
| | Abnormal NCS | n (%) | n (%) | n (%) |
| | Abnormal CS | n (%) | n (%) | n (%) |

Head

path\t\_program.sas date time

Programming note: Table will include all body systems for all target visits and for Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows.

Note: NCS = Not clinically significant, CS = Clinically significant.

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

**Table 14.3.4.3 Neurological Examination by Visit Safety Population** 

| | | AD | bvFTD | All Subjects |
|-------------|--------------|-------|-------|--------------|
| Body System | Time Point | (N= ) | (N= ) | (N= ) |
| Appearance | Baseline [1] | (n=) | (n=) | (n=) |
| | Normal | n (%) | n (%) | n (%) |
| | Abnormal NCS | n (%) | n (%) | n (%) |
| | Abnormal CS | n (%) | n (%) | n (%) |
| | Week 2 | (n=) | (n=) | (n=) |
| | Normal | n (%) | n (%) | n (%) |
| | Abnormal NCS | n (%) | n (%) | n (%) |
| | Abnormal CS | n (%) | n (%) | n (%) |

Behaviour

path\t\_program.sas date time

Programming note: Table will include all body systems for all target visits and for Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows.

Note: NCS = Not clinically significant, CS = Clinically significant.

[1] Baseline is defined as the last non-missing value prior to first dose of study drug.

TRx-237-020

Table 14.3.4.4.1 Serotonin Toxicity (Syndrome) Assessment by Visit Safety Population

| | Time point | AD<br>(N= ) | bvFTD<br>(N= ) | All Subjects<br>(N= ) |
|---|---|---|---|---|
| Sign or Symptom of Serotonin Toxicity (Syndrome)<br>Exhibited [1] | Baseline | (n=)<br>n (%) | (n= )<br>n (%) | (n= )<br>n (%) |
| | Week 2 | (n=)<br>n (%) | (n=)<br>n (%) | (n= )<br>n (%) |

. . . .

Note: Baseline is defined as the last non-missing value prior to first dose of study drug.

path\t program.sas date time

Programming note: Table will include all target visits and Last Available On-Treatment Value. Please see Appendix A for target visits and visit windows.

Programming Note: Repeat table for Table 14.3.4.4.2 Serotonin Toxicity (Syndrome) Assessment by Visit – Non-AChEI/Memantine Users (Safety Population)

<sup>[1]</sup> Subjects are counted if they answered "yes" to any of the signs or symptoms on the Serotinin Toxicity (Syndrome) Assessment form.

## Table 14.3.4.5.1 Central ECG Data by Visit Safety Population

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| ECG Parameter | Time Point | (N= ) | (N= ) | (N= ) |
| W ( 1 D ( (1 ) | p. 1: []] | | | |
| Ventricular Rate (bpm) | Baseline [1] | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Week 26 | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Change from Baseline to Week 26 | | | |
| | N | n | n | n |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx |

PR Interval (msec)

...

path\t\_program.sas date time

Programming note: table will include all target visits and Last Available On-Treatment Value and the following ECG parameters: Ventricular Rate (beats/min), PR Interval (msec), QRS Duration (msec), QTcB Interval (msec), QTcF Interval (msec). See Appendix A for visit windows.

<sup>[1]</sup> Baseline is defined as the mean of the last non-missing triplicate values prior to first dose of study drug. Note: The summaries are based on the measurements from central read (BIOCLINICA).

Table 14.3.4.5.2 Central ECG Data – Change from Baseline in Investigator's Overall Interpretation of Clinical Significance by Visit
Safety Population

| | | $\begin{array}{c} \text{AD} \\ \text{(N= )} \\ \text{Baseline}^{[1]} \end{array}$ | | | bvFTD<br>(N= )<br>Baseline <sup>[1]</sup> | | | All Subjects (N= ) Baseline <sup>[1]</sup> | |
|---|---|---|---|---|---|---|---|---|---|
| Target Visit | Normal | Abnormal<br>CS | Abnormal<br>NCS | Normal | Abnormal<br>CS | Abnormal<br>NCS | Normal | Abnormal<br>CS | Abnormal<br>NCS |
| Week 26 | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal NCS | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal CS | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Week 52 | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal NCS | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal CS | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

. . .

Note: CS = Clinically Significant, NCS = Not Clinically Significant. The clinical significance was determined by the investigator.

path\t program.sas date time

<sup>[1]</sup> Baseline is defined as the last non-missing value among triplicate values prior to first dose of study drug.

Table 14.3.4.5.3 Central ECG Data - QTc Abnormalities **Safety Population** 

| | | AD | bvFTD | All Subjects |
|---|---|---|---|---|
| ECG Parameter | Target Visit | (N= ) | (N= ) | (N= ) |
| | - v III | | | |
| QTcF Interval (msec) | Baseline <sup>[1]</sup> | (n=) | (n=) | (n=) |
| | >450 ms to ≤480 ms | n (%) | n (%) | n (%) |
| | >480 ms to ≤500 ms | n (%) | n (%) | n (%) |
| | >500 ms | n (%) | n (%) | n (%) |
| | Week 26 | (n=) | (n=) | (n=) |
| | >450 ms to ≤480 ms | n (%) | n (%) | n (%) |
| | >480 ms to ≤500 ms | n (%) | n (%) | n (%) |
| | >500 ms | n (%) | n (%) | n (%) |
| | Change from Baseline to Week 26 | (n=) | (n=) | (n=) |
| | >30 ms to ≤60 ms | n (%) | n (%) | n (%) |
| | >60 ms to <90 ms | n (%) | n (%) | n (%) |
| | ≥90 ms | n (%) | n (%) | n (%) |

QTcB Interval (msec)

path\t\_program.sas date time

<sup>[1]</sup> Baseline is defined as the mean of the last non-missing triplicate values prior to first dose of study drug. Note: The categories are based on the average of triplicate measurements from central read (BIOCLINICA).

**Appendix H: Figure Layouts** 

Figure 14.2.4.1 Observed Mean MMSE by Visit Safety Population



Reference: Table 14.2.1.1 path\t\_program.sas date time

Programming Note: Repeat for the figure:

Figure 14.2.4.2 Annualized Mean Change from Baseline in MMSE (Safety Population)

Figure 14.3.5.1.1 Hemoglobin by Visit – Conventional Units Safety Population



Notes: the upper bar is the 90th percentile, the lower bar is the 10th percentile; += Mean, \*= Outlier; Most Frequent Normal Range Used, *Gender* Aged xx-xx. Low = xxx g/L High = xxx g/L path\t\_program.sas date time

Programming Note: Repeat figure for the figures listed on the following page:

| Figure 14.3.5.1.2 | Box Plots of Hemoglobin Change from Baseline by Visit – Conventional Units (Safety Population) |
|---|---|
| Figure 14.3.5.1.3 | Box Plots of Hemoglobin by Visit – SI Units (Safety Population) |
| Figure 14.3.5.1.4 | Box Plots of Hemoglobin Change from Baseline by Visit – SI Units (Safety Population) |
| Figure 14.3.5.2.1 | Box Plots of Reticulocytes by Visit – Conventional Units (Safety Population) |
| Figure 14.3.5.2.2 | Box Plots of Reticulocytes Change from Baseline by Visit – Conventional Units (Safety Population) |
| Figure 14.3.5.2.3 | Box Plots of Reticulocytes by Visit – SI Units (Safety Population) |
| Figure 14.3.5.2.4 | Box Plots of Reticulocytes Change from Baseline by Visit – SI Units (Safety Population) |
| Figure 14.3.5.3.1 | Box Plots of Neutrophils by Visit (Safety Population) |
| Figure 14.3.5.3.2 | Box Plots of Neutrophils Change from Baseline by Visit (Safety Population) |
| Figure 14.3.5.4.1 | Box Plots of Albumin by Visit - Conventional Units (Safety Population) |
| Figure 14.3.5.4.2 | Box Plots of Albumin Change from Baseline by Visit – Conventional Units (Safety Population) |
| Figure 14.3.5.4.3 | Box Plots of Albumin by Visit – SI Units (Safety Population) |
| Figure 14.3.5.4.4 | Box Plots of Albumin Change from Baseline by Visit – SI Units (Safety Population) |
| Figure 14.3.5.5.1 | Box Plots of ALT by Visit (Safety Population) |
| Figure 14.3.5.5.2 | Box Plots of ALT Change from Baseline by Visit (Safety Population) |
| Figure 14.3.5.6.1 | Box Plots of AST by Visit (Safety Population) |
| Figure 14.3.5.6.2 | Box Plots of AST Change from Baseline by Visit (Safety Population) |
| Figure 14.3.5.7.1 | Box Plots of Alkaline Phosphatase by Visit (Safety Population) |
| Figure 14.3.5.7.2 | Box Plots of Alkaline Phosphatase Change from Baseline by Visit (Safety Population) |
| Figure 14.3.5.8.1 | Box Plots of Total Bilirubin by Visit – Conventional Units (Safety Population) |
| Figure 14.3.5.8.2 | Box Plots of Total Bilirubin Change from Baseline by Visit – Conventional Units (Safety Population) |
| Figure 14.3.5.8.3 | Box Plots of Total Bilirubin by Visit – SI Units (Safety Population) |
| Figure 14.3.5.8.4 | Box Plots of Total Bilirubin Change from Baseline by Visit – SI Units (Safety Population) |
| Figure 14.3.5.9.1 | Box Plots of Direct Bilirubin by Visit – Conventional Units (Safety Population) |
| Figure 14.3.5.9.2 | Box Plots of Direct Bilirubin Change from Baseline by Visit - Conventional Units (Safety Population) |
| Figure 14.3.5.9.3 | Box Plots of Direct Bilirubin by Visit – SI Units (Safety Population) |
| Figure 14.3.5.9.4 | Box Plots of Direct Bilirubin Change from Baseline by Visit – SI Units (Safety Population) |
### **Appendix I: Listing Layouts**

#### Listing 16.2.1.1.1 Subjects Who Entered the Study All Enrolled

| Subject<br>ID | Prior Study<br>Subject ID | Prior Study<br>Treatment | Site | Prior Study Site [1] |
|---|---|---|---|---|
| xxxxxx | xxxxxx | XXXXXX | xxxxxx | XXXXXX |
| XXXXXX | xxxxxx | xxxxxx | xxxxxx | XXXXXX |
| xxxxx* | xxxxxx | xxxxxx | XXXXXX | xxxxxx |
| XXXXXX | xxxxxx | xxxxxx | xxxxxx | XXXXXX |
| XXXXXX | xxxxxx | xxxxxx | xxxxxx | XXXXXX |
| xxxxx* | xxxxxx | xxxxxx | XXXXXX | xxxxxx |
| XXXXXX | xxxxxx | xxxxxx | XXXXXX | xxxxxx |

Note: \* indicates a Non-AChEI/Memantine User. Note: # indicates the subject was not dosed in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Add a flag for Non-AChEI/Memantine Users.

<sup>[1]</sup> If a subject did not change sites, this field will be left blank. Note: \* indicates a Non-AChEI/Memantine User.

#### Listing 16.2.1.1.2 Informed Consent All Enrolled

#### Date Caregivers Signed Informed Consent

| | | Protocol | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Version | | | | | | | | | | |
| | Date of | Date of | | | | | Legally | Did a Study | | | | |
| Subject | Informed | Initial | Primary | Secondary | Third | Fourth | Authorized | Participant | Study | Date of | Protocol | Reason for |
| ID | Consent | Consent | Caregiver | Caregiver | Caregiver | Caregiver | Representative | Reconsent? | Participant | Reconsent | Version | Reconsent |
| XXXXXX | date9. | date9. | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | Yes/No | XXXX | date9. | date9. | XXXXXX |

path\l\_program.sas date time

Programming note: Sort by subject ID. Do not include records where reason for reconsent = Reconsent for Additional 12 Months'

TRx-237-020

#### Listing 16.2.1.1.3 Reconsent for Additional 12-Month Treatment Extension All Enrolled

| | | | | | Subject Will Continue in | Primary Reason Subject Did |
|---|---|---|---|---|---|---|
| | Subject ID | Study Participant | Date of Reconsent | Reason for Reconsent | OLEX | Not Reconsent |
| _ | | | | | | |
| | XXXXXX | XXXX | date9. | xxxxxx | Yes/No | XXXXXX |
| | XXXXXX | XXXX | date9. | xxxxxx | Yes/No | xxxxxx |
| | XXXXXX | XXXX | date9. | xxxxxx | Yes/No | XXXXXX |
| | XXXXXX | XXXX | date9. | xxxxxx | Yes/No | xxxxxx |
| | XXXXXX | XXXX | date9. | xxxxxx | Yes/No | XXXXXX |
| | XXXXXX | XXXX | date9. | xxxxxx | Yes/No | xxxxxx |
| | XXXXXX | xxxx | date9. | xxxxxx | Yes/No | xxxxxx |

path\l\_program.sas date time

Programming note: Sort by subject ID. Only include records where reason for reconsent = Reconsent for Additional 12 Months'. Sources for the columns 'Subject Will Continue in OLEX' and 'Primary Reason Subject Did Not Reconsent' are the Visit 6 and Visit 10 CRFs.

#### Listing 16.2.1.2 Subject Disposition All Enrolled

| Subject<br>ID | Date of Study Completion or<br>Discontinuation (Study Day) | End Date of Study Drug<br>Administration | End Time of Study Drug<br>Administration | Reason(s) for Study<br>Completion/Discontinuation |
|---|---|---|---|---|
| xxxxxx | date9. (day) | date9. | time5. | Reason* |
| XXXXXX | date9. (day) | date9. | time5. | Reason {including Other description} |
| XXXXXX | date9. (day) | date9. | time5. | Reason |

Note: \* indicates primary reason.

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. If reasons for study completion/discontinuation are 'Withdrawal of Consent by Subject,' 'Withdrawal of Consent by Caregiver', 'Withdrawal of Consent by Legally Acceptable Representative', and/or 'Physician Decision,' then concatenate additional related reason ro main reason with a colon (':'), i.e., 'Physician Decision: Specified Reason.'

#### Listing 16.2.1.3 Subject Visit Dates All Enrolled

| Subject<br>ID | Last Visit (Date)<br>from<br>Prior Study | Does Visit 1 –<br>Baseline<br>Coincide with<br>Final Visit? | If No, Have 42<br>Days Elapsed Since<br>Final Visit? | Visit | Visit Date<br>(Study Day) | Visit<br>Not Done | If Not Done,<br>Specify Reason |
|---|---|---|---|---|---|---|---|
| xxxxxx | Visit xx Week xx | | | Screening | date | | |
| | (date9.) | Yes/No | Yes/No | D 1' | 1.4 | | |
| | | | | Baseline | date | | |
| | | | | Week 2 | Not Done: Specify | 7 | |
| | | | | Week 6 | date | | |
| | | | | Week 13 | date | | |
| | | | | Week 26 | date | | |
| | | | | Week 39 | date | | |
| | | | | Week 52 | date | | |
| | | | | Week 56 | date | | |
| | | | | Follow-up Visit | date | | |
| xxxxxx | | | | Unscheduled | date | | |

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID and visit date. Display the CRF visit label.

#### Listing 16.2.2.1 Protocol Deviations Safety Population

| Subject | | | | |
|---|---|---|---|---|
| ID | Treatment Group | Protocol Deviation Category | Deviation Type | CSR Impact |
| XXXXXX | XXXXXXXXX | Category | | Impact/No impact |

path\l\_program.sas date time

Programming note: Sort by subject ID.


Listing 16.2.2.2 Withdrawal of Consent Safety Population

| Subject | Study Participant<br>Who Withdrew | |
|---------|-----------------------------------|-----------------|
| ΙĎ | Consent | Withdrawal Date |
| XXXXXX | XXXXXX | date9. |
| XXXXXX | XXXXXX | date9. |
| XXXXXX | XXXXXX | date9. |
| XXXXXX | XXXXXX | date9. |
| XXXXXX | XXXXXX | date9. |
| XXXXXX | XXXXXX | date9. |
| XXXXXX | XXXXXX | date9. |

Programming note: Sort by subject ID.

Listing 16.2.2.3 Inclusion/Exclusion Criteria Safety Population

\

| Subject<br>ID | Did subject meet all eligibility criteria? | Criterion No. | Protocol Version<br>Date |
|---|---|---|---|
| XXXXXX | Yes/No | XXXXXX | date9. |
| XXXXXX | Yes/No | XXXXXX | date9. |
| XXXXXX | Yes/No | XXXXXX | date9. |
| XXXXXX | Yes/No | XXXXXX | date9. |
| XXXXXX | Yes/No | XXXXXX | date9. |
| XXXXXX | Yes/No | XXXXXX | date9. |
| XXXXXX | Yes/No | XXXXXX | date9. |

path\l\_program.sas date time

Programming note: Sort by subject ID.

# Listing 16.2.4.1 Demographics and Baseline Characteristics Safety Population Part 1 of 2

| | | | | Females, | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Childbearing | Main Method | | | | Who Does the |
| | | | | Status | of Adequate | | | Subject's Living | Subject Live |
| Subject ID | Country | Age (years) [1] | Gender | Details <sup>[2]</sup> | Contraception <sup>[3]</sup> | Ethnicity | Race | Accommodation | With? |
| XXXXXX | Country | XX | Male/Female | X | X | Ethnicity | Race | XXXXXX | XXXXXX |

<sup>[1]</sup> Age at informed consent to participation in the prior study.

path\l program.sas date time

<sup>&</sup>lt;sup>[2]</sup> 1=Surgically Sterile (Hysterectomy, Bilateral Salpingectomy or Oophorectomy); 2=Bilateral Tubal Ligation or Occlusion; 3=Post-Menopausal for at Least 1 Year; 4=Using Adequate Contraception.

<sup>[3] 1=</sup>Condoms with spermicidal foam, gel, film, cream, or suppository; 2=Diaphragm with spermicidal foam, gel, film, cream, or suppository; 3=Cervical/Vault caps with spermicidal foam, gel, film, cream, or suppository; 4=Intrauterine device or system; 5=Oral or long-acting injected or implanted hormonal contraceptives for at least 3 months prior to Baseline; 6=Vasectomized partner; 7=True abstinence.

Listing 16.2.4.1
Demographics and Baseline Characteristics
Safety Population
Part 2 of 2

| Subject ID | Height (cm) | Weight (kg) | $\frac{\mathrm{BMI}}{\mathrm{(kg/m^2)}}$ | MMSE | Use of AChEI/Memantine |
|---|---|---|---|---|---|
| XXXXXX | XX | XX | XX.X | XX.X | Yes/No |
| XXXXXX | XX | XX | XX.X | XX.X | Yes/No |
| xxxxxx | XX | XX | XX.X | XX.X | Yes/No |
| xxxxxx | XX | XX | XX.X | XX.X | Yes/No |
| xxxxxx | XX | XX | XX.X | XX.X | Yes/No |
| xxxxxx | XX | XX | XX.X | XX.X | Yes/No |
| XXXXXX | XX | XX | XX.X | XX.X | Yes/No |

Programming note: Sort by subject ID.

#### Listing 16.2.4.2 Medical History at Study Entry Safety Population

| | | CRF | Onset | | |
|---|---|---|---|---|---|
| | MedDRA | Start/Stop | Date | | End Date |
| | System | Date | (Study | | (Study |
| Subject ID | Organ Class Condition // MedDRA Preferred Term | Unknown | Day) | Ongoing/Resolved | Day) |
| • | | | | | |
| XXXXXX | Body System Verbatim term // MedDRA Preferred Term | Checkbox | date9. | Ongoing/Resolved | date9. |
| | Body System Verbatim term // MedDRA Preferred Term | value | date9. | Ongoing/Resolved | date9. |
| | Body System Verbatim term // MedDRA Preferred Term | | date9. | Ongoing/Resolved | date9. |
| XXXXXX | Body System Verbatim term // MedDRA Preferred Term | | date9. | Ongoing/Resolved | date9. |
| | Body System Verbatim term // MedDRA Preferred Term | | date9. | Ongoing/Resolved | date9. |
| | Body System Verbatim term // MedDRA Preferred Term | | date9. | Ongoing/Resolved | date9. |

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programmer note: sort by subject ID and onset date within each subject. Combine data collected from Prior Study – Medical History and Medical History CRF pages and flag Medical History CRF records with asterisk (\*).

<sup>\*=</sup>Medical History additions as of the start of this study.

#### Listing 16.2.4.3.1 **Prior Medications** Safety Population

| | | | | | | | | | Anti-Psychotic | If Yes, |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Verbatim Term // Generic | Start Date | Stop Date | | | Dose | | | Drug? | Reason |
| ID | Name | (Study Day) | (Study Day) | Dose | Units | Form Rout | e Frequency | Indication | | for Use |
| xxxxxx | Verbatim Term // Generic<br>Name | date9. (xx) | date9. (xx) | dose | unit | dose route | e frequency | indication | Yes/No | xxxx |
| | Verbatim Term // Generic<br>Name | date9. (xx) | date9. (xx) | dose | unit | dose route<br>form | e frequency | indication | Yes/No | XXXX |
| | Verbatim Term // Generic<br>Name | date9. (xx) | date9. (xx) | dose | unit | dose route<br>form | e frequency | indication | Yes/No | XXXX |
| xxxxxx | Verbatim Term // Generic<br>Name | date9. (xx) | date9. (xx) | dose | unit | dose route<br>form | e frequency | indication | Yes/No | xxxx |
| | Verbatim Term // Generic<br>Name | date9. (xx) | date9. (xx) | dose | unit | dose route<br>form | e frequency | indication | Yes/No | XXXX |
| | Verbatim Term // Generic<br>Name | date9. (xx) | date9. (xx) | dose | unit | dose route<br>form | e frequency | indication | Yes/No | XXXX |

Note: Prior Medications are those medications that were started or ongoing at the end of the prior study participation and were stopped prior to the 020 first dose date. Study day is calculated as days prior to the date of first dose of study drug in 020. \*Medications with serotonergic potential

path\1 program.sas date time

Programmer note: sort by subject ID and start date and stop date within each subject. Include medications that fit the prior medications definition from both the Concomitant Medications and Prior-Study - Concomitant Medications CRF pages.

Programming Note: Repeat listing for the listings listed below

Concomitant Medications (Safety Population) - see Section 5.6 for sources Listing 16.2.3.3.2

Procedures or Therapies (Safety Population) {include Subject ID, Any Procedures/Therapies Listing 16.2.3.4 Performed? (Y/N), Description, Start and Stop Dates, and Ongoing (Yes, if checked)}

Listing 16.2.5.1 **Drug Accountability and Compliance Safety Population** 

| Subject<br>ID | Visit | Date of<br>Administration<br>(Study Day) | Package ID<br>Dispensed<br>(1 <sup>st</sup> /2 <sup>nd</sup> /3 <sup>rd</sup> ) | Tablets | Package ID<br>Returned<br>(1 <sup>st</sup> /2 <sup>nd</sup> /3 <sup>rd</sup> ) | Tablets | | Compliance <sup>[1]</sup> | Comments |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | Day 1 | date9. (xx) | XX | XX | xx | XX | Yes/No | XX.X | |
| | Week 2 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| | Week 6 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| xxxxxx | Day 1 | date9. (xx) | XX | xx | xx | xx | Yes/No | XX.X | |
| | Week 2 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| | Week 6 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| xxxxxx | Day 1 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| | Week 2 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| | Week 6 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| xxxxxx | Day 1 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| | Week 2 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |
| | Week 6 | date9. (xx) | XX | XX | XX | XX | Yes/No | XX.X | |

...

path\l program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.


Note: Study day is calculated as days since the date of first dose of study drug in 020.

[1] Defined as 100 x (Total Tablets Dispensed – Total Tablets Returned) / (Expected Number of Tablets).

#### Listing 16.2.5.2 By-Subject Summary of Overall Exposure Safety Population

#### Treatment Duration

| Subject<br>ID | Treatment Duration | Accounting for Interruptions [2] | Mean Daily Dose (mg) <sup>[3]</sup> | Modal Daily Dose (mg) |
|---|---|---|---|---|
| xxxxxx | xxx | xxx | x.xx | x.xx |
| xxxxxx | xxx | xxx | x.xx | x.xx |
| xxxxxx | xxx | XXX | X.XX | X.XX |
| xxxxxx | xxx | XXX | X.XX | X.XX |

. . .

path\l program.sas date time

Programming note: Sort by subject ID.


<sup>[1]</sup> Duration of exposure in days is defined as the difference between the last dose date recorded on the study exit CRF page and the first dose date, plus 1 day.

Duration of exposure accounting for interruptions in days is defined as the difference between the last dose date recorded on the study exit CRF page and the first dose date, minus the duration of dose interruption(s), plus 1 day.

<sup>[3]</sup> Defined as the total dose received divided by duration of exposure.

Listing 16.2.5.3
Chronological Study Drug Administration Including Dose Interruption and Adjustment Safety Population

| <u></u> | Subject<br>ID | Start Date of Administration (Study Day) | Stop Date of Administration (Study Day) | Daily Dose | Comment |
|---|---|---|---|---|---|
| | | 1 . 0 | 1 . 0 | | |
| | XXXXXX | date9. | date9. | xx mg | Comment |
| | XXXXXX | date9. | date9. | xx mg | Comment |
| | XXXXXX | date9. | date9. | xx mg | Comment |
| | XXXXXX | date9. | date9. | xx mg | Comment |
| | XXXXXX | date9. | date9. | xx mg | Comment |
| | XXXXXX | date9. | date9. | xx mg | Comment |

Programming note: Sort by subject ID.

Listing 16.2.6.1 RUD Lite Safety Population Part 1 of 6

| | | | | | | | | Caregiver | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Descri | ption of Pi | rimary Ca | regiver | |
| | | | | | Previous | Completed | | | | | # of | | | |
| | | | | | Assessment | within prior 42 | Date of | | | | Children | Live with | | |
| Subject | Int | erview | Start | End | Completed in | days of Prior | Previous | | | Relationship | Living | the | # of Other | Level of |
| ID Vis | sit I | Date | Time | Time | Prior Study? | Study? | Assessement | Age | Gende | to Patient | with | Patient? | Caregivers | Contribution |
| xxxxxx Day | y 1 d | ate9. | time5. | time5. | Yes/No | Yes/No | date9. | $\mathbf{X}\mathbf{X}$ | F/M | Relationship | XX | Yes/No | XX | xx-xx% |
| We | ek Not | Done: | | | | | | | | | | | | |
| 20 | sp | ecify | | | | | | | | | | | | |
| We | ek d | ate9. | time5. | time5. | | | | $\mathbf{X}\mathbf{X}$ | F/M | Relationship | XX | Yes/No | XX | xx-xx% |
| 52 | 2 | | | | | | | | | | | | | |
| xxxxxx Day | v 1 d | ate9. | time5. | time5. | Yes/No | Yes/No | date9. | XX | F/M | Relationship | XX | Yes/No | XX | xx-xx% |
| We | | | time5. | | | | | XX | | Relationship | XX | Yes/No | XX | xx-xx% |
| 20 | 5 | | | | | | | | | 1 | | | | |
| We | ek d | ate9. | time5. | time5. | | | | XX | F/M | Relationship | XX | Yes/No | XX | xx-xx% |
| 52 | 2 | | | | | | | | | • | | | | |
| xxxxxx Day | , 1 d | ate9. | time5. | time5 | Yes/No | Yes/No | date9. | XX | F/M | Relationship | XX | Yes/No | XX | xx-xx% |
| We | | | time5. | | 1 03/110 | 1 05/110 | date). | XX | | Relationship | XX | Yes/No | XX | xx-xx% |
| 20 | | aics. | unics. | umes. | | | | λλ | 1./161 | Relationship | АА | 1 68/110 | AA | AA-AA / 0 |
| We | - | ate9. | time5. | time5 | | | | XX | E/M | Relationship | XX | Yes/No | XX | xx-xx% |
| 52 | | aic). | unics. | unics. | | | | ΛΛ | 1 / IVI | Relationship | ΛΛ | 1 05/110 | ΛΛ | AA-AA/0 |
| •• | • | | | | | | | | | | | | | |

Listing 16.2.6.1 RUD Lite Safety Population Part 2 of 6

| | | | | | Caregiver | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Care | giver T | ime Sp | ent | | | |
| | | | | | | | Assi | sting pa | tient with toilet | A | ssisting | patient with | | | |
| | | | | | Slee | eping | | visi | its, etc. | | shop | oing, etc. | Sup | ervisir | ng the patient |
| | | | | | On a | typical | On a | typical | | On a | typical | | On a | typical | |
| | | | | | care | day | | day | | care | day | | care | day | |
| | | | | | durir | ng last | durir | ıg last | During the last | durir | ng last | During the last | durir | ng last | During the last |
| | | | | | 30 | days | 30 days 30 days | | | days | 30 days | 30 | days | 30 days | |
| Subject | | Interview | Start | End | # of | # of | # of | # of | # of | # of | # of | # of | # of | # of | # of |
| ΙĎ | Visit | Date | Time | Time | Hrs. | Min. | Hrs. | Min. | Days | Hrs. | Min. | Days | Hrs. | Min. | Days |
| XXXXXX | Day 1 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week | Not Done: | | | | | | | | | | | | | |
| | 26 | specify | | | | | | | | | | | | | |
| | Week | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | 52 | | | | | | | | | | | | | | |
| XXXXXX | Day 1 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | 26 | | | | | | | | | | | | | | |
| | Week | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | 52 | | | | | | | | | | | | | | |
| XXXXXX | Day 1 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | 26 | | | | | | | | | | | | | | |
| | Week | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | 52 | | | | | | | | | | | | | | |

Listing 16.2.6.1 RUD Lite Safety Population Part 3 of 6

| | | | | | Ca | aregiver | | | | Patient | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Caregive | er work statu | S | | | tient Living Accon | | | |
| | | | | | # of tin | nes caregiver | If patient made | e perman | ent | If patient moved to | a new location for | more than 24 | hours, # |
| | | | | | status a | ffected work | change since | e last vis | it | of n | ights at temporary le | ocation | |
| | | | | | Missed | | | | | | | | |
| | | | | | a whole | Missed part | | | | | | Long-term | |
| Subject | | Interview | Start | End | day of | of a day of | Current | Date of | Own | Intermediate | Dementia-specific | institutional | Other, |
| ID | Visit | Date | Time | Time | work | work | Accommodations | move | home | Accommodation | accommodation | care | specify |
| xxxxxx | - | date9.<br>Not Done: | | time5 | . xx | xx | xxxxxx | date9. | xx | XX | xx | xx | XX |
| | 26<br>Week<br>52 | specify date9. | time5. | time5 | . XX | xx | xxxxxx | date9. | xx | XX | XX | XX | xx |
| xxxxxx | Day 1 | date9. | time5. | time5 | . xx | XX | xxxxxx | date9. | XX | XX | XX | XX | XX |
| | Week<br>26 | date9. | time5. | time5 | . XX | XX | XXXXXX | date9. | XX | XX | XX | XX | XX |
| | Week<br>52 | date9. | time5. | time5 | . XX | XX | xxxxxx | date9. | XX | XX | XX | XX | XX |
| | <br>Doz. 1 | dataO | time5. | tim 05 | | | | date9. | **** | | | | |
| XXXXXX | • | | | | | XX | XXXXXX | | XX | XX | XX | XX | XX |
| | Week<br>26 | date9. | time5. | umes | . XX | XX | XXXXXX | date9. | XX | XX | XX | XX | XX |
| | Week<br>52 | date9. | time5. | time5 | . XX | XX | xxxxxx | date9. | XX | XX | XX | XX | xx |

Listing 16.2.6.1 RUD Lite Safety Population Part 4 of 6

| | | | | | | | | | Patient | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Patien | t Health ( | Care Resou | rce Utilisation | | |
| | | | | | | | # of nig | hts spent | in hospital | since last visit | | |
| Subject | T- | ntervieu | v Start End | # of times<br>hospitalized<br>in last 30 | | | Internal | | | | | # of times in<br>hospital ER<br>in last 30 |
| | √isit | Date | Time Time | days | Geriatr | ic Psychiatri | | | Neurology | General Ward | Other, specify | days |
| -12 | . 1510 | 2 | 111110 111110 | uujs | 0411441 | 101 0) 01114411 | | | | General Ware | o their, specify | |
| | Veek | Not | time5.time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Done: specify | | | | | | | | | | |
| | 52 | date9. | time5.time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| D | 1 | 1-4-0 | | | | | | | | | | |
| xxxxxx D | • | | time5.time5. | | XX | XX | XX | XX | XX | XX | XX | XX |
| | Veek<br>26 | date9. | time5.time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Veek<br>52 | date9. | time5.time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| xxxxxx D | <br>Oav 1 | date9. | time5.time5. | XX | XX | XX | xx | XX | XX | XX | XX | XX |
| | - | | time5.time5. | | XX | XX | XX | XX | XX | XX | XX | XX |
| | 26 | | | | | | | | | | | |
| | Veek<br>52 | date9. | time5.time5. | XX | XX | XX | XX | xx | XX | XX | XX | XX |
| | • • • | | | | | | | | | | | |

#### Listing 16.2.6.1 RUD Lite Safety Population Part 5 of 6

| | | | | | | Patient Patient Health Care Resource Utilisation | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Patient | Health Ca | are Resou | rce Utilisa | tion | | | |
| | | | | | | | | | | # of | visits | | | | |
| Subject<br>ID | Visit | Interview<br>Date | | End<br>Time | # of times<br>admitted to a<br>hospital since<br>the last visit | None | General<br>Practitioner | Geria-<br>trician | Neuro-<br>logist | Psychi-<br>atrist | | Occupational<br>Therapist | | Psycho-<br>logist | Other, specify |
| xxxxxx | Day 1<br>Week<br>26 | Not<br>Done: | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week 52 | specify date9. | time5. | time5. | xx | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| XXXXXX | Day 1 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week<br>26 | | time5. | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week<br>52 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | 1 . 0 | | | | | | | | | | | | | |
| XXXXXX | | | time5. | | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week<br>26 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Week 52 | date9. | time5. | time5. | XX | XX | XX | XX | XX | XX | xx | XX | XX | XX | XX |

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Listing 16.2.6.1 RUD Lite Safety Population Part 6 of 6

| | | | | | | Patient Patient Health Care Resource Utilisation | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | • | | | | 1 41 | | es servic | | | 11 | | | |
| | | | | | | | | | # 01 11111 | Meals | e was it | eceived | | | | |
| | | | | | | | | Home Help/He | aalthaara | on | | | Transpor | tation | | |
| | | | | | | Dietri | ct Nurse | Assista: | | Wheels | Day | Care | (Care Re | | 0 | ther |
| | | | | | No | Distri | ot Ivuisc | Assista | 111 | WHEELS | Day | Carc | (Care Re | iaicu) | | rifici |
| Subject | т. | ntomion | v Start | End | services | # of | # of | | # of | # of | # of | # of | | | # of | # of |
| Subject<br>ID V | 7isit | Date | | | received | | hrs/visit | # of visits | hrs/visit | | # 01<br>visits | hrs/visit | # of visits | Specify | | hrs/visits |
| 1D V | 1811 | Date | Time | Tille | received | VISITS | III S/ VISIt | # OI VISITS | 1118/ V1811 | VISITS | VISITS | 111 S/ V1S1t | # 01 VISITS | Specify | VISITS | 111 S/ V1S11S |
| xxxxxx D | ay 1<br>Jeek | date9. | time5.t | ime5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | xxxxxx | xx | XX |
| : | | Done: specify | | | | | | | | | | | | | | |
| | Veek<br>52 | date9. | time5.t | ime5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XXXXXX | XX | XX |
| | ••• | | | | | | | | | | | | | | | |
| xxxxxx D | - | | time5.t | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XXXXXX | XX | XX |
| | /eek<br>26 | date9. | time5.t | ime5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XXXXXX | XX | XX |
| | Veek<br>52 | date9. | time5.t | ime5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XXXXXX | XX | XX |
| xxxxxx D | <br>ay 1 | date9. | time5.t | ime5. | xx | XX | XX | XX | XX | XX | XX | xx | XX | xxxxxx | XX | xx |
| | leek<br>26 | date9. | time5.t | ime5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | xxxxxx | XX | XX |
| | Veek<br>52 | date9. | time5.t | ime5. | XX | XX | XX | XX | XX | XX | XX | XX | XX | XXXXXX | XX | XX |
| | • • • | | | | | | | | | | | | | | | |

path\l\_program.sas date time

#### Listing 16.2.6.2.1 EQ-5D-5L Safety Population

| SubjectIDVis | Date Performed (Study sit Day) | Start<br>Time | End<br>Time | Mobility | Self-care | Usual Activities | Pain or<br>Discomfort | Anxiety/<br>Depression | Your<br>Health<br>Today |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxSci | reening date9. (xx) | time5. | time5. | problems in | I have no problems<br>washing or dressing<br>/myself/ I have sligh<br>problems, etc. | doing my usual | I have no pain or<br>discomfort/ I have<br>slight pain, etc. | I am not anxious or<br>depressed/ I am<br>slightly anxious, etc. | XX |
| We | eek 26 date9. (xx) | time5. | time5. | I have no problems in walking about | I have no problems<br>washing or dressing<br>/myself/ I have sligh<br>problems, etc. | doing my usual | I have no pain or<br>discomfort/ I have<br>slight pain, etc. | I am not anxious or<br>depressed/ I am<br>slightly anxious, etc. | XX |
| xxxxxxSci | reening date9. (xx) | time5. | time5. | problems in | I have no problems<br>washing or dressing<br>/myself/ I have sligh<br>problems, etc. | doing my usual | I have no pain or<br>discomfort/ I have<br>slight pain, etc. | I am not anxious or<br>depressed/ I am<br>slightly anxious, etc. | XX |
| We | eek 26 date9. (xx) | time5. | time5. | problems in | I have no problems<br>washing or dressing<br>/myself/ I have sligh<br>problems, etc. | doing my usual | I have no pain or<br>discomfort/ I have<br>slight pain, etc. | I am not anxious or<br>depressed/ I am<br>slightly anxious, etc. | XX |

Note: Study day is calculated as days since the date of first dose of study drug in 020. BP = Blood Pressure.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.

Programming Note: Repeat listing for the listings listed below

Listing 16.2.6.2.2 EQ-5D-5L, Patient Rated (Safety Population)
Listing 16.2.6.2.3 EQ-5D-5L, Caregiver Rated (Safety Population)

#### Listing 16.2.7.1 Adverse Events Safety Population

| | | Start | End | Start after last visit? | | | | Action<br>Taken<br>with | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Verbatim Term // | Date/Time | Date/Time | If Yes, Visit | | | Relationship | Study | Other | | |
| ID | Preferred Term | (Study Day) | (Study Day) | Date? | Serious | Severity | to Study Drug | Drug | Drug | Outcome | AESI |
| | | | | | | | | | | | · |
| XXXXXX | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | | | | | | |
| | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | • | - | | | | |
| | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | - | • | | | | |
| | | , | , | | | | | | | | |
| XXXXXX | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | - | • | | | | |
| | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | • | • | | | | |
| | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | J | 1 | | | | |
| | | ( ) | ( ) | | | | | | | | |
| XXXXXX | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | J | • | | | | |
| | Verbatim Term // | date9./time5. | date9./time5. | No/ | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | | | | т | | | | |
| | Verbatim Term // | date9./time5. | date9./time5. | Yes/Date9. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | (xx) | (xx) | 1 Co. Dates. | 1 25,110 | 22.21109 | | | | 5 <b>2.13</b> 6111 <b>6</b> | 1 25,110 |
| | Treferred Term | (1111) | (AA) | | | | | | | | |

<sup>\*</sup> Prior adverse event

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programmer note: sort by subject ID and onset date and resolution date within each subject.

<sup>#</sup> Pre-existing adverse event

<sup>&</sup>amp; Post-treatment adverse event

#### Listing 16.2.7.2.1 Serious Adverse Events Safety Population

| | | | | E 15 : | | | | Action | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| G 1. | 77 1 · | G | <b>a</b> | End Date | F 1 | | D 1 .: 1: | Taken | | | |
| Subject | Verbatim Term // | Start Date | Start | (Study | End | | Relationship | with Study | | | |
| ID | Preferred Term | (Study Day) | Time | Day) | Time | Severity | to Study Drug | Drug | Other Drug | Outcome | AESI |
| XXXXXX | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | | | | | | | | | | |
| | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | | | | | | | | | | |
| | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | | | | | • | - | | | | |
| xxxxxx | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | | | , , | | • | • | | | | |
| | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | . , | | . , | | • | • | | | | |
| | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | - ( ) | | - ( ) | | , | 1 | | | | |
| xxxxxx | Verbatim Term // | date9. (xx) | time5. | date9. (xx) | time5. | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | Gares (1111) | | . (1111) | | 20.01109 | remaining | | | | 1 00,110 |
| | Verbatim Term // | date9. (xx) | time5 | date9 (xx) | time5 | severity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | auto). (AA) | minos. | auco, (AA) | times. | Se . Silty | retationship | action | action | carcome | 1 55,110 |
| | Verbatim Term // | date9. (xx) | time5 | date0 (vv) | time5 | ceverity | relationship | action | action | outcome | Yes/No |
| | Preferred Term | uaic). (XX) | unics. | uaic). (XX) | unics. | severity | relationship | action | action | outcome | 1 05/110 |
| | Ficiented Term | | | | | | | | | | |

<sup>\*</sup> Prior adverse event

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l program.sas date time

Programmer note: sort by subject ID and onset date and resolution date within each subject

Programmer note: Repeat listing for the following:

Listing 16.2.7.2.2 Fatal Adverse Events (Safety Population)

Listing 16.2.7.2.3 Non-Fatal Serious Adverse Events (Safety Population)

<sup>#</sup> Pre-existing adverse event

<sup>&</sup>amp; Post-treatment adverse event

Listing 16.2.7.2.4
Serious Adverse Events (Additional Information About the SAE Collected on the AE CRF)
Safety Population

| | | | | | | | | Did the SAE | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Result | Date of |
| | | | Hospital | Hospital | | | Autopsy | in Death? | Death |
| Subject | Verbatim Term // | TT 1. 11 .1 | Admission Date | Discharge | Death Certificate | Autopsy | Report | | (Study |
| ID | Preferred Term | Hospitalization | (Study Day) | Date (Study Day) | Available | Performed | Obtained | | Day) |
| xxxxxx | Verbatim Term //<br>Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Verbatim Term // | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Preferred Term | | | | | | | | |
| xxxxxx | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | V 1 4 T // | N/ /NI | D 4 0 | D 4 0 | N7 /N1 | 37 /NI | X7 /X1 | 37 /NI | D 4 0 |
| XXXXXX | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |
| | Verbatim Term // Preferred Term | Yes/No | Date9. | Date9. | Yes/No | Yes/No | Yes/No | Yes/No | Date9. |

path\l program.sas date time

Programmer note: sort by subject ID and onset date and resolution date within each subject

<sup>\*</sup> Prior adverse event

<sup>#</sup> Pre-existing adverse event

<sup>&</sup>amp; Post-treatment adverse event

Listing 16.2.7.2.5
Serious Adverse Events (Collected on the SAE CRF)
Safety Population

| | D | | <b>D</b> 1 | If Yes, | 3 | | |
|---|---|---|---|---|---|---|---|
| | | 5.1 | | | SAE? | | |
| | _ | | • | Description | | | Summary |
| Preferred Term | (Study Day) | Reported? | Tests Done? | | | SAE | |
| Verbatim Term //<br>Preferred Term | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxx | Yes/No | date9. | |
| Verbatim Term // | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| Preferred Term | | | | | | | |
| Verbatim Term // | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| Preferred Term | - ( ) | | | | | | |
| Verbatim Term // | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| Preferred Term | - ( ) | | | | | | |
| Verbatim Term // | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| Preferred Term | · / | | | | | | |
| Verbatim Term // | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| | - ( ) | | | | | | |
| Verbatim Term // | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxx | Yes/No | date9. | |
| | | 1 10 | 2 23/110 | | 2 23/110 | | |
| | date9. (xx) | Yes/No | Yes/No | xxxxxxxxxxxxx | Yes/No | date9. | |
| | antes, (AA) | 1 25/110 | 1 23/110 | | 23/110 | aate). | |
| | Verbatim Term // Preferred Term Verbatim Term // Preferred Term Verbatim Term // Preferred Term Verbatim Term // Preferred Term Verbatim Term // Preferred Term Verbatim Term // Preferred Term Verbatim Term // | Preferred Term (Study Day) Verbatim Term // date9. (xx) Preferred Term Verbatim Term // date9. (xx) | Verbatim Term // Report Relevant Lab Reported? Verbatim Term // date9. (xx) Yes/No Preferred Term Verbatim Term // date9. (xx) Yes/No | Verbatim Term // Preferred TermReport (Study Day)Relevant Lab Reported?Confirmatory Tests Done?Verbatim Term // Preferred Termdate9. (xx)Yes/NoYes/NoVerbatim Term // Preferred TermYes/NoYes/NoYes/No | Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Verbatim Term // Report (Study Day) Relevant Lab Confirmatory Tests Done? Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXX Yes/No Preferred Term Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXXX Yes/No Preferred Term Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXXX Yes/No Preferred Term Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXXX Yes/No Preferred Term Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXXX Yes/No Preferred Term Verbatim Term // date9. (xx) Yes/No Yes/No XXXXXXXXXXXXX Yes/No Preferred Term | Date of Initial Verbatim Term // Report Relevant Lab Preferred Term (Study Day) Reported? Tests Done? Description SAE? Dose Prior to SAE Verbatim Term // date9. (xx) |

<sup>\*</sup> Prior adverse event

path\l program.sas date time

Programmer note: sort by subject ID and onset date and resolution date within each subject

<sup>#</sup> Pre-existing adverse event

<sup>&</sup>amp; Post-treatment adverse event

Listing 16.2.7.3.1

Adverse Events Leading to Dose Reduction, Interruption or Study Drug Withdrawal Safety Population

| Subject<br>ID | Verbatim Term //<br>Preferred Term | Start Date<br>(Study Day) | Start<br>Time | End Date (Study Day) | End<br>Time | Serious | Severity | Relationship to Study Drug | Action Taken<br>with Study<br>Drug | Other Drug | Outcome | AESI |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - 10 | Treferred Term | (Study Duy) | | (Study Day) | Time | Scrious | Beventy | Drug | Diug | Other Drug | Outcome | TIESI |
| xxxxxx | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| xxxxxx | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| xxxxxx | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| xxxxxx | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term //<br>Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |
| | Verbatim Term // Preferred Term | date9. (xx) | time5. | date9. (xx) | time5. | Yes/No | severity | relationship | action | action | outcome | Yes/No |

<sup>\*</sup> Prior adverse event

path\l program.sas date time

Programmer note: sort by subject ID and onset date and resolution date within each subject. Repeat listing for

<sup>#</sup> Pre-existing adverse event

<sup>&</sup>amp; Post-treatment adverse event

Listing 16.2.7.3.2 All AEs for Subjects with Adverse Events Leading to Dose Reduction, Interruption or Study Drug Withdrawal (Safety Population) {Programmer note: Please present the AE leading to dose reduction, interruption or study drug withdrawal along with all AEs for that subject.}

#### Listing 16.2.7.4 Adverse Events of Special Interest Safety Population

| Subject | Verbatim Term // Preferred | Start Date | Start | End Date | End | Relationship to Study | Action<br>Taken<br>with Study | _ | |
|---|---|---|---|---|---|---|---|---|---|
| ID | Term | (Study Day) | Time | (Study Day) | Time Serious Severity | Drug | Drug | Other Drug | Outcome |
| | 101111 | (Study Duy) | 111110 | (Study Buy) | Time Serious Severity | Diag | Drug | Other Drug | Guiconie |
| xxxxxx | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| xxxxxx | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| xxxxxx | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |
| | Verbatim Term // Preferred<br>Term | date9. (xx) | time5. | date9. (xx) | time5. Yes/No severity | relationship | action | action | outcome |

<sup>\*</sup> Prior adverse event

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programmer note: sort by subject ID, onset date and resolution date within each subject.

<sup>#</sup> Pre-existing adverse event

<sup>&</sup>amp; Post-treatment adverse event

## Listing 16.2.8.1.1 Central Laboratory Normal Ranges Safety Population

| | | | Convention | onal Units | SI Unit | ts |
|---|---|---|---|---|---|---|
| Laboratory Test | Gender | Age Range | Normal Range | Unit | Normal Range | Unit |
| WBC | Female<br>Male | min-max<br>min-max | min-max<br>min-max | | min-max<br>min-max | |
| Hematocrit | Female<br>Male | min-max<br>min-max | min-max<br>min-max | | min-max<br>min-max | |
| Hemoglobin<br> | Female<br>Male | min-max<br>min-max | min-max<br>min-max | | min-max<br>min-max | |
| TSH<br> | Female<br>Male | min-max<br>min-max | min-max<br>min-max | | min-max<br>min-max | |

path\l\_program.sas date time

**Listing 16.2.8.1.2** Central Laboratory - Comments on Samples Not Analyzed **Safety Population** 

| Subject<br>ID | Visit | Collection<br>Date<br>(Study Day) | Collection<br>Time | Laboratory<br>Panel | Laboratory Test | Comments |
|---|---|---|---|---|---|---|
| XXXXXX | Baseline | date9. (xx) | time5. | Hematology | XXXXX | XXXXX |
| | Week 2 | date9. (xx) | time5. | Hematology | XXXXX | XXXXX |
| | Week 13 | date9. (xx) | time5. | Chemistry | XXXXX | XXXXX |
| XXXXXX | Baseline | date9. (xx) | time5. | XXXXX | XXXXX | XXXXX |
| | Week 2 | date9. (xx) | time5. | XXXXX | XXXXX | xxxxx |
| | Week 13 | date9. (xx) | time5. | XXXXX | XXXXX | xxxxx |
| | | ` ' | | | | |
| XXXXXX | Baseline | date9. (xx) | time5. | xxxxx | xxxxx | xxxxx |
| | Week 2 | date9. (xx) | time5. | XXXXX | XXXXX | XXXXX |
| | Week 13 | date9. (xx) | time5. | xxxxx | xxxxx | xxxxx |
| | | · / | | | | |
| XXXXXX | Baseline | date9. (xx) | time5. | xxxxx | xxxxx | xxxxx |
| | Week 2 | date9. (xx) | time5. | xxxxx | xxxxx | xxxxx |
| | Week 13 | date9. (xx) | time5. | XXXXX | XXXXX | XXXXX |
| | | - (-mi) | | | | |

Programming note: Display the CRF visit label.

Listing 16.2.8.2.1
Central Lab - Hematology - Conventional Units
Safety Population
Part 1 of 2

| Subject<br>ID | Sex | Age | Visit | Collection<br>Date<br>(Study Day) | Collection<br>Time | Neutro-<br>phils<br>(10 <sup>3</sup> /uL) | Lympho-<br>cytes<br>(10 <sup>3</sup> /uL) | Monocytes (10 <sup>3</sup> /uL) | Baso-<br>phils<br>(10 <sup>3</sup> /uL) | Eosino-<br>phils<br>(10³/uL) | WBC (10 <sup>3</sup> /uL) | RBC<br>(10 <sup>6</sup> /uL) | Platelets (10 <sup>3</sup> /uL) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | M/F | xx | Baseline<br>Week 2<br>Week 13 | date9. (xx) | time5.<br>time5. | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |
| xxxxxx | M/F | XX | Baseline<br>Week 2<br>Week 13 | date9. (xx) | time5.<br>time5. | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |
| xxxxxx | M/F | xx | Baseline<br>Week 2<br>Week 13 | date9. (xx)<br>date9. (xx) | time5.<br>time5. | XX.XX<br>XX.XX<br>XX.XX | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |
| xxxxxx | M/F | xx | Baseline<br>Week 2<br>Week 13 | date9. (xx)<br>date9. (xx) | time5.<br>time5. | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.


#### Listing 16.2.8.2.1 Central Lab - Hematology - Conventional Units Safety Population Part 2 of 2

| Visit | Collection<br>Date<br>(Study Day) | Collection<br>Time | MCV<br>(fl) | MCH<br>(pg) | MCHC<br>(g/dL) | Hemoglobin<br>(g/dL) | Hema-<br>tocrit<br>(%) | Reticulocytes (%) |
|---|---|---|---|---|---|---|---|---|
| Week 2 | date9. (xx)<br>date9. (xx) | time5. | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX |
| Baseline<br>Week 2 | date9. (xx)<br>date9. (xx) | time5. | XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |
| <br>Baseline | date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5. | xx.xx<br>xx.xx<br>xx.xx | xx.xx<br>xx.xx<br>xx.xx | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | xx.xx<br>xx.xx<br>xx.xx | xx.xx<br>xx.xx<br>xx.xx |
| | date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5. | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | xx.xx<br>xx.xx<br>xx.xx | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |
| | Baseline Week 2 Week 13 Baseline Week 2 Week 13 Baseline Week 2 Week 13 Baseline | Date Visit | Date Collection | Date Collection MCV | Date Visit Collection (Study Day) MCV (fl) MCH (pg) Baseline date9. (xx) time5. xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx Baseline date9. (xx) time5. xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx Baseline date9. (xx) time5. xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx Baseline date9. (xx) time5. xx.xx xx.xx | Date Collection MCV MCH MCHC Visit (Study Day) Time (fl) (pg) (g/dL) Baseline date9. (xx) time5. xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. | Date Visit Collection (Study Day) MCV (fl) MCH (pg) MCHC (g/dL) Hemoglobin (g/dL) Baseline date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 2 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Week 13 date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx Baseline date9. (xx) time5. xx.xx xx.xx xx.xx xx.xx | Date Collection MCV MCH MCHC Hemoglobin tocrit |

Note: L=Low, H=High; \*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.

Repeat for Listing 16.2.8.2.2 Central Lab - Hematology - SI Units (Safety Population)

Part 1 of 2

Listing 16.2.8.2.3

Local Lab – Hematology - Conventional Units

Safety Population

| | | Collection | | | | | | | | | | Reticul- | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date | Collection | Hemat- | Hemo- | | | | Reticulocyte | | Erythrocytes | ocyte | | Neutro- |
| ID | Visit | (Study Day) | Time | ocrit | globin N | MCH | MCHC | RBC | (Count) | Heinz Bodies | w/ Heinz Bodies | (%) | WBC | phils (%) |
| XXXXXX | Baseline | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX |
| | Week 13 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | XX.XX | XX.XX X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note; L=Low, H=High; \*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

TRx-237-020

#### Listing 16.2.8.2.3 Local Lab - Hematology - Conventional Units **Safety Population** Part 2 of 2

| Subject<br>ID | Visit | Collection<br>Date<br>(Study Day) | Collection<br>Time | Neutro-<br>phils<br>(abs) | Lymph-<br>ocytes<br>(%) | Lymph-<br>ocytes<br>(abs) | Mono-<br>cytes<br>(%) | Mono-<br>cytes<br>(abs) | Eosino-<br>phils<br>(%) | Eosino-<br>phils<br>(abs) | Baso-<br>phils<br>(%) | Baso-<br>phils<br>(abs) | Platelets | MCV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | Baseline<br>Week 2<br>Week 13 | date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5.<br>time5. | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX | XX.XX<br>XX.XX<br>XX.XX |

Note; L=Low, H=High; \*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.

Repeat for Listing 16.2.8.2.4 Local Lab - Hematology - SI Units (Safety Population)
# Listing 16.2.8.3.1 Central Lab - Serum Chemistry - Conventional Units Safety Population Part 1 of 3

| | | | | Collection | n | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Date | | ALT | AST | Alkaline | | | | Total | | |
| Subject | ~ | | *** | (Study | Collection | (SGPT) | | Phosphatase | | | | | | |
| ID | Sex | Age | Visit | Day) | Time | (U/L) | (U/L) | (U/L) | (U/L) | (g/dL) | (g/dL) | (g/dL) | (mEq/L) | (mEq/L) |
| xxxxxx | M/F | xx | Baseline | date9. | time5. | xxx | xxx | XXX | xxx | x.x | X.X | x.x | xxx | X.X |
| | | | Week 2 | date9. | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XXX | X.X |
| | | | Week 13 | date9.<br>(xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XXX | X.X |
| xxxxxx | M/F | XX | Baseline | date9. (xx) | time5. | XXX | XXX | xxx | XXX | X.X | X.X | x.x | XXX | X.X |
| | | | Week 2 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XXX | X.X |
| | | | Week 13 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XXX | x.x |
| xxxxxx | M/F | XX | Baseline | date9. (xx) | time5. | XXX | xxx | xxx | xxx | x.x | X.X | x.x | xxx | X.X |
| | | | Week 2 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | x.x | XXX | X.X |
| | | | Week 13 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XXX | X.X |
| xxxxxx | M/F | XX | Baseline | date9. (xx) | time5. | XXX | xxx | xxx | xxx | x.x | X.X | x.x | xxx | X.X |
| | | | Week 2 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | X.X | XXX | X.X |
| | | | Week 13 | date9.<br>(xx) | time5. | XXX | XXX | XXX | XXX | X.X | X.X | x.x | XXX | X.X |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l program.sas date time

### Page 2 of x

# Listing 16.2.8.3.1 Central Lab - Serum Chemistry - Conventional Units Safety Population Part 2 of 3

| Subject<br>ID | Visit | Collection Date (Study | | Total<br>Bilirubin | Direct<br>Bilirubin | Indirect<br>Bilirubin | Urea Nit-<br>rogen | Creatinine<br>(Rate<br>Blanked) | Creatinine<br>Clearance (ml/min) | eGFR<br>mL/min/1.73<br>m <sup>2</sup> ) | Creatine<br>Kinase |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | VISIT | Day) | Time | (mg/dL) | (mg/dL) | (mg/dL) | (mg/dL) | (mg/dL) | (1111/111111) | 111 ) | (U/L) |
| xxxxxx | Baseline<br>Week 2 | date9. (xx)<br>date9. (xx) | time5. | X.X<br>X.X | X.X<br>X.X | x.x<br>x.x | XX<br>XX | X.X<br>X.X | X.X<br>X.X | X.X<br>X.X | X.X<br>X.X |
| | Week 13 | date9. (xx) | time5. | X.X | X.X | X.X | XX | X.X | X.X | X.X | X.X |
| xxxxxx | Baseline<br>Week 2<br>Week 13 | date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5.<br>time5. | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | xx<br>xx<br>xx | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X |
| XXXXXX | Baseline | date9. (xx) | time5. | X.X | X.X | x.x | XX | X.X | X.X | X.X | X.X |
| | Week 2 | date9. (xx) | time5. | X.X | X.X | X.X | XX | X.X | X.X | X.X | X.X |
| | Week 13 | date9. (xx) | time5. | X.X | X.X | X.X | XX | X.X | X.X | X.X | X.X |
| xxxxxx | Baseline<br>Week 2<br>Week 13 | date9. (xx)<br>date9. (xx)<br>date9. (xx) | time5.<br>time5.<br>time5. | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | xx<br>xx<br>xx | X.X<br>X.X<br>X.X | x.x<br>x.x<br>x.x | x.x<br>x.x<br>x.x | X.X<br>X.X<br>X.X |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

#### Listing 16.2.8.3.1 Central Lab - Serum Chemistry - Conventional Units Safety Population Part 3 of 3

| | | | ( | Collection | n | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Date | | | | Calcium | | | Triglyceride | S | | Uric |
| Subject | | | | (Study | Collection | nChloride I | Phosphorus | s (EDTA) | Glucose | LDH | (GPO) | Cholesterol(HP | ) Folate | Acid |
| ID | Sex | Age | Visit | Day) | Time | (mEq/L) | (mg/dL) | (mg/dL) | (mg/dL) | (U/L) | (mg/dL) | (mg/dL) | (ng/mL) | (mg/dL) |
| • | | | | | | | | | | | | | | |
| XXXXXX | M/F | XX | Baseline | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | Week 2 | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | Week 13 | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| xxxxxx | M/F | XX | Baseline | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | Week 2 | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | Week 13 | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | | () | | | | | | | | | | |
| xxxxxx | M/F | XX | Baseline | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | Week 2 | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | (xx) | | | | | | | | | | |
| | | | Week 13 | date9. | time5. | XXX | X.X | XX.X | XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | WCCK 13 | (xx) | unics. | AAA | AA | AAA | MAA | AAA | AA.A | AA.A | AAA | AAA |
| | | | | (AA) | | | | | | | | | | |

Note: L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.

Repeat for Listing 16.2.8.3.2 Central Lab – Serum Chemistry - SI Units (Safety Population)

TRx-237-020

## Listing 16.2.8.3.3 Local Lab – Serum Chemistry - Conventional Units Safety Population Part 1 of 3

| | | Collection | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date ( | Collectio | n | | | Hapto- | | | | | |
| ID | Visit | (Study Day) | Time | Fasting? TSH Free T3 | Free T4 | Vitamin B12 | 2Folate globin G6P | DSodium | Potassiun | ıCalcium | Albumin | Total Protein |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | X XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | X XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | X XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No xx.xx xx.xx | XX.XX | XX.XX | XX.XX XX.XX XX.X | x xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |

Note; L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

## Listing 16.2.8.3.3 Local Lab – Serum Chemistry - Conventional Units Safety Population Part 2 of 3

| Subject | | Collection<br>Date | Collection | | Blood Urea | | | | Indirect | | | | | Glucose<br>(not |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | Visit | (Study Day) | Time | Fasting? | Nitrogen | Urea | Bilirubin | Bilirubii | ıBilirubinl | Phosphatase | LDH | GGT ALT | AST | fasted) |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX XX.XX | XX.XX | XX.XX |

Note; L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Listing 16.2.8.3.3 Local Lab - Serum Chemistry - Conventional Units **Safety Population** 

### Part 3 of 3

| | | Collection<br>Date | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | (Study | Collection | | | Creatinine | | C | holester | ol Uric | | | Methylmalor | nic |
| ID | Visit | Day) | Time | Fasting? | Creatinin | eClearance | Phosphate | Triglycerides | (total) | Acid Chloride | Digoxin | Homocysteine | e Acid | Others |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | , , | | | | | | | | | | | | |

Note; L=Low, H=High; \*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.

Repeat for Listing 16.2.8.3.4 Local Lab – Serum Chemistry - SI Units (Safety Population)

TRx-237-020

## Listing 16.2.8.4.1 Local Lab – Urinalysis - Conventional Units Safety Population Part 1 of 3

| | | Collection | | | | | | | | 6 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 0.11 | | Date | G 11 4: | | | c .c | HTD.C | TT 1 | | Squamous | NT 6 | | |
| Subject | | (Study | Collection | | | Specific | WBC | Hyaline | Unclassified | Epitheial | Non-Squamaus | | |
| ID | Visit | Day) | Time | Fasting? | RBC WB | C Gravity | Clumps | Casts | Casts | Cells | Epithelial Cells | Bacteria | Yeast |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX XX.X | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | xx.xx xx.x | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note; L=Low, H=High;\*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label. Only display parameters with at least one result.

TRx-237-020

#### Listing 16.2.8.4.1 Local Lab - Urinalysis - Conventional Units **Safety Population** Part 2 of 3

| | | Collection | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date | Collection | | | | | | | | | |
| ID | Visit | (Study Day) | Time | Fasting? | Crystals | Mucus | Sperm | pН | Glucose | Ketones | Protein | Bilirubin |
| • | | | | | | | | | | | | |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note; L=Low, H=High; \*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label. Only display parameters with at least one result.

## Listing 16.2.8.4.1 Local Lab – Urinalysis - Conventional Units Safety Population Part 3 of 3

| Subject | TT. 14 | Collection<br>Date | Collection | T. (' 0 | DI I | 3777 | ** 131 | 6.1 | m 1:12 | 0.1 |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Visit | (Study Day) | Time | Fasting? | Blood | Nitrites | Urobilinogen | Color | Turbidity | Others |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XXXXXX | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | , , | | | | | | | | |
| xxxxxx | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | . , | | | | | | | | |
| xxxxxx | Baseline | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 2 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Week 13 | date9. (xx) | time5. | Yes/No | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | · / | | | | | | | | |

Note; L=Low, H=High; \*=Potentially Clinically Significant; #=Abnormal/Clinically Significant per Investigator. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label. Only display parameters with at least one result.

Repeat for Listing 16.2.8.4.2 Local Lab - Urinalysis - SI Units (Safety Population)

### Listing 16.2.8.5.1 Hematology Results of Potential Clinical Significance – Conventional Units Safety Population

#### Collection Date

| | | | | Conection Date | • | |
|---|---|---|---|---|---|---|
| Subject ID | Laboratory Test (unit) | Criteria | Visit | (Study Day) | Collection Time | Results |
| XXXXXX | test (unit) | Criteria | Baseline | date9. (xx) | time5. | result |
| | test (unit) | Criteria | Week 2 | date9. (xx) | time5. | result |
| | test (unit) | Criteria | Week 13 | date9. (xx) | time5. | result |
| XXXXXX | test (unit) | Criteria | Baseline | date9. (xx) | time5. | result |
| | test (unit) | Criteria | Week 2 | date9. (xx) | time5. | result |
| | test (unit) | Criteria | Week 13 | date9. (xx) | time5. | result |
| XXXXXX | test (unit) | Criteria | Baseline | date9. (xx) | time5. | result |
| | test (unit) | Criteria | Week 2 | date9. (xx) | time5. | result |
| | test (unit) | Criteria | Week 13 | date9. (xx) | time5. | result |

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\1 program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.

#### Repeat this listing for:

Listing 16.2.8.5.2 Hematology Results of Potential Clincial Significance - SI Units (Safety Population)

Listing 16.2.8.5.3 Hematology Results of Potential Clincial Significance - Includes Only Hgb and Hct reticulocy (Safety Population): If either RBC or Hgb meets PCS for any visit, then both labs values for all visits will be required in format of Listing 16.2.6.2.1.

Listing 16.2.8.5.4 Hematology Results of Potential Clincial Significance - WBCs and Neutrophils (Safety Population): If either parameter meets PCS for any visit, then the values for all visits are required, in format of Listing 16.2.6.2.1

Listing 16.2.8.5.5 Hematology Results of Potential Clincial Significance – Eosinophils (Safety Population)

Listing 16.2.8.5.6 Hematology Results of Potential Clincial Significance – Platelets (Safety Population)

Listing 16.2.8.6.1 Serum Chemistry Results of Potential Clinical Significance – Conventional Units (Safety Population)

Listing 16.2.8.6.2 Serum Chemistry Results of Potential Clinical Significance – SI Units (Safety Population)

Listing 16.2.8.6.3 Serum Chemistry Results of Potential Clinical Significance - Urea (Nitrogen) or Creatinine (Safety Population): If either parameter meets PCS for any visit, then Urea (Nitrogen), Creatinine, plus Creatinine Clearance and eGFR are required for all visits, in format of Listing 16.2.6.3.1

Listing 16.2.8.6.4 Serum Chemistry Results of Potential Clinical Significance - ALT, AST, GGT, bilirubin, alkaline phosphatase (Safety Population): If any of one of these parameters meets PCS, display the results for all 4 parameters.

Listing 16.2.9.1 Vital Signs Safety Population

| Subject<br>ID | Visit | Date of<br>Measurement<br>(Study Day) | Time of<br>Measurement | Temperature<br>(°C) | Temperature<br>Method | SBP<br>(mmHg) | DBP<br>(mmHg) | Pulse<br>(beats/min) | Weight<br>(kg) | Any<br>Findings<br>Abnormal? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | Baseline | date9. (xx) | time5. | XX.X. | xxx.x | xx.x | xx | xxx | xxx | Yes:<br>CS/NCS / |
| | Week 2 | date9. (xx) | time5. | | xxx.x | xx.x | xx | xxx | xxx | No<br>Yes:<br>CS/NCS / |
| | Week 13 | date9. (xx) | time5. | | xxx.x | XX.X | XX | xxx | xxx | No<br>Yes:<br>CS/NCS /<br>No |
| xxxxxx | Baseline | date9. (xx) | time5. | XX.X. | xxx.x | XX.X | XX | xxx | xxx | Yes:<br>CS/NCS / |
| | Week 2 | date9. (xx) | time5. | | xxx.x | xx.x | XX | xxx | xxx | No<br>Yes:<br>CS/NCS / |
| | Week 13 | date9. (xx) | time5. | | xxx.x | xx.x | xx | xxx | XXX | No<br>Yes:<br>CS/NCS /<br>No |
| xxxxxx | Baseline | date9. (xx) | time5. | XX.X. | xxx.x | xx.x | XX | xxx | xxx | Yes:<br>CS/NCS / |
| | Week 2 | date9. (xx) | time5. | | xxx.x | xx.x | xx | xxx | xxx | No<br>Yes:<br>CS/NCS / |
| | Week 13 | date9. (xx) | time5. | | xxx.x | XX.X | XX | xxx | xxx | No<br>Yes:<br>CS/NCS /<br>No |

Note: CS= Clinically Significant; NCS = Not Clinically Significant; \*=Potentially Clinically Significant. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

#### Listing 16.2.9.2.1 Vital Sign Results of Potential Clinical Significance Safety Population

| Subject ID | Parameter (unit) | Criteria | Target<br>Visit | Collection Date<br>(Study Day) | Collection Time | Results |
|---|---|---|---|---|---|---|
| xxxxxx | Temperature (°C) | criteria | Baseline<br>Week 2 | date9. (xx) | time5. | result |
| | SBP (mmHg) | criteria | Baseline<br>Week 2 | date9. (xx) | time5. | result |
| xxxxxx | Temperature (°C) | criteria | Baseline<br>Week 2 | date9. (xx) | time5. | result |
| | SBP (mmHg) | criteria | Baseline<br>Week 2 | date9. (xx) | time5. | result |
| XXXXXX | Temperature (°C) | criteria | Baseline<br>Week 2 | date9. (xx) | time5. | result |
| | SBP (mmHg) | criteria | Baseline<br>Week 2 | date9. (xx) | time5. | result |

Note: CS= Clinically Significant; NCS = Not Clinically Significant. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID.

### Listing 16.2.9.2.2 Subjects with Potentially Clinically Significant Vital Sign Results Safety Population

| Subject ID | Parameter (unit) | Target<br>Visit | Collection Date<br>(Study Day) | Collection Time | Results |
|---|---|---|---|---|---|
| xxxxxx | Temperature (°C) | Week 2 | date9. (xx) | time5. | result |
| | SBP (mmHg) | Baseline | date9. (xx) | time5. | result |
| xxxxxx | Temperature (°C) | Week 2 | date9. (xx) | time5. | result |
| | SBP (mmHg) | Baseline | date9. (xx) | time5. | result |
| xxxxxx | Temperature (°C) | Week 2 | date9. (xx) | time5. | result |
| | SBP (mmHg) | Baseline | date9. (xx) | time5. | result |

Note: \*=Potentially Clinically Significant. Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Programming note: Sort by subject ID. Listing will include all vital sign results for those parameters and subjects that have one or more results that meet criteria.

#### Listing 16.2.9.2.3 Respiratory Rate Safety Population

| Subject<br>ID | | | Respiratory Rate t(breaths per min) |
|---|---|---|---|
| xxxxxx | Baseline date9. (xx)<br>Week 2 date9. (xx) | time5. | xx.x. |
| | Week 2 date9. (xx) Week 13 date9. (xx) | time5. | |
| xxxxxx | Baseline date9. (xx) Week 2 date9. (xx) Week 13 date9. (xx) | time5.<br>time5.<br>time5. | xx.x. |
| xxxxxx | Baseline date9. (xx) Week 2 date9. (xx) Week 13 date9. (xx) | time5.<br>time5.<br>time5. | XX.X. |

Note: Study day is calculated as days since the date of first dose of study drug in 020.

path\l\_program.sas date time

Listing 16.2.9.3 Pregnancy Test Safety Population

| | | | Date of | |
|---------|----------|-----------|-------------|-------------------|
| Subject | | | Collection | |
| ID | Visit | Performed | (Study Day) | Result |
| XXXXXX | Baseline | Yes/No | date9. (xx) | Negative/Positive |
| | Week 2 | Yes/No | date9. (xx) | Negative/Positive |
| | Week 13 | Yes/No | date9. (xx) | Negative/Positive |
| | | | | - |
| XXXXXX | Baseline | Yes/No | date9. (xx) | Negative/Positive |
| | Week 2 | Yes/No | date9. (xx) | Negative/Positive |
| | Week 13 | Yes/No | date9. (xx) | Negative/Positive |
| | | | ` ´ | |
| XXXXXX | Baseline | Yes/No | date9. (xx) | Negative/Positive |
| | Week 2 | Yes/No | date9. (xx) | Negative/Positive |
| | Week 13 | Yes/No | date9. (xx) | Negative/Positive |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

#### Listing 16.2.9.4 Physical Examination Safety Population

| | | Visit | | | | |
|---|---|---|---|---|---|---|
| Subject | | Date | | | | Clinically |
| ID | Visit | (Study Day) | Body System | Overall Assessment | Description of Abnormality | Significant |
| XXXXXX | Baseline | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | Week 2 | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | Week 13 | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | . , | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | ••• | | | | | |
| XXXXXX | Baseline | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | Week 2 | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | . , | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal | Description | Yes/No |
| | Week 13 | date9. (xx) | Body System 1 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal | Description | Yes/No |
| | | | Body System 2 Body System 3 | Normal/Abnormal | Description | Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

#### Listing 16.2.9.5 Neurological Examination Safety Population

| 0.1. | | Visit | | | | C1: : 11 |
|---|---|---|---|---|---|---|
| Subject | *** | Date | D 1 6 | <b>a</b> | 5 | Clinically |
| ID | Visit | (Study Day) | Body System | Status | Description of Abnormality | Significant |
| | Baseline | data() (vvv) | Dodry Crystam 1 | Name of Alexander of Alexand | Description | Yes/No |
| XXXXXX | Daseillie | date9. (xx) | Body System 1 | Normal/Abnormal/Absent | | |
| | | | Body System 2 | Normal/Abnormal/Absent | • | Yes/No |
| | | | Body System 3 | Normal/Abnormal/Absent | Description | Yes/No |
| | Week 2 | date9. (xx) | Body System 1 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal/Absent | • | Yes/No |
| | | | Body System 3 | Normal/Abnormal/Absent | | Yes/No |
| | | | Body System 5 | 1 tollian / tollollian / toselit | Description | 1 65/110 |
| | Week 13 | date9. (xx) | Body System 1 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal/Absent | • | Yes/No |
| xxxxxx | Baseline | date9. (xx) | Body System 1 | Normal/Abnormal/Absent | Description | Yes/No |
| ALL LANGE | Визение | dates. (AA) | Body System 2 | Normal/Abnormal/Absent | • | Yes/No |
| | | | Body System 2 Body System 3 | Normal/Abnormal/Absent | | Yes/No |
| | | | Body System 5 | Tvorman/Tvonorman/Tvosent | Description | 1 65/140 |
| | Week 2 | date9. (xx) | Body System 1 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal/Absent | Description | Yes/No |
| | Week 13 | date9. (xx) | Body System 1 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 2 | Normal/Abnormal/Absent | Description | Yes/No |
| | | | Body System 3 | Normal/Abnormal/Absent | Description | Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time

#### Listing 16.2.9.6 Serotonin Toxicity Assessment Safety Population Part 1 of 3

| | | | | | Autonomic Findings | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date Performed | Start | End | Rater's | Diaph- I | | Pyrexia/ | | Dyspnea/ | | |
| ID | Visit | (Study Day) | Time | Time | Initials | Shivering | oresis | Diarrhea | Fever | Tachycardia | Tachypnea | Seated BP |
| XXXXXX | Screening | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | | | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXXXXX | Screening | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | | | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXXXXX | Screening | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | | | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXXXXX | Screening | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | date9. (xx) | time5. | time5. | XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug. BP = Blood Pressure.

path\l\_program.sas date time

#### Listing 16.2.9.6 Serotonin Toxicity Assessment Safety Population Part 2 of 3

| | | | Neuromuscular Changes | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Visit | Myo-<br>clonus | Tremor at rest | Mydri-<br>asis | Nystag-<br>mus | Clonus | Hyper-<br>reflexia | Hyper-<br>tonia | Dizzi-<br>ness | Incoord-<br>ination |
| xxxxxx | Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXXXXX | Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXXXXX | Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXXXXX | Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug. BP = Blood Pressure.

path\l\_program.sas date time

#### Listing 16.2.9.6 Serotonin Toxicity Assessment Safety Population Part 3 of 3

Mental State/Other CNS Changes

| Visit | Delirium | Agitation/<br>Akathisia | Elevated<br>Mood | Insomnia | Any Additional Findings |
|---|---|---|---|---|---|
| Si | | | | | |
| Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Screening | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Week 26 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | Screening Week 26 Screening Week 26 Screening Week 26 Screening | Screening Yes/No Week 26 Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Screening Yes/No Screening Yes/No Yes/No Yes/No | Visit Delirium Akathisia Screening Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Screening Yes/No Yes/No | Visit Delirium Akathisia Mood Screening Yes/No Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No | Visit Delirium Akathisia Mood Insomnia Screening Yes/No Yes/No Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Week 26 Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Yes/No Screening Yes/No Yes/No Yes/No Yes/No |

Note: Study day is calculated as days since the date of first dose of study drug. BP = Blood Pressure.

path\l\_program.sas date time

#### **Listing 16.2.9.7** Mini-Mental State Examination (MMSE) **Safety Population** Part 1 of 3

| | | | | | | Orientation to Time | | | | | Orientation to Place | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | What is | | | | |
| | | | | | | | | the | What is | | | |
| | | Date | | | | What | What is | month | the day | What | What is the | What is the |
| Subject | | Performed | | | Rater's | is the | the | of the | of the | is the | state | country (or |
| IĎ | Visit | (Study Day) | Start Time | End Time | Initials | year? | season? | year? | week? | date? | (province)? | city/town?) |
| XXXXXX | Screening | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | Week 26 | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| xxxxxx | Screening | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | Week 26 | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | | 1 . 0 | | | | 0.14 | 0.14 | 0.44 | 0.11 | 0.14 | 0.44 | 0.44 |
| XXXXXX | 0 | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | Week 26 | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| xxxxxx | Screening | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | Week 26 | date9. (xx) | time5. | time5. | XX | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label. Include data collected from both the MMSE and MMSE W/O World Backwards CRF pages.

 $<sup>^{[1]}</sup>$  'N/A' is displayed if the version of the MMSE used did not include this question.  $^{[2]}$  Calculated total score may include imputation of missing items.

#### **Listing 16.2.9.7** Mini-Mental State Examination (MMSE) Safety Population Part 2 of 3

| | | Or | Registration | | | Attention and Calculation | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | What is the city/town | What is the building | What is the floor of the building | | | | What is<br>100<br>taken | Keep | Keep | Keep | Keep | |
| Subject | | (or part of city/ | (name | (room number | Word | Word | Word | away | going | going | going | going | Spell |
| IĎ | Visit | neighborhood)? | or type)? | or address)? | 1 | 2 | 3 | 7? | #1 | #2 | #3 | #4 | WORLD <sup>[1]</sup> |
| xxxxxx | Screening | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/5 |
| | Week 26 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/5 |

<sup>[1] &#</sup>x27;N/A' is displayed if the version of the MMSE used did not include this question. [2] Calculated total score may include imputation of missing items.

path\l program.sas date time

**Listing 16.2.9.7** Mini-Mental State Examination (MMSE) Safety Population Part 3 of 3

| | | ] | Recall | | Nan | ning | | Comprehension | | _ | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Fold | Put | | | | ( | Calculated |
| Subject | | Word | Word | Word | l 1.What | 2.What | : | Take in Right | in | on | | | | Total | Total |
| ID | Visit | 1 | 2 | 3 | is this? | is this? | Repetition | Hand | Half | Floo | r Reading V | Vriting | Drawing | Score | Score [2] |
| XXXXXX | Screening | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| | Week 26 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| xxxxxx | Screening | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| | Week 26 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| XXXXXX | Screening | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| | Week 26 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| xxxxxx | Screening | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |
| | Week 26 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | XX | XX |

<sup>[1] &#</sup>x27;N/A' is displayed if the version of the MMSE used did not include this question. [2] Calculated total score may include imputation of missing items.

path\l program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.


#### Listing 16.2.9.8.1 Central Electrocardiogram **Safety Population**

| Subject<br>ID Visit | Assessment Date (Study Day) Measurement | Assessment<br>Time | Heart<br>Rate<br>(bpm) | PR<br>Interval<br>(ms) | RR<br>Interval<br>(ms) | QRS<br>Interval<br>(ms) | - | QTc Interval<br>(Fridericia)<br>(ms) | QTc Interval<br>(Bazett)<br>(ms) | If Abnormal,<br>Describe <sup>[2]</sup> | Any Findings<br>Abnormal? <sup>[3]</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx Screening<br>Week 26 | date9. (xx) 1st Reading<br>date9. (xx) 1st Reading<br>2nd Reading<br>3rd Reading<br>Average [1] | time5.<br>time5.<br>time5. | XXX<br>XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX<br>XXX | | Yes: CS/NCS / No<br>Yes: CS/NCS / No<br>Yes: CS/NCS / No<br>Yes: CS/NCS / No<br>Yes: CS/NCS / No |
| Week 52 | date9. (xx) 1st Reading<br>2nd Reading<br>3rd Reading<br>Average [1] | time5.<br>time5.<br>time5. | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx<br>xxx | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | | Yes: CS/NCS / No<br>Yes: CS/NCS / No<br>Yes: CS/NCS / No<br>Yes: CS/NCS / No |
| xxxxxx Screening | date9. (xx) 1st Reading | time5. | xxx | xxx | xxx | xxx | xxx | xxx | xxx | | Yes: CS/NCS / No |

Note: Study day is calculated as days since the date of first dose of study drug.

[1] Average of triplicate (or available) measurements within a visit.

[2] As reported by the investigator on the ECG central read CRF.

[3] Investigator interpretation of ECG and clinical significance

path\l\_program.sas date time

Programming note: Sort by subject ID. Display the CRF visit label.


#### Listing 16.2.9.8.2 Local Electrocardiogram Safety Population

| | | Assessment | | Heart | PR | RR | QRS | QT | QTc IntervalO | QTc Interva | 1 | If | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date | Assessment | Rate | Interval | Interval | Interval | Interva | l (Fridericia) | (Bazett) | | Abnormal, | Any Findings |
| ID | Visit | (Study Day) | Time | (bpm) | (ms) | (ms) | (ms) | (ms) | (ms) | (ms) | Interpretation | Describe | Abnormal? |
| XXXXXX | Screening | date9. (xx) | time5. | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | Yes: CS/NCS / No |
| | Week 26 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | Yes: CS/NCS / No |
| | Week 52 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | Yes: CS/NCS / No |
| XXXXXX | Screening | date9. (xx) | time5. | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | |
| | Week 26 | date9. (xx) | time5. | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | |

Note: Study day is calculated as days since the date of first dose of study drug.

path\l\_program.sas date time